CLINICAL TRIAL: NCT00413699
Title: A Long-term, Open-label Follow-up Study Of Tofacitinib (Cp-690,550) For Treatment Of Rheumatoid Arthritis
Brief Title: Long-Term Effectiveness And Safety Of CP-690,550 For The Treatment Of Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3921024; 2006-005035-19 (EudraCT Number)
Record Dates: First submitted 2006-12-18; First posted 2006-12-20 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: long-term; open-label; safety
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open-Label Active Treatment Enrolled from Phase 2 (Experimental): Patients enrolling from Phase 2 studies
  Interventions: Drug: CP-690,550
- Open-Label Active Treatment Enrolled from Phase 3 (Experimental): Patients enrolling from Phase 3 studies
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — 5 mg PO BID open label; may increase to 10 mg PO BID to provide greater control of RA if no related AEs are present. May be off study drug temporarily for up to 28 days for mild to moderate AEs.
  Arms: Open-Label Active Treatment Enrolled from Phase 2
Drug: CP-690,550 — 10 mg PO BID open label; may decrease to 5 mg PO BID for mild to moderate AEs. May be off study drug temporarily for up to 28 days for mild to moderate AEs.
  Arms: Open-Label Active Treatment Enrolled from Phase 3

SUMMARY:
The purpose of this study is to determine the long-term effectiveness and safety of CP-690,550 for the treatment of rheumatoid arthritis. Subjects are eligible for this study only after participating in another "qualifying" study of CP-690,550

A sub-study will be conducted within the A3921024 study, this study will evaluate the immune response to pneumococcal and influenza vaccines in patients receiving CP-690,550

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have participated in a randomized "qualifying" study of CP-690,550 for the treatment of rheumatoid arthritis

Vaccine sub-study visit

* Subjects actively participating in Study A3921024 must have completed at least 3 months of continuous 10 mg BID CP-690,550 treatment in A3921024 as defined by >80% compliance with prescribed dose consumption of CP-690,550 over the previous 3 months.

Exclusion Criteria:

* Serious medical conditions that would make treatment with CP-690,550 potentially unsafe

Vaccine sub-study visit

1. Any documented influenza or pneumococcal infection within the last 3 months prior to randomization in this study
2. Received any vaccine within 1 month prior to randomization in this study
3. Received an influenza vaccine within 6 months or a pneumococcal vaccine within 5 years of randomization in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4488 (Actual)
Dates: Start 2007-02-05 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (465):
- United States (147):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Arthrocare, Arthritis Care & Research, PC, Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Radiant Research, Inc., Scottsdale, Arizona
  - Catalina Pointe Clinical Research, Tucson, Arizona
  - CHI St. Vincent Medical Group Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Osborne Research Center, LLC, Little Rock, Arkansas
  - Little Rock Diagnostic Clinic, PA, Little Rock, Arkansas
  - Med Investigations, Inc., Fair Oaks, California
  - Talbert Medical Group, Huntington Beach, California
  - University of California San Diego Center for Innovative Therapy, La Jolla, California
  - Keck Medicine of USC, Los Angeles, California
  - University of Southern California (USC) Norris Comprehensive Cancer Center-, Los Angeles, California
  - University of Southern California (USC) Norris Comprehensive Cancer Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Office of Anupama Bhat, MD, Roseville, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Stanford Health Services - Medical Specialty Clinics, Stanford, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Boulder Medical Center, PC, Boulder, Colorado
  - Arthritis Associates and Osteoporosis Center of Colorado Springs, Colorado Springs, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Arthritis & Osteoporosis Center, PC, Hamden, Connecticut
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Delaware Arthritis and Osteoporosis Center, Newark, Delaware
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Allergy, Asthma, Arthritis, & Lung, Daytona Beach, Florida
  - Physicians Research Alliance LLC, DeBary, Florida
  - Southeastern Arthritis Center, Gainesville, Florida
  - Southeastern Imaging and Diagnostics, Gainesville, Florida
  - Southeastern Integrated Medical PL d/b/a Florida Medical Research Institute, Gainesville, Florida
  - Southeastern Integrated Medical, PL, d/b/a Florida Medical Research Institute, Gainesville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Florida Arthritis Center, P.L., Lake Mary, Florida
  - BayCare Outpatient Imaging at Bardmoor, Largo, Florida
  - Center for Arthritis and Rheumatic Diseases, Miami, Florida
  - Jeffrey Alper MD Research, Naples, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Dr. Jeffrey E. Poiley, MD , Office of, Orlando, Florida
  - Millennium Research, Ormond Beach, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - Florida Arthritis & Osteoporosis Center, Port Richey, Florida
  - Gulf Coast Medical Center, Port Richey, Florida
  - Arthritis & Rheumatic Care Center, South Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Suncoast Medical Clinic, St. Petersburg, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - BayCare Medical Group, Inc, Tampa, Florida
  - Lovelace Scientific Resources, Venice, Florida
  - Venice Arthritis Center, Venice, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Arthritis and Rheumatology of Georgia P.C., Atlanta, Georgia
  - Jeffrey D. Lieberman, MD, PC, Decatur, Georgia
  - Marietta Rheumatology Associates, Marietta, Georgia
  - St. Luke's Clinic - Rheumatology, Boise, Idaho
  - St. Luke's Clinic, Boise, Idaho
  - St. Luke's Intermountain Research Center, Boise, Idaho
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - St. Luke's Clinic - Rhematology, Meridian, Idaho
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois Bone and Joint Institute, LLC, Morton Grove, Illinois
  - Rockford Health Physicians, Rockford, Illinois
  - Rockford Orthopedic Associates, Rockford, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Clinic - Clinical Research, Springfield, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Diagnostic Rheumatology And Research PC, Indianapolis, Indiana
  - Physician's Clinic of Iowa, P.C., Cedar Rapids, Iowa
  - Medical Associates Clinic, PC, Dubuque, Iowa
  - Kansas City Internal Medicine, Overland Park, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Via Christi Clinic, P.A., Wichita, Kansas
  - Bluegrass Community Research, Inc., Lexington, Kentucky
  - Ochsner Clinic Foundation - Baton Rouge, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Rheumatology Associates, Portland, Maine
  - Klein and Associates, MD, PA, Cumberland, Maryland
  - The Arthritis Treatment Center, Frederick, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Research Center of Cape Cod, Inc., Hyannis, Massachusetts
  - Reliant Medical Group, Inc., Worcester, Massachusetts
  - Reliant Medical Group, Inc. at Worcester Medical Center, Worcester, Massachusetts
  - Bronson Internal Medicine and Rheumatology, Battle Creek, Michigan
  - QUEST Research Institiute, Bingham Farms, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - Farmbrook Radiology Associates, Southfield, Michigan
  - Arthritis and Rheumatology Consultants, P.A., Edina, Minnesota
  - North Mississippi Medical Clinics, Inc., Tupelo, Mississippi
  - University Physicians - Woodrail Clinic, Columbia, Missouri
  - University Of Missouri-Columbia, Columbia, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Clinical Pharmacology Study Group, Massachusetts, Nebraska
  - Westroads Clinical Research, Inc., Omaha, Nebraska
  - Heartland Clinic Research, Inc., Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Rheumatology Associates of North Jersey, Teaneck, New Jersey
  - Arthritis, Rheumatic & Back Disease Associates, Voorhees Township, New Jersey
  - The Center for Rheumatology, LLP, Albany, New York
  - Regional Rheumatology Associates, Binghamton, New York
  - Southern Tier Arthritis and Rheumatism, Olean, New York
  - Buffalo Rheumatology and Medicine, PLLC, Orchard Park, New York
  - AAIR Research Center, Rochester, New York
  - Asheville Rheumatology & Osteoporosis Research Associates, P.A., Asheville, North Carolina
  - Asheville Rheumatology & Osteoporosis Research Associates, PA, Asheville, North Carolina
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - PMG Research Hickory, LLC, Hickory, North Carolina
  - PMG Research of Hickory, Hickory, North Carolina
  - Boice-Willis Clinic, Rocky Mount, North Carolina
  - Trinity Health Center - Medical Arts, Minot, North Dakota
  - Cincinnati Rheumatic Disease Study Group, Inc., Cincinnati, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Office of David R. Mandel, MD, Inc., Mayfield, Ohio
  - Oklahoma Medical Research Foundation (OMRF), Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Rheumatic Disease Associates, Ltd., Willow Grove, Pennsylvania
  - Clinical Research Center of Reading LLP, Wyomissing, Pennsylvania
  - Piedmont Arthritis Clinic, PA, Greenville, South Carolina
  - Arthritis Associates, PLLC, Hixson, Tennessee
  - Arthritis Clinic, Jackson, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - Rheumatology Consultants, PLLC, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Office of John P. Lavery, MD, PA, Allen, Texas
  - Austin Rheumatology Research, PA, Austin, Texas
  - Arthritis Care and Diagnostic Center, P.A., Dallas, Texas
  - Baylor Research Institute, Dallas, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - University of North Texas Health Science Center at Fort Worth, Fort Worth, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Arthritis and Osteoporosis Associates, LLP, Lubbock, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Rheumatology Associates, Seattle, Washington
  - The Seattle Arthritis Clinic, Seattle, Washington
  - Tacoma Center of Arthritis Research, PS, Tacoma, Washington
  - The Vancouver Clinic, Inc. PS, Vancouver, Washington
  - Mountain State Clinical Research, Clarksburg, West Virginia
  - Gundersen Clinic, Ltd, Onalaska, Wisconsin
- Argentina (6):
  - OMI- Organizacion Medica de Investigacion, Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Reumatologicas y Osteologicas -CIRO, Buenos Aires, Buenos Aires F.D.
  - Hospital Sirio Libanes, Buenos Aires
  - OMI - Organización Médica de Investigación, Buenos Aires
  - Saint Dennis Medical Group S.A., Buenos Aires
  - Consultorios Reumatologicos Pampa, Buenos Aires
- Australia (7):
  - Optimus Clinical Research Pty. Ltd., Kogarah, New South Wales
  - Rheumatology Research, Cairns, Queensland
  - Rheumatology Research Unit Sunshine Coast, Maroochydore, Queensland
  - Queen Elizabeth Hospital, Department of Rheumatology, Woodville, South Australia
  - Emeritus Research, Malvern East, Victoria
  - Goatcher Clinical Research Unit, Perth, Western Australia
  - Royal North Shore Hospital, St Leonards
- Austria (3):
  - Medizinische Universitaet Wien / AKH, Vienna
  - Rheuma-Ordination Favoriten, Vienna
  - Sozialmedizinisches Zentrum Sued - Kaiser Franz Josef Spital, Vienna
- Belgium (3):
  - Universitair Ziekenhuis Gent - Reumatologie, Ghent, Oost-vlaanderen
  - AZ Groeninge, Kortrijk
  - Centre Hospitalier Universitaire de Liège, Liège
- University Clinical Center Sarajevo, Sarajevo, Bosnia and Herzegovina
- Brazil (9):
  - CIP - Centro Internacional de Pesquisa, Goiânia, Goiás
  - Centro de Estudos em Terapias Inovadoras, Curitiba, Paraná
  - CCBR Brasil Centro de Pesquisas e Analises Clinicas Ltda, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo (HC-FMUSP), São Paulo, São Paulo
  - IMA Brasil -Instituto de Pesquisa Clinica e Medicina Avancada, São Paulo, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica e Servicos Medicos Ltda, São Paulo
- Bulgaria (10):
  - Revmatologichen kabinet, DKTs Sveti Pantaleimon OOD, Pleven
  - Revmatologichno Otdelenie, MBAL - Plovdiv, Plovdiv
  - UMBAL Kaspela Plovdiv, Plovdiv
  - MBAL Akta Medika OOD, Sevlievo
  - Clinic of Cardiology and Rheumatology Military Medical Academy, Sofia
  - Clinic of Rheumatology Multiprofile Hospital for Active treatment Sveti Ivan Rilski, Sofia
  - MBAL Sveti Ivan Rilski Sofia, Sofia
  - DKTs "Sveta Anna" Sofia, Konsultativen kabinet po Revmatologia, Sofia
  - DKTs "Sveta Anna", Sofia / Diagnostic Consultative Center "Sveta Anna", Sofia
  - MOBAL "D-r Stefan Cherkezov" AD,, Veliko Tarnovo
- Canada (22):
  - Rheumatology Research Associates Ltd., Edmonton, Alberta
  - Dr. Alice Klinkhoff, Inc., Vancouver, British Columbia
  - Percuro Clinical Research Limited, Victoria, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Dr. William G. Bensen Medicine Professional Corporation, Hamilton, Ontario
  - Office of Dr. Fernando Bianchi, Hamilton, Ontario
  - Cividino Medicine Professional Corporation, Hamilton, Ontario
  - KW Musculoskeletal Research Inc., Kitchener, Ontario
  - St Joseph's Health Centre, London, Ontario
  - Credit Valley Rheumatology, Missisauga, Ontario
  - The Arthritis Program Research Group Inc., Newmarket, Ontario
  - Rheumatology and Osteoporosis Clinic, Oakville, Ontario
  - Rheumatology Research Associates, Ottawa, Ontario
  - Niagara Peninsula Arthritis Centre, St. Catharines, Ontario
  - Clinical Research and Arthritis Centre, Windsor, Ontario
  - Institut de Rhumatologie de Montreal, Montreal, Quebec
  - West Island Rheumatology Research Associates, Pointe-Claire, Quebec
  - Groupe De Recherche En Rhumatologie Et Maladies Osseuses Inc., Québec, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
  - Arthritis Research Center, Royal University Hospital, Saskatoon, Saskatchewan
- Chile (9):
  - Hospital Base Valdivia, Policlinico de Reumatologia, Valdivia, Region XIV
  - Consulta Privada Dra. Lucia Ponce, Temuco, Región de la Araucanía
  - Centro de Estudios Reumatologicos, Santiago, RM
  - Consulta Privada Dra. Marta Aliste, Santiago, RM
  - Centro de Diagnostico y Tratamiento Hospital San Borja Arriaran, Santiago, Santiago Metropolitan
  - Clinica Santa Maria, Seccion Reumatologia, Providencia, Santiago, RM
  - Hospital Regional de Rancagua, Rancagua
  - Clinica Santa Maria, Santiago
  - Estudios Clinicos V Region, Vina Del Mar, V Region
- China (20):
  - Beijing Chaoyang Hospital, Capital University of Medical Science, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Centre-south University, Changsha, Hunan
  - Xijing Hospital, The Fourth Military Medical University, Xi'an, Shaan'xi
  - QiLu Hospital of Shandong University, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Peking University People's Hospital/Rheumatology and Immunology Department, Beijing
  - PLA General Hospital, Beijing
  - Si Chuan Huaxi Hospital, Chengdu
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Anhui Province Hospital, Hefei
  - An Hui Medical University 1st Hospital, Hefei
  - Jiangsu Province Hospital, Nanjing
  - Rheumatology and Immunology Dept., Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Changhai Hospital, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - "Department of Infectious Diseases & Immunology, Tianjin
- Colombia (4):
  - Centro de Reumatologia y Ortopedia S.A.S., Barranquilla, Atlántico
  - Riesgo de Fractura S.A., Bogota D.C., Cundinamarca
  - Centro de Investigacion en Reumatologia y Especialidades Medicas S.A.S CIREEM S.A.S, Bogota, D.C., Cundinamarca
  - Servimed S.A.S., Bucaramanga, Santander Department
- Costa Rica (3):
  - Centro de Reumatologia y Osteoporosis, Cartago, Cartago
  - Hospital Cima San Jose, San José
  - Oficina Privada Del Colegio deMedicos, San José
- Croatia (5):
  - University Hospital Center Osijek, Osijek
  - University Hospital Split, Department for Internal Medicine, Division of Clinical Rheumatology, Split
  - Clinical Hospital "Sveti Duh", Zagreb
  - University Hospital Center "Zagreb", Zagreb
  - University Hospital Center Zagreb, Zagreb
- Czechia (18):
  - X-MEDICA s.r.o., Brno
  - Revmacentrum MUDr. Mostera, s.r.o., Brno
  - Fakultni Nemocnice Brno, Interni hematoonkologicka klinika, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - HESTE s.r.o. Revmatologie, Česká Lípa
  - MEDIPONT Plus sro, České Budějovice
  - L.K.N. Arthrocentrum, s.r.o., Hlučín
  - ARTMEDI UPD s r.o, Hostivice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Revmatologicka ambulance, Ostrava
  - ARTHROMED, s. r. o. Revmatologicka ambulance, Pardubice
  - Revmatologicky ustav, Prague
  - Revmatologicka ambulance, Prague
  - Fakultni Thomayerova nemocnice s poliklinikou, Prague
  - Nuselska poliklinika RTG, Prague
  - Affidea Praha, s.r.o., Praha 11 - Chodov
  - Nemocnice Atlas, a.s., Zlín
  - PV-Medical s.r.o., Zlín
- Frederiksberg Hospital, Frederiksberg, Denmark
- Hospital Central de las Fuerzas Armadas, Santo Domingo, Dominican Republic
- Finland (3):
  - Helsingin Reumakeskus Oy, Helsinki
  - Kiljavan Laaketutkimus Oy, Hyvinkää
  - TAYS/Reumakeskus/Finn-Medi 1, Tampere
- France (6):
  - Hopital Nord, Amiens
  - Hôpital Nord, Amiens
  - *CHR Hopital Porte Madeleine IPROS, Orléans
  - CHR ORLEANS - Service IPROS, Orléans
  - Hôpital Saint-Antoine, Paris
  - Hopital Cochin, Paris
- Germany (18):
  - Privat-Praxis, Aachen
  - Charite Campus Mitte, Medizinische Klinik mit Schwerpunkt Rheumatologie und Klinische Immunologie, Berlin
  - Schlosspark-Klinik Innere Medizin II, Rheumatologie, Berlin
  - Ambulantes Rheumazentrum Dr Soerensen, Berlin
  - Universitaetsklinikum Koeln Klinik I fuer Innere Medizin, Haus 16, 1. OG, Raum 1.008, Cologne
  - Krankenhaus Friedrichstadt, I. Medizinische Klinik, Dresden
  - Studienambulanz Universitaetsklinikum Erlangen Medizinische Klinik 3, Erlangen
  - J.W.-Goethe-Universitaetsklinik, Medizinische Klinik II, Abteilung fuer Rheumatologie, Frankfurt am Main
  - Schwerpunktpraxis Rheumatologie, Halle
  - Schoen Klinik Hamburg-Eilbek, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Universitaetsklinik Leipzig, Klinik fur Gastroenterologie und Rheumatologie, Sektion Rheumatologie, Leipzig
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Universitaet Muenchen, Campus Innenstadt, Rheuma-Einheit, München
  - Arztpraxis, Internist - Rheumatologie, Nuremberg
  - Rheumaforschung- Studienambulanz, Ratingen
  - Schwerpunktpraxis fuer Rheumatologie, Rheine
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (2):
  - General Hospital Euromedica "KYANOUS STAVROS", Thessaloniki
  - 424 General Army Hospital, Thessaloniki
- Hungary (5):
  - Drug Research Center Kft, Balatonfüred
  - Orszagos Reumatologiai Es Fizioterapias Intezet, Budapest
  - Revita Reumatologiai Rendelo, Budapest
  - Synexus Magyarorszag Kft., Budapest
  - MAV Korhaz es Rendelointezet, Reumatologiai szakrendeles, Szolnok
- India (10):
  - Mahavir Hospital & Research Center, Hyderabad, Andhra Pradesh
  - Rheumatic Diseases Clinic, Ahmedabad, Gujarat
  - Shalby Hospitals, Ahmedabad, Gujarat
  - Chanre Rheumatology and Immunology Center and Research, Bangalore, Karnataka
  - St. John's Medical College and Hospital., Bangalore, Karnataka
  - Shirdi Sai Hospital, Bangalore, Karnataka
  - Chanre Rheumatology & Immunology Center & Research, Bangalore, Karnataka
  - Arthritis Research and Care Foundation Centre for Rheumatic Diseases, Pune, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra
  - Krishna Institute of Medical Sciences Ltd, Secunderabad, Telangana
- St. Vincent's University Hospital, Elm Park, Dublin, Ireland
- Italy (2):
  - A.O.U. Careggi - SOD Medicina Interna 1 e Reumatologia, Florence, FI
  - U.O. Clinica Reumatologica, Genova
- Malaysia (7):
  - Hospital Putrajaya, Dept. of Medicine, Putrajaya, Kuala Lumpur
  - Hospital Tuanku Ja'afar, Seremban, Negeri Sembilan
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Selayang, Batu Caves, Selangor
  - Sunway Medical Centre, Petaling Jaya, Selangor
  - Subang Jaya Medical Centre, Subang Jaya, Selangor
- Mexico (18):
  - Centro de Investigacion del Noroeste, Tijuana, BAJA California Norte
  - Unidad de Enfermedades Reumaticas y Cronico Degenerativas SC, Torreón, Coahuila
  - Centro Integral en Reumatologia, SA de CV, Guadalajara, Jalisco
  - Unidad de Investigacion en Enfermedades Cronico Degenerativas, Guadalajara, Jalisco
  - Centro de Investigacion Clinica Especializada, SC, Coyoacán, Mexico City
  - Hospital Angeles del Pedregal, Mexico City, Mexico City
  - Centro de Investigacion Clinica de Morelia, Morelia, Michoacán
  - Clinica de Enfermedades Cronicas y Procedimientos Especiales SC, Morelia, Michoacán
  - Fundacion El Hospitalito, Cuernavaca, Morelos
  - Hospital Universitario Doctor Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Centro Medico Toluca, Metepec, State of Mexico
  - Unidad Reumatologica Las Americas SCP, Mérida, Yucatán
  - Investigacion y Biomedica de Chihuahua, SC, Chihuahua City
  - Hospital Angeles Mocel, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Centro Reumatologico Queretaro, Querétaro
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi, S.C., San Luis Potosí City
  - Hospital Central Dr Ignacio Morones Prieto Unidad Regional de Reumatologia y Osteoporosis, San Luis Potosí City
- New Zealand (3):
  - The Canterbury Geriatric Medical Research Trust, c/- The Princess Margaret Hospital, Christchurch
  - Waikato Hospital, Rheumatology, Hamilton
  - Clinical Trials Unit, Timaru Hospital, Timaru
- Peru (3):
  - Hospital Nacional IV Alberto Sabogal Sologuren, Callao
  - Centro Medico Corpac/Investigaciones en Reumatologia, Lima
  - Instituto Peruano del Hueso y la Articulacion SAC-Privado-Lima/Centro de Investigacion IPHAR, Lima
- Philippines (7):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - De La Salle University Health Sciences Campus Clinical Epidemiology Unit, Dasmariñas, Cavite
  - Angeles University Foundation Medical Center, Angeles City, Pampanga
  - University of Perpetual Help Rizal Dalta Medical Center, Las Piñas, Philippines
  - Chong Hua Hospital, Cebu City
  - Southern Philippine Medical Center, Davao City
  - University of Santo Tomas Hospital, Manila
- Poland (11):
  - "ZDROWIE OSTEO-MEDIC" s.c. Lidia I Artur Racewicz, Agnieszka I Jerzy Supronik, Bialystok
  - ClinicMed Badurski i wspolnicy Spolka Jawna, Bialystok
  - NSZOZ Medicus II, Cieszyn
  - Szpital im. Teodora Dunina, Kościan
  - Krakowskie Centrum Medyczne NZOZ, Krakow
  - Centrum Badan Klinicznych s.c. Wieslawa Porawska, Lukasz Porawski, Poznan
  - Wojewodzki Zespol Reumatologiczny im. dr Jadwigi Titz-Kosko, Sopot
  - Nzoz "Nasz Lekarz", Torun
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Rheuma-Medicus - Specjalistyczne Centrum Reumatologii i Osteoporozy, Warsaw
  - SYNEXUS Polska Sp. z.o.o., Wroclaw
- Puerto Rico (3):
  - Mindful Medical Research, San Juan, PR
  - Ponce School Of Medicine, Ponce
  - Edificio Parra, Ponce
- Romania (2):
  - Spitalul Clinic "Sf. Maria", Bucharest
  - Spitalul Clinic De Recuperare, Iași
- Russia (19):
  - City Clinical Hospital # 1, Novosibirsk, Novosibirsk Oblast
  - "Consultative Diagnostic Rheumatology Center ""Healthy Joints"", LLC", Novosibirsk, Novosibirsk Oblast
  - State Healthcare Institution City Hospital # 40 of Administrative Health Resort District, Saint Petersburg, Sestroretsk, Russia
  - Smolensk State Medical Academy, Smolensk, Smolensk Oblast
  - State Healthcare Institution Regional Clinical Hospital, Barnaul
  - State Healthcare Institution Regional Clinical Hospital for War Veterans, Kemerovo
  - Russian State Medical University Moscow Faculty City Clinical Hospital #4, Moscow
  - Rheumatology Research Institute of Russian Academy of Medical Sciences, Moscow
  - GUZ Republican Hospital n.a. Baranov, Petrozavodsk
  - Saint-Petersburg State Budgetary Healthcare Institution "Clinical Rheumathology Hospital #25", Saint Petersburg
  - Clinical Hospital #122 named after L.G. Sokolov of the Federal Medical-Biological Agency, Saint Petersburg
  - Federal North-West Medical Research Centre, Saint Petersburg
  - St. Petersburg State Institution of Healthcare Consultative-diagnostic Center #85, Saint Petersburg
  - Regional State Budget Institution Of Healthcare, Tomsk
  - Regional State Budgetary Healthcare Institution of Tomsk Regional Clinical Hospital, Tomsk
  - State Healthcare Institution, Yekaterinburg
  - State Educational Institution of Higher Professional Education Ural State Medical Academy of Federal, Yekaterinburg
  - State Educational Institution of Higher Professional Education, Yekaterinburg
  - Ltd.Medical Association "Novaya Bolnitsa", Yekaterinburg
- Slovakia (10):
  - Reumatologicka ambulancia, Poliklinika Ruzinov, Bratislava
  - NOVAPHARM s.r.o -Zeleznicna NaP, Reumatologicka ambulancia, Bratislava
  - AAGS, s.r.o. , nestatne zdravotnicke zariadenie, Dunajská Streda
  - Interna a reumatologicka ambulancia, Košice
  - Ecclesia, s.r.o Reumatologicka ambulancia, Nové Zámky
  - Narodny Ustav Reumatickych Chorob, Piešťany
  - Reumatologicka ambulancia, MUDr. Zuzana Cizmarikova, s.r.o., Poprad
  - Reumatologicka ambulancia, REUMEX, s.r.o., Rimavská Sobota
  - Reumatologicka ambulancia, Nestatne zdravotnicke zariadenie, Senica
  - Nestatna reumatologicka ambulancia, MUDr. Pavol Polak s.r.o., Žilina
- South Korea (14):
  - Inha University Hospital, Jung-gu, Incheon
  - Eulji University Hospital, Daejeon, Republic of Korea
  - Dong-A University Hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Seoul
  - Hanyang University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center-University of Ulsan College of Medicine, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital-Yonsei University Health System, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul St. Mary's Hospital-The Catholic University of Korea, Seoul
- Spain (15):
  - Hospital Nuestra Senora de la Esperanza, Santiago de Compostela, A Coruna
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruna
  - Hospital de Merida, Mérida, Badajoz
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital de Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Del Mar, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario De La Paz, Madrid
  - Hospital Civil. Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital El Tomillar, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Sweden (6):
  - Falu lasarett, Falun
  - Lanssjukhuset Ryhov, Jönköping
  - Skanes Universitetssjukhus i Malmo Reumamottagningen, Malmo
  - Sundsvalls Sjukhus, Sundsvall
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska University Hospital, Uppsala
- Taiwan (9):
  - Chang Gung Medical Foundation-, Niao Sung Hsiang, Kaohsiung County
  - Chang Gung Medical Foundation-Linkou Branch, Kwei-Shan, Taoyuan County
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (5):
  - Rheumatology Unit, Department of Internal Medicine, Phramongkutklao Hospital, Rajathevee, Bangkok
  - Division of Rheumatology, Department of Internal Medicine, Faculty of Medicine,, Amphoe Mueang, Chiang Mai
  - Division of Allergy-Immunology-Rheumatology, Department of Medicine, Faculty of Medicine, Muang District, Khonkaen
  - Rheumatology Unit, Department of Internal Medicine, Rajavithi Hospital, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok
- Turkey (Türkiye) (3):
  - Ege University Medical Faculty, Bornova, İzmir
  - Hacettepe University Medical Faculty, Ankara
  - Dokuz Eylul Universitesi Arastirma Uygulama Hastanesi, Izmir
- Ukraine (10):
  - Crimean Republican Institution "Clinical Territorial Medical Association "University Clinic",, Simferopol, Autonomous Republic of Crimea
  - CRIMEAN Republican Institution, "Clinical Hospital n.a. M.O. Semashko", Simferopol Crimea, Ukraine
  - Municipal Establishment of Health Care "Kharkiv City Clinical Hospital #8", Dept. of Rheumatology, Kharkiv
  - State Institution Republican Clinical Hospital of the Ministry of Health of Ukraine, Kyiv
  - State Establishment "Institute of Gerontology of NAMS of Ukraine n.a. D.F. Chebotareva", Kyiv
  - Municipal City Clinical Hospital #4, Policlinic Care, Lviv
  - "Multifield Medical Center of Odesa National Medical University ""University Clinic #1""", Odesa
  - Multifield Medical Center of Odesa National Medical University "University Clinic #1", Odesa
  - Vinnitsa Regional Clinical Hospital n.a. Pirogov, Vinnitsa
  - Municipal Establishment "City Hospital#7of Zaporizhzhia State Medical University, Zaporizhzhia
- United Kingdom (4):
  - Dudley Group of Hospitals NHS Trust, Dudley, WEST Midlands
  - The Royal Wolverhampton NHS Trust, Cannock
  - Wirral University Teaching Hospital NHS Foundation Trust-Arrowe Park Hospital, Metropolitan Borough of Wirral
  - Royal Victoria Infirmary, Newcastle upon Tyne

REFERENCES:
- [Derived] Strand V, Schulze-Koops H, Al-Emadi S, Kinch CD, Gruben D, Germino R, Connell CA, Mysler E. Sex differences in the efficacy, safety and persistence of tofacitinib in patients with rheumatoid arthritis: a post hoc analysis of phase III and long-term extension trials. BMJ Open. 2025 Dec 24;15(12):e082366. doi: 10.1136/bmjopen-2023-082366. PMID 41448717
- [Derived] Pope J, Finckh A, Silva-Fernandez L, Mandl P, Fan H, Rivas JL, Valderrama M, Montoro M. Tofacitinib Monotherapy in Rheumatoid Arthritis: Clinical Trials and Real-World Data Contextualization of Patients, Efficacy, and Treatment Retention. Open Access Rheumatol. 2024 Jun 11;16:115-126. doi: 10.2147/OARRR.S446431. eCollection 2024. PMID 38883150
- [Derived] Curtis JR, Wollenhaupt J, Tas SW, Chatzidionysiou K, Wang L, Roberts K, Tsekouras V. Determinants of tofacitinib discontinuation in adult patients with rheumatoid arthritis during long-term extension studies up to 9.5 years. Rheumatol Adv Pract. 2024 May 11;8(2):rkae063. doi: 10.1093/rap/rkae063. eCollection 2024. PMID 38854417
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Mueller RB, Schulze-Koops H, Furst DE, Cohen SB, Kwok K, Wang L, Killeen T, von Kempis J. Effect of dose adjustments on the efficacy and safety of tofacitinib in patients with rheumatoid arthritis: a post hoc analysis of an open-label, long-term extension study (ORAL Sequel). Clin Rheumatol. 2022 Apr;41(4):1045-1055. doi: 10.1007/s10067-021-05908-z. Epub 2022 Jan 1. PMID 34973077
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] van der Heijde D, Landewe RBM, Wollenhaupt J, Strengholt S, Terry K, Kwok K, Wang L, Cohen S. Assessment of radiographic progression in patients with rheumatoid arthritis treated with tofacitinib in long-term studies. Rheumatology (Oxford). 2021 Apr 6;60(4):1708-1716. doi: 10.1093/rheumatology/keaa476. PMID 33057725
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Kaine J, Tesser J, Takiya L, DeMasi R, Wang L, Snyder M, Soma K, Fan H, Bandi V, Wollenhaupt J. Re-establishment of efficacy of tofacitinib, an oral JAK inhibitor, after temporary discontinuation in patients with rheumatoid arthritis. Clin Rheumatol. 2020 Jul;39(7):2127-2137. doi: 10.1007/s10067-020-04956-1. Epub 2020 Feb 12. PMID 32048083
- [Derived] Wollenhaupt J, Lee EB, Curtis JR, Silverfield J, Terry K, Soma K, Mojcik C, DeMasi R, Strengholt S, Kwok K, Lazariciu I, Wang L, Cohen S. Safety and efficacy of tofacitinib for up to 9.5 years in the treatment of rheumatoid arthritis: final results of a global, open-label, long-term extension study. Arthritis Res Ther. 2019 Apr 5;21(1):89. doi: 10.1186/s13075-019-1866-2. PMID 30953540
- [Derived] Li ZG, Liu Y, Xu HJ, Chen ZW, Bao CD, Gu JR, Zhao DB, An Y, Hwang LJ, Wang L, Kremer J, Wu QZ. Efficacy and Safety of Tofacitinib in Chinese Patients with Rheumatoid Arthritis. Chin Med J (Engl). 2018 Nov 20;131(22):2683-2692. doi: 10.4103/0366-6999.245157. PMID 30425195
- [Derived] Hall S, Nash P, Rischmueller M, Bossingham D, Bird P, Cook N, Witcombe D, Soma K, Kwok K, Thirunavukkarasu K. Tofacitinib, an Oral Janus Kinase Inhibitor: Pooled Efficacy and Safety Analyses in an Australian Rheumatoid Arthritis Population. Rheumatol Ther. 2018 Dec;5(2):383-401. doi: 10.1007/s40744-018-0118-2. Epub 2018 Jun 11. PMID 29949132
- [Derived] Fleischmann R, Wollenhaupt J, Takiya L, Maniccia A, Kwok K, Wang L, van Vollenhoven RF. Safety and maintenance of response for tofacitinib monotherapy and combination therapy in rheumatoid arthritis: an analysis of pooled data from open-label long-term extension studies. RMD Open. 2017 Dec 18;3(2):e000491. doi: 10.1136/rmdopen-2017-000491. eCollection 2017. PMID 29435359
- [Derived] Fleischmann R, Wollenhaupt J, Cohen S, Wang L, Fan H, Bandi V, Andrews J, Takiya L, Bananis E, Weinblatt ME. Effect of Discontinuation or Initiation of Methotrexate or Glucocorticoids on Tofacitinib Efficacy in Patients with Rheumatoid Arthritis: A Post Hoc Analysis. Rheumatol Ther. 2018 Jun;5(1):203-214. doi: 10.1007/s40744-018-0093-7. Epub 2018 Feb 7. PMID 29417430
- [Derived] Mariette X, Chen C, Biswas P, Kwok K, Boy MG. Lymphoma in the Tofacitinib Rheumatoid Arthritis Clinical Development Program. Arthritis Care Res (Hoboken). 2018 May;70(5):685-694. doi: 10.1002/acr.23421. Epub 2018 Apr 2. PMID 28941219
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Genovese MC, van Vollenhoven RF, Wilkinson B, Wang L, Zwillich SH, Gruben D, Biswas P, Riese R, Takiya L, Jones TV. Switching from adalimumab to tofacitinib in the treatment of patients with rheumatoid arthritis. Arthritis Res Ther. 2016 Jun 23;18:145. doi: 10.1186/s13075-016-1049-3. PMID 27334658
- [Derived] Winthrop KL, Silverfield J, Racewicz A, Neal J, Lee EB, Hrycaj P, Gomez-Reino J, Soma K, Mebus C, Wilkinson B, Hodge J, Fan H, Wang T, Bingham CO 3rd. The effect of tofacitinib on pneumococcal and influenza vaccine responses in rheumatoid arthritis. Ann Rheum Dis. 2016 Apr;75(4):687-95. doi: 10.1136/annrheumdis-2014-207191. Epub 2015 Mar 20. PMID 25795907
- [Derived] Boyle DL, Soma K, Hodge J, Kavanaugh A, Mandel D, Mease P, Shurmur R, Singhal AK, Wei N, Rosengren S, Kaplan I, Krishnaswami S, Luo Z, Bradley J, Firestein GS. The JAK inhibitor tofacitinib suppresses synovial JAK1-STAT signalling in rheumatoid arthritis. Ann Rheum Dis. 2015 Jun;74(6):1311-6. doi: 10.1136/annrheumdis-2014-206028. Epub 2014 Nov 14. PMID 25398374
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921024&StudyName=Long-Term%20Effectiveness%20And%20Safety%20Of%20CP-690%2C550%20For%20The%20Treatment%20Of%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial period (IP): conducted at multiple sites, participants were assigned to Tofacitinib 5 mg and 10 mg BID. Extension period (EP): participants who took part initially in IP, completed 2 years of lymphocyte assessment in IP, given consent, were enrolled in EP and assigned to "Extension Period: Tofacitinib 5 mg". EP was conducted in 2 countries.
Pre-assignment Details: Participants had previously participated in qualifying studies (A3921019, A3921025, A3921032, A3921035, A3921044, A3921045, A3921046, A3921064, A3921068, A3921069, A3921073, A3921109, A3921129, A3921130, A3921152, A3921237) prior to enrollment in initial period.
Groups:
- Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID): Participants with non-zero average total daily dose across study <15 were assigned to 5 mg BID.
- Initial Period: Tofacitinib 10 mg BID: Participants with average total daily dose across study >=15 were assigned to 10 mg BID.
- Extension Period: Tofacitinib 5 mg: Participants who completed 2 years of lymphocyte assessment in Initial period and enrolled for Extension period received Tofacitinib (CP-690,550) 5 mg orally, twice daily up to 12 months.
Period: Initial Period
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Extension Period: Tofacitinib 5 mg
Started | 1123 | 3358 | 0
Completed | 484 | 1653 | 0
Not Completed | 639 | 1705 | 0
Not completed — Death | 25 | 30 | 0
Not completed — Lack of Efficacy | 59 | 115 | 0
Not completed — Lost to Follow-up | 31 | 101 | 0
Not completed — Protocol Violation | 38 | 89 | 0
Not completed — Pregnancy | 10 | 8 | 0
Not completed — Did not meet entrance criteria | 2 | 2 | 0
Not completed — Medication error without adverse event | 0 | 1 | 0
Not completed — Study terminated by Sponsor | 0 | 1 | 0
Not completed — Other | 67 | 211 | 0
Not completed — Adverse event related to study drug | 178 | 527 | 0
Not completed — Adverse event not related to study drug | 113 | 248 | 0
Not completed — Missing end of study page | 0 | 4 | 0
Not completed — No longer willing to participate | 116 | 368 | 0
Period: Extension Period
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Extension Period: Tofacitinib 5 mg
Started | 0 | 0 | 48
Completed | 0 | 0 | 43
Not Completed | 0 | 0 | 5
Not completed — No Longer Willing to Participate | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Total
Number analyzed (Participants) | 1123 | 3358 | 4481
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  18 to 64 years | 916 | 2838 | 3754
  >=65 years | 207 | 520 | 727
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 927 | 2744 | 3671
  Male | 196 | 614 | 810

OUTCOME MEASURES:

1. Primary Outcome: Initial Period: Primary Endpoints Were Standard Laboratory Safety Data (Chemistry, Hematology, Etc.) and Adverse Event (AE) Reports
Description: Treatment-emergent non serious AEs by System Organ Class (SOC) (all causalities) and Laboratory Test Abnormalities (without regard to baseline) The stated number of participants analyzed was the total number of participants in each group (AEs). The actual number of participants analyzed for each laboratory parameter varied, and is provided for each.
  Abs=absolute; ALT=alanine aminotransferase; AST=aspartate aminotransferase; ESR=erythrocyte sedimentation rate; GGT=gamma glutamyl transferase; hgb=hemoglobin; HDL=high density lipids; LDL=low density lipids; LLN=lower limit of normal; qual=qualitative; Tot=total; ULN=upper limit of normal; WBC=white blood cell
Time Frame: Includes laboratory test abnormality data for all visits and adverse event data up to 999 days after last dose of study drug
Population: For abnormal laboratory results, those listed include both mandatory and optional laboratory tests. The number of participants analyzed is the number with at least one evaluable observation of the given laboratory test. Fasting lipids were only collected from participants who enrolled more than 14 days after last visit of their qualifying study.
Measure: Number; unit: Number of participants
Groups:
- Initial Period: All Tofacitinib: All participants treated with tofacitinib 5 mg BID and 10 mg BID groups in initial period.
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib
Number analyzed (Participants) | 1123 | 3358 | 4481
Number of participants
  Participants with non-serious AEs | 991 | 2963 | 3954
  Blood and lymphatic system disorders | 159 | 395 | 554
  Cardiac disorders | 93 | 185 | 278
  Congenital, familial and genetic disorders | 6 | 16 | 22
  Ear and labyrinth disorders | 67 | 138 | 205
  Endocrine disorders | 29 | 94 | 123
  Eye disorders | 117 | 259 | 376
  Gastrointestinal disorders | 393 | 1011 | 1404
  General disorders and admin site conditions | 169 | 477 | 646
  Hepatobiliary disorders | 60 | 176 | 236
  Immune system disorders | 18 | 87 | 105
  Infections and infestations | 704 | 2200 | 2904
  Injury, poisoning and procedural complications | 244 | 721 | 965
  Investigations | 402 | 995 | 1397
  Metabolism and nutrition disorders | 184 | 562 | 746
  Musculoskeletal and connective tissue disorders | 425 | 1314 | 1739
  Neoplasms benign, malignant and unspecified | 80 | 219 | 299
  Nervous system disorders | 222 | 639 | 861
  Pregnancy, puerperium and perinatal conditions | 1 | 0 | 1
  Product issues | 2 | 8 | 10
  Psychiatric disorders | 97 | 280 | 377
  Renal and urinary disorders | 123 | 265 | 388
  Reproductive system and breast disorders | 89 | 206 | 295
  Respiratory, thoracic and mediastinal disorders | 208 | 634 | 842
  Skin and subcutaneous tissue disorders | 201 | 682 | 883
  Social circumstances | 1 | 5 | 6
  Surgical and medical procedures | 2 | 4 | 6
  Vascular disorders | 207 | 468 | 675
  Participants evaluable for lab abnormalities | 1118 | 3346 | 4464
  Participants with laboratory abnormalities | 1095 | 3208 | 4303
  Hemoglobin <0.8x LLN: number analyzed (Participants) | 1117 | 3343 | 4460
  Hemoglobin <0.8x LLN | 57 | 148 | 205
  Hematocrit <0.8x LLN: number analyzed (Participants) | 1117 | 3343 | 4460
  Hematocrit <0.8x LLN | 29 | 67 | 96
  Red blood cell count <0.8x LLN: number analyzed (Participants) | 1049 | 3343 | 4392
  Red blood cell count <0.8x LLN | 32 | 142 | 174
  Reticulocytes (Abs) <0.5x LLN: number analyzed (Participants) | 570 | 75 | 645
  Reticulocytes (Abs) <0.5x LLN | 44 | 5 | 49
  Reticulocytes (Abs) >1.5x ULN: number analyzed (Participants) | 570 | 75 | 645
  Reticulocytes (Abs) >1.5x ULN | 49 | 9 | 58
  Platelets <0.5x LLN: number analyzed (Participants) | 1116 | 3343 | 4459
  Platelets <0.5x LLN | 5 | 2 | 7
  Platelets >1.75x ULN: number analyzed (Participants) | 1116 | 3343 | 4459
  Platelets >1.75x ULN | 5 | 25 | 30
  Reticulocyte count (%) <0.5x LLN: number analyzed (Participants) | 46 | 34 | 80
  Reticulocyte count (%) <0.5x LLN | 1 | 1 | 2
  Reticulocyte count (%) >1.5x ULN: number analyzed (Participants) | 46 | 34 | 80
  Reticulocyte count (%) >1.5x ULN | 24 | 17 | 41
  WBC count <0.6x LLN: number analyzed (Participants) | 1117 | 3343 | 4460
  WBC count <0.6x LLN | 21 | 33 | 54
  WBC count >1.5x ULN: number analyzed (Participants) | 1117 | 3343 | 4460
  WBC count >1.5x ULN | 29 | 71 | 100
  Lymphocytes (Abs) <0.8x LLN: number analyzed (Participants) | 1117 | 3343 | 4460
  Lymphocytes (Abs) <0.8x LLN | 254 | 789 | 1043
  Lymphocytes (Abs) >1.2x ULN: number analyzed (Participants) | 1117 | 3343 | 4460
  Lymphocytes (Abs) >1.2x ULN | 23 | 94 | 117
  Lymphocytes (%) <0.8x LLN: number analyzed (Participants) | 1043 | 3343 | 4386
  Lymphocytes (%) <0.8x LLN | 401 | 1267 | 1668
  Lymphocytes (%) >1.2x ULN: number analyzed (Participants) | 1043 | 3343 | 4386
  Lymphocytes (%) >1.2x ULN | 23 | 75 | 98
  Tot neutrophils (Abs) <0.8x LLN: number analyzed (Participants) | 1117 | 3343 | 4460
  Tot neutrophils (Abs) <0.8x LLN | 105 | 305 | 410
  Tot neutrophils (Abs) >1.2x ULN: number analyzed (Participants) | 1117 | 3343 | 4460
  Tot neutrophils (Abs) >1.2x ULN | 239 | 617 | 856
  Neutrophils (%) <0.8x LLN: number analyzed (Participants) | 1042 | 3343 | 4385
  Neutrophils (%) <0.8x LLN | 23 | 75 | 98
  Neutrophils (%) >1.2x ULN: number analyzed (Participants) | 1042 | 3343 | 4385
  Neutrophils (%) >1.2x ULN | 29 | 93 | 122
  Basophils (Abs) >1.2x ULN: number analyzed (Participants) | 1117 | 3343 | 4460
  Basophils (Abs) >1.2x ULN | 19 | 10 | 29
  Basophils (%) >1.2x ULN: number analyzed (Participants) | 1043 | 3343 | 4386
  Basophils (%) >1.2x ULN | 76 | 221 | 297
  Eosinophils (Abs) >1.2x ULN: number analyzed (Participants) | 1117 | 3343 | 4460
  Eosinophils (Abs) >1.2x ULN | 24 | 58 | 82
  Eosinophils (%) >1.2x ULN: number analyzed (Participants) | 1043 | 3343 | 4386
  Eosinophils (%) >1.2x ULN | 36 | 118 | 154
  Monocytes (Abs) >1.2x ULN: number analyzed (Participants) | 1117 | 3343 | 4460
  Monocytes (Abs) >1.2x ULN | 65 | 107 | 172
  Monocytes (%) >1.2x ULN: number analyzed (Participants) | 1043 | 3343 | 4386
  Monocytes (%) >1.2x ULN | 128 | 405 | 533
  ESR >1.5x ULN: number analyzed (Participants) | 1113 | 3343 | 4456
  ESR >1.5x ULN | 872 | 2411 | 3283
  Total bilirubin >1.5x ULN: number analyzed (Participants) | 1117 | 3345 | 4462
  Total bilirubin >1.5x ULN | 18 | 38 | 56
  Direct bilirubin >1.5x ULN: number analyzed (Participants) | 1088 | 3344 | 4432
  Direct bilirubin >1.5x ULN | 5 | 14 | 19
  Indirect bilirubin >1.5x ULN: number analyzed (Participants) | 1041 | 3344 | 4385
  Indirect bilirubin >1.5x ULN | 4 | 18 | 22
  AST >3.0x ULN: number analyzed (Participants) | 1117 | 3344 | 4461
  AST >3.0x ULN | 52 | 111 | 163
  ALT >3.0x ULN: number analyzed (Participants) | 1117 | 3345 | 4462
  ALT >3.0x ULN | 87 | 189 | 276
  GGT >3.0x ULN: number analyzed (Participants) | 1118 | 3345 | 4463
  GGT >3.0x ULN | 82 | 239 | 321
  Alkaline phosphatase >3.0x ULN: number analyzed (Participants) | 1118 | 3345 | 4463
  Alkaline phosphatase >3.0x ULN | 3 | 10 | 13
  Total protein <0.8x LLN: number analyzed (Participants) | 1118 | 3345 | 4463
  Total protein <0.8x LLN | 1 | 0 | 1
  Total protein >1.2x ULN: number analyzed (Participants) | 1118 | 3345 | 4463
  Total protein >1.2x ULN | 2 | 4 | 6
  Albumin <0.8x LLN: number analyzed (Participants) | 1118 | 3345 | 4463
  Albumin <0.8x LLN | 11 | 28 | 39
  Albumin >1.2x ULN: number analyzed (Participants) | 1118 | 3345 | 4463
  Albumin >1.2x ULN | 0 | 0 | 0
  Blood urea nitrogen >1.3x ULN: number analyzed (Participants) | 1118 | 3345 | 4463
  Blood urea nitrogen >1.3x ULN | 87 | 126 | 213
  Creatinine >1.3x ULN: number analyzed (Participants) | 1118 | 3345 | 4463
  Creatinine >1.3x ULN | 52 | 95 | 147
  Cholesterol >1.3x ULN: number analyzed (Participants) | 1104 | 3345 | 4449
  Cholesterol >1.3x ULN | 42 | 130 | 172
  HDL Cholesterol <0.8x LLN: number analyzed (Participants) | 1097 | 3301 | 4398
  HDL Cholesterol <0.8x LLN | 32 | 59 | 91
  LDL Cholesterol >1.2x ULN: number analyzed (Participants) | 1094 | 3293 | 4387
  LDL Cholesterol >1.2x ULN | 69 | 145 | 214
  Triglycerides >1.3x ULN: number analyzed (Participants) | 1096 | 3300 | 4396
  Triglycerides >1.3x ULN | 196 | 373 | 569
  Sodium <0.95x LLN: number analyzed (Participants) | 1118 | 3345 | 4463
  Sodium <0.95x LLN | 6 | 19 | 25
  Sodium >1.05x ULN: number analyzed (Participants) | 1118 | 3345 | 4463
  Sodium >1.05x ULN | 11 | 18 | 29
  Potassium <0.9x LLN: number analyzed (Participants) | 1118 | 3345 | 4463
  Potassium <0.9x LLN | 28 | 62 | 90
  Potassium >1.1x ULN: number analyzed (Participants) | 1118 | 3345 | 4463
  Potassium >1.1x ULN | 11 | 25 | 36
  Chloride <0.9x LLN: number analyzed (Participants) | 1118 | 3345 | 4463
  Chloride <0.9x LLN | 3 | 5 | 8
  Chloride >1.1x ULN: number analyzed (Participants) | 1118 | 3345 | 4463
  Chloride >1.1x ULN | 0 | 1 | 1
  Calcium <0.9x LLN: number analyzed (Participants) | 1041 | 3345 | 4386
  Calcium <0.9x LLN | 2 | 8 | 10
  Calcium >1.1x ULN: number analyzed (Participants) | 1041 | 3345 | 4386
  Calcium >1.1x ULN | 6 | 9 | 15
  Bicarbonate (venous) <0.9x LLN: number analyzed (Participants) | 1117 | 3345 | 4462
  Bicarbonate (venous) <0.9x LLN | 106 | 277 | 383
  Bicarbonate (venous) >1.1x ULN: number analyzed (Participants) | 1117 | 3345 | 4462
  Bicarbonate (venous) >1.1x ULN | 1 | 5 | 6
  Glucose <0.6x LLN: number analyzed (Participants) | 1118 | 3345 | 4463
  Glucose <0.6x LLN | 3 | 4 | 7
  Glucose >1.5x ULN: number analyzed (Participants) | 1118 | 3345 | 4463
  Glucose >1.5x ULN | 125 | 345 | 470
  Creatine Kinase >2.0x ULN: number analyzed (Participants) | 1041 | 3345 | 4386
  Creatine Kinase >2.0x ULN | 203 | 908 | 1111
  C-reactive protein >1.25x ULN: number analyzed (Participants) | 697 | 242 | 939
  C-reactive protein >1.25x ULN | 365 | 106 | 471
  Urine specific gravity <1.003: number analyzed (Participants) | 1098 | 3319 | 4417
  Urine specific gravity <1.003 | 2 | 7 | 9
  Urine specific gravity >1.030: number analyzed (Participants) | 1098 | 3319 | 4417
  Urine specific gravity >1.030 | 203 | 303 | 506
  Urine pH <4.5: number analyzed (Participants) | 1098 | 3319 | 4417
  Urine pH <4.5 | 0 | 0 | 0
  Urine pH >8: number analyzed (Participants) | 1098 | 3319 | 4417
  Urine pH >8 | 20 | 17 | 37
  Urine glucose (qual) ≥1: number analyzed (Participants) | 1095 | 3319 | 4414
  Urine glucose (qual) ≥1 | 60 | 148 | 208
  Urine ketones (qual) ≥1: number analyzed (Participants) | 686 | 103 | 789
  Urine ketones (qual) ≥1 | 2 | 1 | 3
  Urine protein (qual) ≥1: number analyzed (Participants) | 1097 | 3319 | 4416
  Urine protein (qual) ≥1 | 65 | 222 | 287
  Urine blood/hgb (qual) ≥1: number analyzed (Participants) | 1098 | 3319 | 4417
  Urine blood/hgb (qual) ≥1 | 444 | 1260 | 1704
  Urine leukocyte esterase ≥1: number analyzed (Participants) | 687 | 132 | 819
  Urine leukocyte esterase ≥1 | 158 | 23 | 181
  Urine red blood cells ≥20: number analyzed (Participants) | 678 | 1498 | 2176
  Urine red blood cells ≥20 | 198 | 491 | 689
  Urine WBC ≥20: number analyzed (Participants) | 689 | 1603 | 2292
  Urine WBC ≥20 | 219 | 507 | 726
  Urine epithelial cells ≥6: number analyzed (Participants) | 422 | 38 | 460
  Urine epithelial cells ≥6 | 205 | 20 | 225
  Urine casts >1: number analyzed (Participants) | 420 | 38 | 458
  Urine casts >1 | 0 | 0 | 0
  Urine granular casts >1: number analyzed (Participants) | 0 | 2 | 2
  Urine granular casts >1 |  | 0 | 0
  Urine hyaline casts >1: number analyzed (Participants) | 14 | 60 | 74
  Urine hyaline casts >1 | 0 | 0 | 0
  Urine bacteria >20: number analyzed (Participants) | 384 | 35 | 419
  Urine bacteria >20 | 0 | 0 | 0

2. Primary Outcome: Extension Period: Number of Participants With Treatment Emergent Adverse Events (AEs), Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Day 1 at Entry of Extension Period) up to 28 days after last study drug dose in Extension Period (13 Months)
Population: Safety analysis set included all participants who enrolled for extension period and received at least 1 dose of open label study medication in extension period.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Period: Tofacitinib 5 mg
Number analyzed (Participants) | 48
Participants
  Participants with AEs | 16
  Participants with SAEs | 5

3. Primary Outcome: Extension Period: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for laboratory abnormalities: hemoglobin (Hg), hematocrit, red blood cell (RBC), high density lipoprotein (HDL) cholesterol:<0.8*lower limit of normal (LLN), platelet<0.5*LLN/>1.75*upper limit of normal (ULN), white blood cell (WBC)<0.6*LLN/>1.5*ULN, lymphocyte, neutrophil, protein, albumin <0.8*LLN/>1.2*ULN, basophil, eosinophil, monocyte, low density lipoprotein (LDL) cholesterol: >1.2*ULN; bilirubin>1.5*ULN, aspartate amino transferase(AT), alanine AT, gammaglutamyl transferase, alkaline phosphatase:>3.0*ULN; blood urea nitrogen, creatinine, cholesterol, triglyceride:>1.3*ULN; sodium <0.95*LLN/>1.05*ULN, potassium, chloride, calcium, bicarbonate: <0.9*LLN/>1.1*ULN; glucose<0.6*LLN/>1.5*ULN; Urine (specific gravity<1.003/>1.030, pH<4.5/>8, glucose, ketone, protein, blood/Hg(>=1; RBC, WBC>=20; creatinine kinase>2*ULN).
Time Frame: Baseline (Day 1 at Entry of Extension Period) up to 28 days after last study drug dose in Extension Period (13 Months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Period: Tofacitinib 5 mg
Number analyzed (Participants) | 48
Participants | 30

4. Primary Outcome: Initial Period: The Long Term Safety and Tolerability of CP-690,550 5 Milligrams (mg) Twice Daily (BID) and 10 mg BID for the Treatment of Rheumatoid Arthritis
Description: Treatment-emergent AEs by SOC (all causalities) - all participants, by time. Data presented for Post Month 96 includes data up to and including Month 114.
Time Frame: Includes AEs for every visit and up to 999 days after last dose of study drug
Population: The stated number of participants analyzed is the total number of participants enrolled in each group. The number of evaluable participants is the number remaining in the study in the given time period.
Measure: Number; unit: Number of participants
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib
Number analyzed (Participants) | 1123 | 3358 | 4481
Number of participants
  Evaluable for AEs at Months 0 to 6 | 1123 | 3358 | 4481
  Percent with AEs at Months 0 to 6 | 59.4 | 61.8 | 61.2
  Percent discontinued due to AEs at Months 0 to 6 | 4.2 | 4.0 | 4.0
  Evaluable for AEs at Months 6 to 12 | 1033 | 3121 | 4154
  Percent with AEs at Months 6 to 12 | 45.1 | 47.7 | 47.1
  Percent discontinued due to AEs at Months 6 to 12 | 2.1 | 3.7 | 3.3
  Evaluable for AEs at Months 12 to 18 | 969 | 2865 | 3834
  Percent with AEs at Months 12 to 18 | 41.2 | 46.8 | 45.4
  Percent discontinued due to AEs at Months 12 to 18 | 3.2 | 3.4 | 3.3
  Evaluable at Months 18 to 24 | 896 | 2660 | 3556
  Percent with AEs at Months 18 to 24 | 38.1 | 43.2 | 41.9
  Percent discontinued due to AEs at Months 18 to 24 | 2.8 | 2.9 | 2.9
  Evaluable for AEs at Months 24 to 30 | 820 | 2461 | 3281
  Percent with AEs at Months 24 to 30 | 40.7 | 44.5 | 43.5
  Percent discontinued due to AEs at Months 24 to 30 | 3.2 | 2.8 | 2.9
  Evaluable for AEs at Months 30 to 36 | 774 | 2288 | 3062
  Percent with AEs at Months 30 to 36 | 39.0 | 40.7 | 40.3
  Percent discontinued due to AEs at Months 30 to 36 | 2.6 | 2.5 | 2.5
  Evaluable for AEs at Months 36 to 42 | 729 | 2162 | 2891
  Percent with AEs at Months 36 to 42 | 38.1 | 37.5 | 37.6
  Percent discontinued due to AEs at Months 36 to 42 | 2.5 | 2.5 | 2.5
  Evaluable for AEs at Months 42 to 48 | 652 | 1843 | 2495
  Percent with AEs at Months 42 to 48 | 37.9 | 34.3 | 35.3
  Percent discontinued due to AEs at Months 42 to 48 | 2.8 | 2.9 | 2.9
  Evaluable for AEs at Months 48 to 54 | 558 | 1471 | 2029
  Percent with AEs at Months 48 to 54 | 36.0 | 36.4 | 36.3
  Percent discontinued due to AEs at Months 48 to 54 | 2.0 | 2.5 | 2.4
  Evaluable for AEs at Months 54 to 60 | 466 | 1172 | 1638
  Percent with AEs at Months 54 to 60 | 37.1 | 35.4 | 35.9
  Percent discontinued due to AEs at Months 54 to 60 | 3.6 | 2.7 | 3.0
  Evaluable for AEs at Months 60 to 66 | 414 | 918 | 1332
  Percent with AEs at Months 60 to 66 | 33.8 | 31.4 | 32.1
  Percent discontinued due to AEs at Months 60 to 66 | 2.4 | 1.9 | 2.0
  Evaluable for AEs at Months 66 to 72 | 379 | 670 | 1049
  Percent with AEs at Months 66 to 72 | 33.5 | 21.6 | 25.9
  Percent discontinued due to AEs at Months 66 to 72 | 3.2 | 0.7 | 1.6
  Evaluable for AEs at Months 72 to 78 | 336 | 262 | 598
  Percent with AEs at Months 72 to 78 | 33.6 | 22.5 | 28.8
  Percent discontinued due to AEs at Months 72 to 78 | 0.9 | 0.4 | 0.7
  Evaluable for AEs at Months 78 to 84 | 302 | 86 | 388
  Percent with AEs at Months 78 to 84 | 36.8 | 26.7 | 34.5
  Percent discontinued due to AEs at Months 78 to 84 | 3.3 | 1.2 | 2.8
  Evaluable for AEs at Months 84 to 90 | 273 | 42 | 315
  Percent with AEs at Months 84 to 90 | 30.8 | 35.7 | 31.4
  Percent discontinued due to AEs at Months 84 to 90 | 1.8 | 0 | 1.6
  Evaluable for AEs at Months 90 to 96 | 234 | 34 | 268
  Percent with AEs at Months 90 to 96 | 21.8 | 29.4 | 22.8
  Percent discontinued due to AEs at Months 90 to 96 | 0.9 | 0 | 0.7
  Evaluable for AEs post Month 96 | 130 | 15 | 145
  Percent with AEs post Month 96 | 20.8 | 46.7 | 23.4
  Percent discontinued due to AEs post Month 96 | 1.5 | 0 | 1.4

5. Primary Outcome: Extension Period: Percentage of Participants With Adverse Events and Who Discontinued Treatment Due to Adverse Events to Assess Long-term Safety and Tolerability of Tofacitinib
Description: Long term safety and tolerability of Tofacitinib was measured as following: percentage (%) of participants with AEs, percentage of participants who discontinued due to AEs. An AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline (Day 1 at Entry of Extension Period) up to Month 6 of Extension Period; Month 6 of Extension Period to Month 12 of Extension Period
Population: Safety analysis set included all participants who enrolled for extension period and received at least 1 dose of open label study medication in extension period. Here, "Number Analyzed" signifies number of participants evaluable for specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Extension Period: Tofacitinib 5 mg
Number analyzed (Participants) | 48
Percentage of participants
  Baseline to Month 6: % of Participants with AEs | 31.3
  Baseline to Month6:% of Participants Discontinued | 4.2
  Month 6 to 12: % of Participants with AEs: number analyzed (Participants) | 17
  Month 6 to 12: % of Participants with AEs | 17.6
  Month 6 to 12: % of Participants Discontinued: number analyzed (Participants) | 17
  Month 6 to 12: % of Participants Discontinued | 0

6. Secondary Outcome: Initial Period: Percentage of Patients With American College of Rheumatology (ACR) 20, 50, and 70 Responses
Description: The stated number of participants analyzed was the total number of participants in each group. The actual number of participants analyzed on each occasion varied, and is provided for each visit presented. ACR20 is defined as a 20% improvement from baseline in tender/painful joint count and swollen joint count, and at least 3 of the following 5 variables: Subject's Global Assessment of Arthritis, Physician's Global Assessment of Arthritis, Subject's Assessment of Arthritis Pain, Health Assessment Questionnaire - Disability Index, C-Reactive Protein (CRP). ACR50 is a 50% improvement and ACR70 a 70% improvement in these variables.
Time Frame: Every visit until study completion
Population: The number of participants analyzed is the number remaining in the study who had evaluable data for the measure at the given time point.
Measure: Number; unit: Percent of participants
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib
Number analyzed (Participants) | 1123 | 3358 | 4481
Percent of participants
  ACR20 at Month 1: number analyzed (Participants) | 1114 | 3307 | 4421
  ACR20 at Month 1 | 70.65 | 73.60 | 72.86
  ACR20 at Month 2: number analyzed (Participants) | 1080 | 3254 | 4334
  ACR20 at Month 2 | 74.81 | 76.06 | 75.75
  ACR20 at Month 3: number analyzed (Participants) | 1069 | 3228 | 4297
  ACR20 at Month 3 | 75.68 | 78.00 | 77.43
  ACR20 at Month 6: number analyzed (Participants) | 1040 | 3132 | 4172
  ACR20 at Month 6 | 75.58 | 77.36 | 76.92
  ACR20 at Month 9: number analyzed (Participants) | 1003 | 3022 | 4025
  ACR20 at Month 9 | 76.57 | 77.53 | 77.29
  ACR20 at Month 12: number analyzed (Participants) | 972 | 2891 | 3863
  ACR20 at Month 12 | 77.88 | 78.24 | 78.15
  ACR20 at Month 15: number analyzed (Participants) | 938 | 2775 | 3713
  ACR20 at Month 15 | 76.76 | 78.67 | 78.18
  ACR20 at Month 18: number analyzed (Participants) | 910 | 2665 | 3575
  ACR20 at Month 18 | 77.91 | 78.46 | 78.32
  ACR20 at Month 21: number analyzed (Participants) | 860 | 2565 | 3425
  ACR20 at Month 21 | 77.91 | 79.42 | 79.04
  ACR20 at Month 24: number analyzed (Participants) | 824 | 2464 | 3288
  ACR20 at Month 24 | 79.61 | 78.37 | 78.68
  ACR20 at Month 27: number analyzed (Participants) | 796 | 2361 | 3157
  ACR20 at Month 27 | 79.15 | 79.16 | 79.16
  ACR20 at Month 30: number analyzed (Participants) | 770 | 2288 | 3058
  ACR20 at Month 30 | 80.00 | 79.90 | 79.92
  ACR20 at Month 33: number analyzed (Participants) | 749 | 2219 | 2968
  ACR20 at Month 33 | 80.51 | 79.81 | 79.99
  ACR20 at Month 36: number analyzed (Participants) | 730 | 2157 | 2887
  ACR20 at Month 36 | 81.78 | 79.37 | 79.98
  ACR20 at Month 39: number analyzed (Participants) | 690 | 2073 | 2763
  ACR20 at Month 39 | 78.55 | 81.23 | 80.56
  ACR20 at Month 42: number analyzed (Participants) | 657 | 1907 | 2564
  ACR20 at Month 42 | 78.69 | 80.49 | 80.03
  ACR20 at Month 45: number analyzed (Participants) | 616 | 1658 | 2274
  ACR20 at Month 45 | 82.14 | 79.55 | 80.26
  ACR20 at Month 48: number analyzed (Participants) | 581 | 1486 | 2067
  ACR20 at Month 48 | 78.31 | 80.69 | 80.02
  ACR20 at Month 51: number analyzed (Participants) | 490 | 1355 | 1845
  ACR20 at Month 51 | 83.47 | 80.30 | 81.14
  ACR20 at Month 54: number analyzed (Participants) | 471 | 1208 | 1679
  ACR20 at Month 54 | 79.19 | 78.97 | 79.04
  ACR20 at Month 57: number analyzed (Participants) | 441 | 1021 | 1462
  ACR20 at Month 57 | 80.73 | 82.37 | 81.87
  ACR20 at Month 60: number analyzed (Participants) | 411 | 920 | 1331
  ACR20 at Month 60 | 81.75 | 82.39 | 82.19
  ACR20 at Month 63: number analyzed (Participants) | 396 | 692 | 1230
  ACR20 at Month 63 | 80.30 | 82.97 | 82.11
  ACR20 at Month 66: number analyzed (Participants) | 382 | 705 | 1087
  ACR20 at Month 66 | 79.84 | 81.42 | 80.86
  ACR20 at Month 69: number analyzed (Participants) | 358 | 486 | 844
  ACR20 at Month 69 | 82.68 | 83.54 | 83.18
  ACR20 at Month 72: number analyzed (Participants) | 339 | 287 | 626
  ACR20 at Month 72 | 82.01 | 82.58 | 82.27
  ACR20 at Month 75: number analyzed (Participants) | 309 | 171 | 480
  ACR20 at Month 75 | 82.20 | 78.95 | 81.04
  ACR20 at Month 78: number analyzed (Participants) | 295 | 91 | 386
  ACR20 at Month 78 | 81.69 | 80.22 | 81.35
  ACR20 at Month 81: number analyzed (Participants) | 286 | 54 | 340
  ACR20 at Month 81 | 82.52 | 79.63 | 82.06
  ACR20 at Month 84: number analyzed (Participants) | 271 | 44 | 315
  ACR20 at Month 84 | 82.66 | 81.82 | 82.54
  ACR20 at Month 87: number analyzed (Participants) | 264 | 41 | 305
  ACR20 at Month 87 | 84.47 | 70.73 | 82.62
  ACR20 at Month 90: number analyzed (Participants) | 241 | 39 | 280
  ACR20 at Month 90 | 82.57 | 74.36 | 81.43
  ACR20 at Month 93: number analyzed (Participants) | 196 | 28 | 224
  ACR20 at Month 93 | 82.14 | 78.57 | 81.70
  ACR20 at Month 96: number analyzed (Participants) | 144 | 16 | 160
  ACR20 at Month 96 | 78.47 | 81.25 | 78.75
  ACR20 at Month 99: number analyzed (Participants) | 65 | 11 | 76
  ACR20 at Month 99 | 83.08 | 90.91 | 84.21
  ACR20 at Month 102: number analyzed (Participants) | 22 | 4 | 26
  ACR20 at Month 102 | 77.27 | 50.00 | 73.08
  ACR20 at Month 105: number analyzed (Participants) | 15 | 3 | 18
  ACR20 at Month 105 | 73.33 | 66.67 | 72.22
  ACR20 at Month 108: number analyzed (Participants) | 8 | 1 | 9
  ACR20 at Month 108 | 62.50 | 100.00 | 66.67
  ACR20 at Month 111: number analyzed (Participants) | 3 | 1 | 4
  ACR20 at Month 111 | 100.00 | 100.00 | 100.00
  ACR20 at Month 114: number analyzed (Participants) | 1 | 0 | 1
  ACR20 at Month 114 | 100.00 |  | 100.00
  ACR50 at Month 1: number analyzed (Participants) | 1114 | 3307 | 4421
  ACR50 at Month 1 | 47.67 | 49.56 | 49.08
  ACR50 at Month 2: number analyzed (Participants) | 1080 | 3254 | 4334
  ACR50 at Month 2 | 50.19 | 53.29 | 52.51
  ACR50 at Month 3: number analyzed (Participants) | 1069 | 3228 | 4297
  ACR50 at Month 3 | 51.45 | 54.52 | 53.76
  ACR50 at Month 6: number analyzed (Participants) | 1040 | 3132 | 4172
  ACR50 at Month 6 | 52.79 | 55.75 | 55.01
  ACR50 at Month 9: number analyzed (Participants) | 1003 | 3022 | 4025
  ACR50 at Month 9 | 53.24 | 55.96 | 55.28
  ACR50 at Month 12: number analyzed (Participants) | 972 | 2891 | 3863
  ACR50 at Month 12 | 52.98 | 56.73 | 55.79
  ACR50 at Month 15: number analyzed (Participants) | 938 | 2775 | 3713
  ACR50 at Month 15 | 55.76 | 56.61 | 56.40
  ACR50 at Month 18: number analyzed (Participants) | 910 | 2665 | 3575
  ACR50 at Month 18 | 55.16 | 57.30 | 56.76
  ACR50 at Month 21: number analyzed (Participants) | 860 | 2565 | 3425
  ACR50 at Month 21 | 54.77 | 59.10 | 58.01
  ACR50 at Month 24: number analyzed (Participants) | 824 | 2464 | 3288
  ACR50 at Month 24 | 57.77 | 57.67 | 57.69
  ACR50 at Month 27: number analyzed (Participants) | 796 | 2361 | 3157
  ACR50 at Month 27 | 56.91 | 58.58 | 58.16
  ACR50 at Month 30: number analyzed (Participants) | 770 | 2288 | 3058
  ACR50 at Month 30 | 58.83 | 58.65 | 58.70
  ACR50 at Month 33: number analyzed (Participants) | 749 | 2219 | 2968
  ACR50 at Month 33 | 57.68 | 59.31 | 58.89
  ACR50 at Month 36: number analyzed (Participants) | 730 | 2157 | 2887
  ACR50 at Month 36 | 58.49 | 58.51 | 58.50
  ACR50 at Month 39: number analyzed (Participants) | 690 | 2073 | 2763
  ACR50 at Month 39 | 59.28 | 59.29 | 59.28
  ACR50 at Month 42: number analyzed (Participants) | 657 | 1907 | 2564
  ACR50 at Month 42 | 58.60 | 59.99 | 59.63
  ACR50 at Month 45: number analyzed (Participants) | 616 | 1658 | 2274
  ACR50 at Month 45 | 59.42 | 60.07 | 59.89
  ACR50 at Month 48: number analyzed (Participants) | 581 | 1486 | 2067
  ACR50 at Month 48 | 58.00 | 57.60 | 57.72
  ACR50 at Month 51: number analyzed (Participants) | 490 | 1355 | 1845
  ACR50 at Month 51 | 62.45 | 59.19 | 60.05
  ACR50 at Month 54: number analyzed (Participants) | 471 | 1208 | 1679
  ACR50 at Month 54 | 58.60 | 59.44 | 59.20
  ACR50 at Month 57: number analyzed (Participants) | 441 | 1021 | 1462
  ACR50 at Month 57 | 61.45 | 61.12 | 61.22
  ACR50 at Month 60: number analyzed (Participants) | 411 | 920 | 1331
  ACR50 at Month 60 | 62.53 | 60.65 | 61.23
  ACR50 at Month 63: number analyzed (Participants) | 396 | 834 | 1230
  ACR50 at Month 63 | 64.39 | 61.99 | 62.76
  ACR50 at Month 66: number analyzed (Participants) | 382 | 705 | 1087
  ACR50 at Month 66 | 60.73 | 60.85 | 60.81
  ACR50 at Month 69: number analyzed (Participants) | 358 | 486 | 844
  ACR50 at Month 69 | 58.10 | 61.11 | 59.83
  ACR50 at Month 72: number analyzed (Participants) | 339 | 287 | 626
  ACR50 at Month 72 | 62.54 | 59.93 | 61.34
  ACR50 at Month 75: number analyzed (Participants) | 309 | 171 | 480
  ACR50 at Month 75 | 61.49 | 56.14 | 59.58
  ACR50 at Month 78: number analyzed (Participants) | 295 | 91 | 386
  ACR50 at Month 78 | 60.00 | 58.24 | 59.59
  ACR50 at Month 81: number analyzed (Participants) | 286 | 54 | 340
  ACR50 at Month 81 | 63.99 | 51.85 | 62.06
  ACR50 at Month 84: number analyzed (Participants) | 271 | 44 | 315
  ACR50 at Month 84 | 63.10 | 54.55 | 61.90
  ACR50 at Month 87: number analyzed (Participants) | 264 | 41 | 305
  ACR50 at Month 87 | 67.05 | 43.90 | 63.93
  ACR50 at Month 90: number analyzed (Participants) | 241 | 39 | 280
  ACR50 at Month 90 | 61.00 | 46.15 | 58.93
  ACR50 at Month 93: number analyzed (Participants) | 196 | 28 | 224
  ACR50 at Month 93 | 61.22 | 57.14 | 60.71
  ACR50 at Month 96: number analyzed (Participants) | 144 | 16 | 160
  ACR50 at Month 96 | 61.11 | 56.25 | 60.63
  ACR50 at Month 99: number analyzed (Participants) | 65 | 11 | 76
  ACR50 at Month 99 | 53.85 | 54.55 | 53.95
  ACR50 at Month 102: number analyzed (Participants) | 22 | 4 | 26
  ACR50 at Month 102 | 54.55 | 25.00 | 50.00
  ACR50 at Month 105: number analyzed (Participants) | 15 | 3 | 18
  ACR50 at Month 105 | 66.67 | 33.33 | 61.11
  ACR50 at Month 108: number analyzed (Participants) | 8 | 1 | 9
  ACR50 at Month 108 | 50.00 | 0.00 | 44.44
  ACR50 at Month 111: number analyzed (Participants) | 3 | 1 | 4
  ACR50 at Month 111 | 100.00 | 0.00 | 75.00
  ACR50 at Month 114: number analyzed (Participants) | 1 | 0 | 1
  ACR50 at Month 114 | 100.00 |  | 100.00
  ACR70 at Month 1: number analyzed (Participants) | 1114 | 3307 | 4421
  ACR70 at Month 1 | 26.66 | 28.82 | 28.27
  ACR70 at Month 2: number analyzed (Participants) | 1080 | 3254 | 4334
  ACR70 at Month 2 | 27.78 | 31.53 | 30.60
  ACR70 at Month 3: number analyzed (Participants) | 1069 | 3228 | 4297
  ACR70 at Month 3 | 29.37 | 33.09 | 32.16
  ACR70 at Month 6: number analyzed (Participants) | 1040 | 3132 | 4172
  ACR70 at Month 6 | 31.06 | 33.75 | 33.08
  ACR70 at Month 9: number analyzed (Participants) | 1003 | 3022 | 4025
  ACR70 at Month 9 | 31.80 | 34.91 | 34.14
  ACR70 at Month 12: number analyzed (Participants) | 972 | 2891 | 3863
  ACR70 at Month 12 | 31.38 | 35.84 | 34.71
  ACR70 at Month 15: number analyzed (Participants) | 938 | 2775 | 3713
  ACR70 at Month 15 | 32.94 | 36.54 | 35.63
  ACR70 at Month 18: number analyzed (Participants) | 910 | 2665 | 3575
  ACR70 at Month 18 | 35.82 | 36.40 | 36.25
  ACR70 at Month 21: number analyzed (Participants) | 860 | 2565 | 3425
  ACR70 at Month 21 | 33.49 | 37.66 | 36.61
  ACR70 at Month 24: number analyzed (Participants) | 824 | 2464 | 3288
  ACR70 at Month 24 | 35.44 | 38.15 | 37.47
  ACR70 at Month 27: number analyzed (Participants) | 796 | 2361 | 3157
  ACR70 at Month 27 | 36.06 | 38.33 | 37.76
  ACR70 at Month 30: number analyzed (Participants) | 770 | 2288 | 3058
  ACR70 at Month 30 | 37.27 | 38.99 | 38.55
  ACR70 at Month 33: number analyzed (Participants) | 749 | 2219 | 2968
  ACR70 at Month 33 | 33.64 | 38.26 | 37.10
  ACR70 at Month 36: number analyzed (Participants) | 730 | 2157 | 2887
  ACR70 at Month 36 | 36.71 | 37.41 | 37.24
  ACR70 at Month 39: number analyzed (Participants) | 690 | 2073 | 2763
  ACR70 at Month 39 | 38.41 | 38.88 | 38.76
  ACR70 at Month 42: number analyzed (Participants) | 657 | 1907 | 2564
  ACR70 at Month 42 | 35.77 | 38.91 | 38.10
  ACR70 at Month 45: number analyzed (Participants) | 616 | 1658 | 2274
  ACR70 at Month 45 | 36.69 | 38.18 | 37.77
  ACR70 at Month 48: number analyzed (Participants) | 581 | 1486 | 2067
  ACR70 at Month 48 | 35.97 | 37.01 | 36.72
  ACR70 at Month 51: number analyzed (Participants) | 490 | 1355 | 1845
  ACR70 at Month 51 | 39.59 | 37.34 | 37.94
  ACR70 at Month 54: number analyzed (Participants) | 471 | 1208 | 1679
  ACR70 at Month 54 | 36.73 | 39.32 | 38.59
  ACR70 at Month 57: number analyzed (Participants) | 441 | 1021 | 1462
  ACR70 at Month 57 | 38.78 | 39.47 | 39.26
  ACR70 at Month 60: number analyzed (Participants) | 411 | 920 | 1331
  ACR70 at Month 60 | 37.96 | 38.91 | 38.62
  ACR70 at Month 63: number analyzed (Participants) | 396 | 834 | 1230
  ACR70 at Month 63 | 38.64 | 39.33 | 39.11
  ACR70 at Month 66: number analyzed (Participants) | 382 | 705 | 1087
  ACR70 at Month 66 | 38.22 | 40.14 | 39.47
  ACR70 at Month 69: number analyzed (Participants) | 358 | 486 | 844
  ACR70 at Month 69 | 38.55 | 41.56 | 40.28
  ACR70 at Month 72: number analyzed (Participants) | 339 | 287 | 626
  ACR70 at Month 72 | 40.12 | 36.59 | 38.50
  ACR70 at Month 75: number analyzed (Participants) | 309 | 171 | 480
  ACR70 at Month 75 | 40.13 | 36.84 | 38.96
  ACR70 at Month 78: number analyzed (Participants) | 295 | 91 | 386
  ACR70 at Month 78 | 42.37 | 32.97 | 40.16
  ACR70 at Month 81: number analyzed (Participants) | 286 | 54 | 340
  ACR70 at Month 81 | 41.26 | 35.19 | 40.29
  ACR70 at Month 84: number analyzed (Participants) | 271 | 44 | 315
  ACR70 at Month 84 | 42.07 | 31.82 | 40.63
  ACR70 at Month 87: number analyzed (Participants) | 264 | 41 | 305
  ACR70 at Month 87 | 42.80 | 21.95 | 40.00
  ACR70 at Month 90: number analyzed (Participants) | 241 | 39 | 280
  ACR70 at Month 90 | 38.17 | 25.64 | 36.43
  ACR70 at Month 93: number analyzed (Participants) | 196 | 28 | 224
  ACR70 at Month 93 | 41.84 | 39.29 | 41.52
  ACR70 at Month 96: number analyzed (Participants) | 144 | 16 | 160
  ACR70 at Month 96 | 43.75 | 31.25 | 42.50
  ACR70 at Month 99: number analyzed (Participants) | 65 | 11 | 76
  ACR70 at Month 99 | 40.00 | 18.18 | 36.84
  ACR70 at Month 102: number analyzed (Participants) | 22 | 4 | 26
  ACR70 at Month 102 | 40.91 | 25.00 | 38.46
  ACR70 at Month 105: number analyzed (Participants) | 15 | 3 | 18
  ACR70 at Month 105 | 46.67 | 33.33 | 44.44
  ACR70 at Month 108: number analyzed (Participants) | 8 | 1 | 9
  ACR70 at Month 108 | 25.00 | 0.00 | 22.22
  ACR70 at Month 111: number analyzed (Participants) | 3 | 1 | 4
  ACR70 at Month 111 | 100.00 | 0.00 | 75.00
  ACR70 at Month 114: number analyzed (Participants) | 1 | 0 | 1
  ACR70 at Month 114 | 100.00 |  | 100.00

7. Secondary Outcome: Extension Period: Percentage of Participants With American College of Rheumatology (ACR) 20, 50, and 70 Responses
Description: ACR20=20 percent (%) improvement from baseline (Month 0 at entry of Initial Period) in tender/painful joint count and swollen joint count, and in at least 3 of 5 variables: participant's global assessment of arthritis (PtGA), physician's global assessment of arthritis (PGA), participant's assessment of arthritis pain (PtA), HAQ-DI, C-reactive protein. ACR50 is a 50% improvement and ACR70 is a 70% improvement in these variables. PtGA: participant assessed overall disease activity, score: 0 (no arthritis) to 10 (extreme arthritis), higher score=more arthritis. PGA: physician judged participant's overall disease activity, score: 0 (no arthritis) to 10 (extreme arthritis), higher score=more arthritis. PtA: participant assessed arthritis pain by 100 millimeter (mm) visual analogue scale, score: 0 mm (no pain) to 100 mm (extreme pain), higher score=more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score=more disability.
Time Frame: Month 3, 6, 9 and 12 of Extension Period
Population: Full analysis set included all participants who enrolled for extension period and received at least 1 dose of open label study medication in extension period. Here, "Number Analyzed" signifies number of participants who were evaluable for specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Extension Period: Tofacitinib 5 mg
Number analyzed (Participants) | 48
Percentage of participants
  ACR20 at Month 3: number analyzed (Participants) | 47
  ACR20 at Month 3 | 70.21
  ACR20 at Month 6: number analyzed (Participants) | 36
  ACR20 at Month 6 | 66.67
  ACR20 at Month 9: number analyzed (Participants) | 15
  ACR20 at Month 9 | 86.67
  ACR20 at Month 12: number analyzed (Participants) | 2
  ACR20 at Month 12 | 50.00
  ACR50 at Month 3: number analyzed (Participants) | 47
  ACR50 at Month 3 | 48.94
  ACR50 at Month 6: number analyzed (Participants) | 36
  ACR50 at Month 6 | 55.56
  ACR50 at Month 9: number analyzed (Participants) | 15
  ACR50 at Month 9 | 60.00
  ACR50 at Month 12: number analyzed (Participants) | 2
  ACR50 at Month 12 | 50.00
  ACR70 at Month 3: number analyzed (Participants) | 47
  ACR70 at Month 3 | 23.40
  ACR70 at Month 6: number analyzed (Participants) | 36
  ACR70 at Month 6 | 36.11
  ACR70 at Month 9: number analyzed (Participants) | 15
  ACR70 at Month 9 | 40.00
  ACR70 at Month 12: number analyzed (Participants) | 2
  ACR70 at Month 12 | 50.00

8. Secondary Outcome: Initial Period: Area Under American College of Rheumatology (ACR) n Curve
Description: No data were collected for this endpoint because it was removed from the protocol in a previous amendment.
Time Frame: Not applicable as no data were collected for this endpoint.
Population: No data were collected for this endpoint as it was removed from the protocol in a protocol amendment.
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Initial Period: Disease Activity Score (DAS)28 (C-reactive Protein [CRP]) and DAS28 (Erythrocyte Sedimentation Rate [ESR])
Description: Descriptive statistics for DAS28-3 (CRP) and DAS28-4 (ESR). The stated number of participants analyzed was the total number of participants in each group. The actual number of participants analyzed on each occasion varied, and is provided for each visit presented.
  DAS28 is a composite score, calculated using a mathematical formula, and is derived from the number of tender/painful joints (out of 28), number of swollen joints (out of 28), and a blood marker of inflammation (ESR or CRP). DAS28-4 also includes a score of general health in the formula.
  The score range is from 0 to 9.4, with a higher score indicating more disease activity. A score of >5.1 indicates active disease, a score of ≤3.2 indicates low disease activity, and a score of <2.6 indicates disease remission.
Time Frame: Every visit until study completion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score calculated from formula
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib
Number analyzed (Participants) | 1123 | 3358 | 4481
Score calculated from formula
  DAS28-4 (ESR) Baseline: number analyzed (Participants) | 1002 | 3296 | 4298
  DAS28-4 (ESR) Baseline | 6.27 (1.02) | 6.39 (1.04) | 6.36 (1.04)
  DAS28-4 (ESR) Month 1: number analyzed (Participants) | 1036 | 3254 | 4290
  DAS28-4 (ESR) Month 1 | 3.81 (1.32) | 3.78 (1.36) | 3.79 (1.35)
  DAS28-4 (ESR) Month 2: number analyzed (Participants) | 1026 | 3222 | 4248
  DAS28-4 (ESR) Month 2 | 3.72 (1.27) | 3.66 (1.32) | 3.68 (1.31)
  DAS28-4 (ESR) Month 3: number analyzed (Participants) | 1033 | 3203 | 4236
  DAS28-4 (ESR) Month 3 | 3.75 (1.32) | 3.61 (1.30) | 3.65 (1.31)
  DAS28-4 (ESR) Month 6: number analyzed (Participants) | 1015 | 3110 | 4125
  DAS28-4 (ESR) Month 6 | 3.67 (1.33) | 3.61 (1.30) | 3.62 (1.31)
  DAS28-4 (ESR) Month 9: number analyzed (Participants) | 992 | 3003 | 3995
  DAS28-4 (ESR) Month 9 | 3.60 (1.31) | 3.58 (1.32) | 3.59 (1.31)
  DAS28-4 (ESR) Month 12: number analyzed (Participants) | 967 | 2862 | 3829
  DAS28-4 (ESR) Month 12 | 3.61 (1.26) | 3.56 (1.30) | 3.57 (1.29)
  DAS28-4 (ESR) Month 15: number analyzed (Participants) | 922 | 2759 | 3681
  DAS28-4 (ESR) Month 15 | 3.54 (1.26) | 3.53 (1.30) | 3.53 (1.29)
  DAS28-4 (ESR) Month 18: number analyzed (Participants) | 899 | 2655 | 3554
  DAS28-4 (ESR) Month 18 | 3.57 (1.26) | 3.50 (1.28) | 3.52 (1.28)
  DAS28-4 (ESR) Month 21: number analyzed (Participants) | 850 | 2547 | 3397
  DAS28-4 (ESR) Month 21 | 3.58 (1.25) | 3.45 (1.27) | 3.48 (1.26)
  DAS28-4 (ESR) Month 24: number analyzed (Participants) | 818 | 2441 | 3259
  DAS28-4 (ESR) Month 24 | 3.54 (1.21) | 3.46 (1.26) | 3.48 (1.25)
  DAS28-4 (ESR) Month 27: number analyzed (Participants) | 787 | 2343 | 3130
  DAS28-4 (ESR) Month 27 | 3.52 (1.20) | 3.44 (1.25) | 3.46 (1.24)
  DAS28-4 (ESR) Month 30: number analyzed (Participants) | 764 | 2257 | 3021
  DAS28-4 (ESR) Month 30 | 3.54 (1.23) | 3.43 (1.25) | 3.46 (1.24)
  DAS28-4 (ESR) Month 33: number analyzed (Participants) | 746 | 2199 | 2945
  DAS28-4 (ESR) Month 33 | 3.51 (1.22) | 3.42 (1.27) | 3.45 (1.26)
  DAS28-4 (ESR) Month 36: number analyzed (Participants) | 720 | 2141 | 2861
  DAS28-4 (ESR) Month 36 | 3.51 (1.23) | 3.42 (1.27) | 3.44 (1.26)
  DAS28-4 (ESR) Month 39: number analyzed (Participants) | 679 | 2056 | 2735
  DAS28-4 (ESR) Month 39 | 3.56 (1.27) | 3.39 (1.24) | 3.43 (1.25)
  DAS28-4 (ESR) Month 42: number analyzed (Participants) | 642 | 1890 | 2532
  DAS28-4 (ESR) Month 42 | 3.53 (1.26) | 3.40 (1.26) | 3.43 (1.26)
  DAS28-4 (ESR) Month 45: number analyzed (Participants) | 609 | 1641 | 2250
  DAS28-4 (ESR) Month 45 | 3.45 (1.20) | 3.37 (1.21) | 3.39 (1.20)
  DAS28-4 (ESR) Month 48: number analyzed (Participants) | 570 | 1471 | 2041
  DAS28-4 (ESR) Month 48 | 3.46 (1.16) | 3.36 (1.21) | 3.39 (1.20)
  DAS28-4 (ESR) Month 51: number analyzed (Participants) | 481 | 1344 | 1825
  DAS28-4 (ESR) Month 51 | 3.43 (1.20) | 3.39 (1.24) | 3.40 (1.23)
  DAS28-4 (ESR) Month 54: number analyzed (Participants) | 467 | 1194 | 1661
  DAS28-4 (ESR) Month 54 | 3.54 (1.23) | 3.38 (1.25) | 3.42 (1.25)
  DAS28-4 (ESR) Month 57: number analyzed (Participants) | 438 | 1006 | 1444
  DAS28-4 (ESR) Month 57 | 3.48 (1.19) | 3.36 (1.21) | 3.40 (1.20)
  DAS28-4 (ESR) Month 60: number analyzed (Participants) | 408 | 908 | 1316
  DAS28-4 (ESR) Month 60 | 3.51 (1.27) | 3.34 (1.20) | 3.39 (1.22)
  DAS28-4 (ESR) Month 63: number analyzed (Participants) | 388 | 825 | 1213
  DAS28-4 (ESR) Month 63 | 3.51 (1.15) | 3.30 (1.16) | 3.37 (1.16)
  DAS28-4 (ESR) Month 66: number analyzed (Participants) | 379 | 700 | 1079
  DAS28-4 (ESR) Month 66 | 3.58 (1.12) | 3.34 (1.17) | 3.42 (1.15)
  DAS28-4 (ESR) Month 69: number analyzed (Participants) | 355 | 483 | 838
  DAS28-4 (ESR) Month 69 | 3.51 (1.18) | 3.35 (1.20) | 3.41 (1.19)
  DAS28-4 (ESR) Month 72: number analyzed (Participants) | 338 | 284 | 622
  DAS28-4 (ESR) Month 72 | 3.45 (1.20) | 3.42 (1.19) | 3.44 (1.20)
  DAS28-4 (ESR) Month 75: number analyzed (Participants) | 299 | 169 | 468
  DAS28-4 (ESR) Month 75 | 3.43 (1.11) | 3.41 (1.14) | 3.43 (1.12)
  DAS28-4 (ESR) Month 78: number analyzed (Participants) | 291 | 91 | 382
  DAS28-4 (ESR) Month 78 | 3.44 (1.14) | 3.32 (1.20) | 3.41 (1.16)
  DAS28-4 (ESR) Month 81: number analyzed (Participants) | 284 | 54 | 338
  DAS28-4 (ESR) Month 81 | 3.40 (1.11) | 3.56 (1.24) | 3.42 (1.13)
  DAS28-4 (ESR) Month 84: number analyzed (Participants) | 271 | 44 | 315
  DAS28-4 (ESR) Month 84 | 3.32 (1.13) | 3.42 (1.37) | 3.34 (1.16)
  DAS28-4 (ESR) Month 87: number analyzed (Participants) | 263 | 41 | 304
  DAS28-4 (ESR) Month 87 | 3.33 (1.13) | 3.19 (1.15) | 3.31 (1.13)
  DAS28-4 (ESR) Month 90: number analyzed (Participants) | 237 | 39 | 276
  DAS28-4 (ESR) Month 90 | 3.34 (1.14) | 3.28 (1.10) | 3.33 (1.13)
  DAS28-4 (ESR) Month 93: number analyzed (Participants) | 191 | 28 | 219
  DAS28-4 (ESR) Month 93 | 3.33 (1.14) | 3.23 (1.12) | 3.32 (1.13)
  DAS28-4 (ESR) Month 96: number analyzed (Participants) | 142 | 16 | 158
  DAS28-4 (ESR) Month 96 | 3.30 (1.12) | 3.48 (1.06) | 3.32 (1.11)
  DAS28-4 (ESR) Month 99: number analyzed (Participants) | 65 | 11 | 76
  DAS28-4 (ESR) Month 99 | 3.26 (1.07) | 3.04 (1.24) | 3.23 (1.09)
  DAS28-4 (ESR) Month 102: number analyzed (Participants) | 22 | 4 | 26
  DAS28-4 (ESR) Month 102 | 3.34 (1.47) | 3.10 (1.76) | 3.30 (1.48)
  DAS28-4 (ESR) Month 105: number analyzed (Participants) | 14 | 3 | 17
  DAS28-4 (ESR) Month 105 | 3.64 (1.52) | 2.65 (0.97) | 3.46 (1.46)
  DAS28-4 (ESR) Month 108: number analyzed (Participants) | 8 | 1 | 9
  DAS28-4 (ESR) Month 108 | 3.36 (1.76) | 4.65 (0) | 3.51 (1.70)
  DAS28-4 (ESR) Month 111: number analyzed (Participants) | 3 | 1 | 4
  DAS28-4 (ESR) Month 111 | 2.03 (0.69) | 3.59 (0) | 2.42 (0.96)
  DAS28-4 (ESR) Month 114: number analyzed (Participants) | 1 | 0 | 1
  DAS28-4 (ESR) Month 114 | 1.28 (0) |  | 1.28 (0)
  DAS28-3 (CRP) Baseline: number analyzed (Participants) | 1112 | 3340 | 4452
  DAS28-3 (CRP) Baseline | 5.31 (0.95) | 5.34 (0.98) | 5.33 (0.97)
  DAS28-3 (CRP) Month 1: number analyzed (Participants) | 1096 | 3234 | 4330
  DAS28-3 (CRP) Month 1 | 3.10 (1.19) | 2.96 (1.22) | 2.99 (1.21)
  DAS28-3 (CRP) Month 2: number analyzed (Participants) | 1070 | 3180 | 4250
  DAS28-3 (CRP) Month 2 | 3.01 (1.15) | 2.87 (1.17) | 2.90 (1.17)
  DAS28-3 (CRP) Month 3: number analyzed (Participants) | 1057 | 3190 | 4247
  DAS28-3 (CRP) Month 3 | 2.98 (1.15) | 2.81 (1.15) | 2.85 (1.15)
  DAS28-3 (CRP) Month 6: number analyzed (Participants) | 1026 | 3106 | 4132
  DAS28-3 (CRP) Month 6 | 2.89 (1.16) | 2.79 (1.15) | 2.81 (1.16)
  DAS28-3 (CRP) Month 9: number analyzed (Participants) | 993 | 3008 | 4001
  DAS28-3 (CRP) Month 9 | 2.82 (1.12) | 2.74 (1.16) | 2.76 (1.15)
  DAS28-3 (CRP) Month 12: number analyzed (Participants) | 962 | 2874 | 3836
  DAS28-3 (CRP) Month 12 | 2.81 (1.11) | 2.72 (1.13) | 2.74 (1.13)
  DAS28-3 (CRP) Month 15: number analyzed (Participants) | 923 | 2761 | 3684
  DAS28-3 (CRP) Month 15 | 2.73 (1.10) | 2.69 (1.13) | 2.70 (1.12)
  DAS28-3 (CRP) Month 18: number analyzed (Participants) | 899 | 2654 | 3553
  DAS28-3 (CRP) Month 18 | 2.72 (1.11) | 2.66 (1.11) | 2.68 (1.11)
  DAS28-3 (CRP) Month 21: number analyzed (Participants) | 856 | 2556 | 3412
  DAS28-3 (CRP) Month 21 | 2.75 (1.12) | 2.62 (1.09) | 2.65 (1.09)
  DAS28-3 (CRP) Month 24: number analyzed (Participants) | 813 | 2456 | 3269
  DAS28-3 (CRP) Month 24 | 2.96 (1.07) | 2.63 (1.11) | 2.64 (1.10)
  DAS28-3 (CRP) Month 27: number analyzed (Participants) | 793 | 2345 | 3138
  DAS28-3 (CRP) Month 27 | 2.66 (1.06) | 2.60 (1.09) | 2.62 (1.08)
  DAS28-3 (CRP) Month 30: number analyzed (Participants) | 766 | 2271 | 3037
  DAS28-3 (CRP) Month 30 | 2.65 (1.07) | 2.59 (1.09) | 2.60 (1.08)
  DAS28-3 (CRP) Month 33: number analyzed (Participants) | 745 | 2209 | 2954
  DAS28-3 (CRP) Month 33 | 2.64 (1.06) | 2.58 (1.10) | 2.60 (1.09)
  DAS28-3 (CRP) Month 36: number analyzed (Participants) | 724 | 2142 | 2866
  DAS28-3 (CRP) Month 36 | 2.64 (1.07) | 2.59 (1.08) | 2.60 (1.08)
  DAS28-3 (CRP) Month 39: number analyzed (Participants) | 686 | 2057 | 2743
  DAS28-3 (CRP) Month 39 | 2.65 (1.10) | 2.57 (1.07) | 2.59 (1.08)
  DAS28-3 (CRP) Month 42: number analyzed (Participants) | 653 | 1893 | 2546
  DAS28-3 (CRP) Month 42 | 2.63 (1.09) | 2.57 (1.09) | 2.59 (1.09)
  DAS28-3 (CRP) Month 45: number analyzed (Participants) | 611 | 1644 | 2255
  DAS28-3 (CRP) Month 45 | 2.57 (1.04) | 2.53 (1.03) | 2.54 (1.03)
  DAS28-3 (CRP) Month 48: number analyzed (Participants) | 579 | 1469 | 2048
  DAS28-3 (CRP) Month 48 | 2.59 (1.03) | 2.54 (1.05) | 2.56 (1.04)
  DAS28-3 (CRP) Month 51: number analyzed (Participants) | 487 | 1348 | 1835
  DAS28-3 (CRP) Month 51 | 2.59 (0.99) | 2.57 (1.07) | 2.57 (1.05)
  DAS28-3 (CRP) Month 54: number analyzed (Participants) | 468 | 1198 | 1666
  DAS28-3 (CRP) Month 54 | 2.68 (1.07) | 2.56 (1.05) | 2.59 (1.06)
  DAS28-3 (CRP) Month 57: number analyzed (Participants) | 439 | 1011 | 1450
  DAS28-3 (CRP) Month 57 | 2.63 (1.03) | 2.54 (1.04) | 2.56 (1.03)
  DAS28-3 (CRP) Month 60: number analyzed (Participants) | 407 | 913 | 1320
  DAS28-3 (CRP) Month 60 | 2.66 (1.09) | 2.53 (1.03) | 2.57 (1.05)
  DAS28-3 (CRP) Month 63: number analyzed (Participants) | 390 | 824 | 1214
  DAS28-3 (CRP) Month 63 | 2.67 (1.01) | 2.51 (0.98) | 2.56 (0.99)
  DAS28-3 (CRP) Month 66: number analyzed (Participants) | 376 | 702 | 1078
  DAS28-3 (CRP) Month 66 | 2.70 (1.02) | 2.53 (1.01) | 2.59 (1.02)
  DAS28-3 (CRP) Month 69: number analyzed (Participants) | 355 | 483 | 838
  DAS28-3 (CRP) Month 69 | 2.67 (1.06) | 2.55 (1.00) | 2.60 (1.03)
  DAS28-3 (CRP) Month 72: number analyzed (Participants) | 337 | 285 | 622
  DAS28-3 (CRP) Month 72 | 2.65 (1.04) | 2.64 (1.03) | 2.64 (1.04)
  DAS28-3 (CRP) Month 75: number analyzed (Participants) | 304 | 170 | 474
  DAS28-3 (CRP) Month 75 | 2.63 (1.05) | 2.59 (1.02) | 2.61 (1.04)
  DAS28-3 (CRP) Month 78: number analyzed (Participants) | 292 | 91 | 383
  DAS28-3 (CRP) Month 78 | 2.59 (1.02) | 2.68 (1.01) | 2.61 (1.02)
  DAS28-3 (CRP) Month 81: number analyzed (Participants) | 285 | 54 | 339
  DAS28-3 (CRP) Month 81 | 2.54 (0.96) | 2.82 (1.13) | 2.59 (0.99)
  DAS28-3 (CRP) Month 84: number analyzed (Participants) | 269 | 44 | 313
  DAS28-3 (CRP) Month 84 | 2.49 (0.94) | 2.84 (1.20) | 2.54 (0.99)
  DAS28-3 (CRP) Month 87: number analyzed (Participants) | 264 | 41 | 305
  DAS28-3 (CRP) Month 87 | 2.52 (0.97) | 2.56 (0.91) | 2.52 (0.96)
  DAS28-3 (CRP) Month 90: number analyzed (Participants) | 240 | 39 | 279
  DAS28-3 (CRP) Month 90 | 2.55 (1.00) | 2.58 (0.95) | 2.55 (0.99)
  DAS28-3 (CRP) Month 93: number analyzed (Participants) | 196 | 28 | 224
  DAS28-3 (CRP) Month 93 | 2.59 (1.00) | 2.59 (0.85) | 2.59 (0.98)
  DAS28-3 (CRP) Month 96: number analyzed (Participants) | 144 | 16 | 160
  DAS28-3 (CRP) Month 96 | 2.59 (0.93) | 2.68 (0.80) | 2.60 (0.92)
  DAS28-3 (CRP) Month 99: number analyzed (Participants) | 64 | 11 | 75
  DAS28-3 (CRP) Month 99 | 2.58 (0.89) | 2.49 (1.12) | 2.57 (0.92)
  DAS28-3 (CRP) Month 102: number analyzed (Participants) | 13 | 3 | 16
  DAS28-3 (CRP) Month 102 | 2.66 (0.78) | 2.29 (1.01) | 2.59 (0.81)
  DAS28-3 (CRP) Month 105: number analyzed (Participants) | 12 | 2 | 14
  DAS28-3 (CRP) Month 105 | 3.31 (1.23) | 1.76 (0.34) | 3.09 (1.26)
  DAS28-3 (CRP) Month 108: number analyzed (Participants) | 7 | 1 | 8
  DAS28-3 (CRP) Month 108 | 3.46 (1.59) | 3.70 (0) | 3.49 (1.47)
  DAS28-3 (CRP) Month 111: number analyzed (Participants) | 3 | 1 | 4
  DAS28-3 (CRP) Month 111 | 1.82 (0.50) | 2.49 (0) | 1.98 (0.53)
  DAS28-3 (CRP) Month 114: number analyzed (Participants) | 1 | 0 | 1
  DAS28-3 (CRP) Month 114 | 2.67 (0) |  | 2.67 (0)

10. Secondary Outcome: Extension Period: Change From Baseline in Disease Activity Score (DAS) 28-3 C-Reactive Protein (CRP)(DAS28-3 CRP) and DAS28-4 Erythrocyte Sedimentation Rate (ESR)(DAS28-4 ESR) at Month 3, 6, 9 and 12
Description: DAS28 is composite score, calculated using mathematical formula, derived from: 1) tender/painful joints count, out of 28 joints (TJC28), 2) swollen joints count, out of 28 joints (SJC28), 3) blood marker of inflammation (ESR [millimeter per hour] or CRP [milligram per liter]). DAS28-4 also include score of general health (GH). GH is general health or participants' global assessment of disease activity on 100 mm visual analog scale (GH score: 0 mm [very well] to 100 mm [extremely bad], higher scores = worse health condition). DAS28-3(CRP) = (0.56*sqrt[TJC28] + 0.28*sqrt[SJC28] + 0.36*ln[CRP+1]) *1.10 + 1.15) and DAS28-4(ESR) = (0.56*sqrt[TJC28] + 0.28*sqrt[SJC28] + 0.70*ln[ESR] + 0.014*GH), where sqrt = square root, ln = natural logarithm. DAS28-4 ESR and DAS28-3 CRP: score ranges from 0 (none) to 9.4 (extreme disease activity), with a higher score indicating more disease activity. Score of <=3.2 indicate low disease activity and score of <2.6 indicate disease remission.
Time Frame: Baseline (Month 0 at the entry of Initial period); Month 3, 6, 9 and 12 of Extension Period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Extension Period: Tofacitinib 5 mg
Number analyzed (Participants) | 48
Scores on a scale
  DAS28-4 (ESR) Baseline: number analyzed (Participants) | 47
  DAS28-4 (ESR) Baseline | 5.68 (1.26)
  DAS28-4 (ESR): Change at Month 3: number analyzed (Participants) | 43
  DAS28-4 (ESR): Change at Month 3 | -2.82 (1.52)
  DAS28-4 (ESR): Change at Month 6: number analyzed (Participants) | 34
  DAS28-4 (ESR): Change at Month 6 | -3.02 (1.50)
  DAS28-4 (ESR): Change at Month 9: number analyzed (Participants) | 15
  DAS28-4 (ESR): Change at Month 9 | -3.13 (1.66)
  DAS28-4 (ESR): Change at Month 12: number analyzed (Participants) | 2
  DAS28-4 (ESR): Change at Month 12 | -2.55 (3.70)
  DAS28-3 (CRP): Baseline | 4.67 (1.24)
  DAS28-3 (CRP): Change at Month 3: number analyzed (Participants) | 42
  DAS28-3 (CRP): Change at Month 3 | -2.36 (1.25)
  DAS28-3 (CRP): Change at Month 6: number analyzed (Participants) | 34
  DAS28-3 (CRP): Change at Month 6 | -2.49 (1.30)
  DAS28-3 (CRP): Change at Month 9: number analyzed (Participants) | 15
  DAS28-3 (CRP): Change at Month 9 | -3.04 (1.49)
  DAS28-3 (CRP): Change at Month 12: number analyzed (Participants) | 1
  DAS28-3 (CRP): Change at Month 12 | 0.29 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.

11. Secondary Outcome: Initial Period: Number (%) of Participants With DAS28-4 (ESR) and DAS28-3 (CRP) <2.6 and ≤3.2
Description: Percent participants with DAS28-4 (ESR) <2.6 and ≤3.2 and percent participants with DAS28-3 (CRP) <2.6 and ≤3.2. The stated number of participants analyzed was the total number of participants in each group. The actual number of participants analyzed on each occasion varied, and is provided for each visit presented.
  DAS28 is a composite score, calculated using a mathematical formula, and is derived from the number of tender/painful joints (out of 28), number of swollen joints (out of 28), and a blood marker of inflammation (ESR or CRP). DAS28-4 also includes a score of general health in the formula.
  The score range is from 0 to 9.4, with a higher score indicating more disease activity. A score of >5.1 indicates active disease, a score of ≤3.2 indicates low disease activity, and a score of <2.6 indicates disease remission.
Time Frame: Every visit until study completion
Population: Full Analysis Set - No Imputation. The number of participants analyzed is the number remaining in the study who had evaluable data for the measure at the given time point.
Measure: Number; unit: Percent of participants
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib
Number analyzed (Participants) | 1123 | 3358 | 4481
Percent of participants
  DAS28-4 (ESR) <2.6 Baseline: number analyzed (Participants) | 1002 | 3296 | 4298
  DAS28-4 (ESR) <2.6 Baseline | 0.2 | 0.3 | 0.3
  DAS28-4 (ESR) <2.6 Month 1: number analyzed (Participants) | 1036 | 3254 | 4290
  DAS28-4 (ESR) <2.6 Month 1 | 19.9 | 20.4 | 20.3
  DAS28-4 (ESR) <2.6 Month 2: number analyzed (Participants) | 1026 | 3222 | 4248
  DAS28-4 (ESR) <2.6 Month 2 | 20.5 | 22.5 | 22.0
  DAS28-4 (ESR) <2.6 Month 3: number analyzed (Participants) | 1033 | 3203 | 4236
  DAS28-4 (ESR) <2.6 Month 3 | 20.0 | 22.9 | 22.2
  DAS28-4 (ESR) <2.6 Month 6: number analyzed (Participants) | 1015 | 3110 | 4125
  DAS28-4 (ESR) <2.6 Month 6 | 22.9 | 23.4 | 23.3
  DAS28-4 (ESR) <2.6 Month 9: number analyzed (Participants) | 992 | 3003 | 3995
  DAS28-4 (ESR) <2.6 Month 9 | 24.4 | 25.1 | 24.9
  DAS28-4 (ESR) <2.6 Month 12: number analyzed (Participants) | 967 | 2862 | 3829
  DAS28-4 (ESR) <2.6 Month 12 | 22.3 | 24.4 | 23.9
  DAS28-4 (ESR) <2.6 Month 15: number analyzed (Participants) | 922 | 2759 | 3681
  DAS28-4 (ESR) <2.6 Month 15 | 23.8 | 25.7 | 25.2
  DAS28-4 (ESR) <2.6 Month 18: number analyzed (Participants) | 899 | 2655 | 3554
  DAS28-4 (ESR) <2.6 Month 18 | 25.3 | 26.9 | 26.4
  DAS28-4 (ESR) <2.6 Month 21: number analyzed (Participants) | 850 | 2547 | 3397
  DAS28-4 (ESR) <2.6 Month 21 | 22.2 | 27.1 | 25.9
  DAS28-4 (ESR) <2.6 Month 24: number analyzed (Participants) | 818 | 2441 | 3259
  DAS28-4 (ESR) <2.6 Month 24 | 22.7 | 26.8 | 25.8
  DAS28-4 (ESR) <2.6 Month 27: number analyzed (Participants) | 787 | 2343 | 3130
  DAS28-4 (ESR) <2.6 Month 27 | 22.6 | 27.9 | 26.5
  DAS28-4 (ESR) <2.6 Month 30: number analyzed (Participants) | 764 | 2257 | 3021
  DAS28-4 (ESR) <2.6 Month 30 | 24.6 | 27.7 | 26.9
  DAS28-4 (ESR) <2.6 Month 33: number analyzed (Participants) | 746 | 2199 | 2945
  DAS28-4 (ESR) <2.6 Month 33 | 23.7 | 28.3 | 27.1
  DAS28-4 (ESR) <2.6 Month 36: number analyzed (Participants) | 720 | 2141 | 2861
  DAS28-4 (ESR) <2.6 Month 36 | 25.6 | 28.9 | 28.1
  DAS28-4 (ESR) <2.6 Month 39: number analyzed (Participants) | 679 | 2056 | 2735
  DAS28-4 (ESR) <2.6 Month 39 | 23.9 | 28.4 | 27.3
  DAS28-4 (ESR) <2.6 Month 42: number analyzed (Participants) | 642 | 1890 | 2532
  DAS28-4 (ESR) <2.6 Month 42 | 24.3 | 27.9 | 27.0
  DAS28-4 (ESR) <2.6 Month 45: number analyzed (Participants) | 609 | 1641 | 2250
  DAS28-4 (ESR) <2.6 Month 45 | 24.1 | 27.5 | 26.6
  DAS28-4 (ESR) <2.6 Month 48: number analyzed (Participants) | 570 | 1471 | 2041
  DAS28-4 (ESR) <2.6 Month 48 | 23.5 | 28.0 | 26.8
  DAS28-4 (ESR) <2.6 Month 51: number analyzed (Participants) | 481 | 1344 | 1825
  DAS28-4 (ESR) <2.6 Month 51 | 28.3 | 27.3 | 27.6
  DAS28-4 (ESR) <2.6 Month 54: number analyzed (Participants) | 467 | 1194 | 1661
  DAS28-4 (ESR) <2.6 Month 54 | 21.4 | 28.3 | 26.4
  DAS28-4 (ESR) <2.6 Month 57: number analyzed (Participants) | 438 | 1006 | 1444
  DAS28-4 (ESR) <2.6 Month 57 | 23.1 | 28.0 | 26.5
  DAS28-4 (ESR) <2.6 Month 60: number analyzed (Participants) | 408 | 908 | 1316
  DAS28-4 (ESR) <2.6 Month 60 | 24.0 | 28.6 | 27.2
  DAS28-4 (ESR) <2.6 Month 63: number analyzed (Participants) | 388 | 825 | 1213
  DAS28-4 (ESR) <2.6 Month 63 | 22.4 | 29.5 | 27.2
  DAS28-4 (ESR) <2.6 Month 66: number analyzed (Participants) | 379 | 700 | 1079
  DAS28-4 (ESR) <2.6 Month 66 | 19.5 | 26.9 | 24.3
  DAS28-4 (ESR) <2.6 Month 69: number analyzed (Participants) | 355 | 483 | 838
  DAS28-4 (ESR) <2.6 Month 69 | 23.9 | 26.3 | 25.3
  DAS28-4 (ESR) <2.6 Month 72: number analyzed (Participants) | 338 | 284 | 622
  DAS28-4 (ESR) <2.6 Month 72 | 25.7 | 25.0 | 25.4
  DAS28-4 (ESR) <2.6 Month 75: number analyzed (Participants) | 299 | 169 | 468
  DAS28-4 (ESR) <2.6 Month 75 | 23.7 | 26.0 | 24.6
  DAS28-4 (ESR) <2.6 Month 78: number analyzed (Participants) | 291 | 91 | 382
  DAS28-4 (ESR) <2.6 Month 78 | 24.7 | 33.0 | 26.7
  DAS28-4 (ESR) <2.6 Month 81: number analyzed (Participants) | 284 | 54 | 338
  DAS28-4 (ESR) <2.6 Month 81 | 24.6 | 22.2 | 24.3
  DAS28-4 (ESR) <2.6 Month 84: number analyzed (Participants) | 271 | 44 | 315
  DAS28-4 (ESR) <2.6 Month 84 | 27.3 | 27.3 | 27.3
  DAS28-4 (ESR) <2.6 Month 87: number analyzed (Participants) | 263 | 41 | 304
  DAS28-4 (ESR) <2.6 Month 87 | 31.2 | 31.7 | 31.3
  DAS28-4 (ESR) <2.6 Month 90: number analyzed (Participants) | 237 | 39 | 276
  DAS28-4 (ESR) <2.6 Month 90 | 28.7 | 25.6 | 28.3
  DAS28-4 (ESR) <2.6 Month 93: number analyzed (Participants) | 191 | 28 | 219
  DAS28-4 (ESR) <2.6 Month 93 | 28.3 | 28.6 | 28.3
  DAS28-4 (ESR) <2.6 Month 96: number analyzed (Participants) | 142 | 16 | 158
  DAS28-4 (ESR) <2.6 Month 96 | 25.4 | 18.8 | 24.7
  DAS28-4 (ESR) <2.6 Month 99: number analyzed (Participants) | 65 | 11 | 76
  DAS28-4 (ESR) <2.6 Month 99 | 27.7 | 36.4 | 28.9
  DAS28-4 (ESR) <2.6 Month 102: number analyzed (Participants) | 22 | 4 | 26
  DAS28-4 (ESR) <2.6 Month 102 | 31.8 | 50.0 | 34.6
  DAS28-4 (ESR) <2.6 Month 105: number analyzed (Participants) | 14 | 3 | 17
  DAS28-4 (ESR) <2.6 Month 105 | 28.6 | 33.3 | 29.4
  DAS28-4 (ESR) <2.6 Month 108: number analyzed (Participants) | 8 | 1 | 9
  DAS28-4 (ESR) <2.6 Month 108 | 25.0 | 0 | 22.2
  DAS28-4 (ESR) </=3.2 Baseline: number analyzed (Participants) | 1002 | 3296 | 4298
  DAS28-4 (ESR) </=3.2 Baseline | 0.4 | 0.7 | 0.6
  DAS28-4 (ESR) </=3.2 Month 1: number analyzed (Participants) | 1036 | 3254 | 4290
  DAS28-4 (ESR) </=3.2 Month 1 | 34.2 | 37.6 | 36.8
  DAS28-4 (ESR) </=3.2 Month 2: number analyzed (Participants) | 1026 | 3222 | 4248
  DAS28-4 (ESR) </=3.2 Month 2 | 36.7 | 40.5 | 39.6
  DAS28-4 (ESR) </=3.2 Month 3: number analyzed (Participants) | 1033 | 3203 | 4236
  DAS28-4 (ESR) </=3.2 Month 3 | 36.6 | 41.6 | 40.4
  DAS28-4 (ESR) </=3.2 Month 6: number analyzed (Participants) | 1015 | 3110 | 4125
  DAS28-4 (ESR) </=3.2 Month 6 | 39.8 | 42.5 | 41.9
  DAS28-4 (ESR) </=3.2 Month 9: number analyzed (Participants) | 992 | 3003 | 3995
  DAS28-4 (ESR) </=3.2 Month 9 | 41.3 | 43.8 | 43.2
  DAS28-4 (ESR) </=3.2 Month 12: number analyzed (Participants) | 967 | 2862 | 3829
  DAS28-4 (ESR) </=3.2 Month 12 | 42.1 | 42.5 | 42.4
  DAS28-4 (ESR) </=3.2 Month 18: number analyzed (Participants) | 899 | 2655 | 3554
  DAS28-4 (ESR) </=3.2 Month 18 | 42.7 | 45.0 | 44.4
  DAS28-4 (ESR) </=3.2 Month 21: number analyzed (Participants) | 850 | 2547 | 3397
  DAS28-4 (ESR) </=3.2 Month 21 | 41.9 | 47.2 | 45.9
  DAS28-4 (ESR) </=3.2 Month 24: number analyzed (Participants) | 818 | 2441 | 3259
  DAS28-4 (ESR) </=3.2 Month 24 | 42.5 | 46.5 | 45.5
  DAS28-4 (ESR) </=3.2 Month 27: number analyzed (Participants) | 787 | 2343 | 3130
  DAS28-4 (ESR) </=3.2 Month 27 | 44.9 | 46.9 | 46.4
  DAS28-4 (ESR) </=3.2 Month 30: number analyzed (Participants) | 764 | 2257 | 3021
  DAS28-4 (ESR) </=3.2 Month 30 | 42.8 | 47.4 | 46.2
  DAS28-4 (ESR) </=3.2 Month 33: number analyzed (Participants) | 746 | 2199 | 2945
  DAS28-4 (ESR) </=3.2 Month 33 | 42.8 | 47.5 | 46.3
  DAS28-4 (ESR) </=3.2 Month 36: number analyzed (Participants) | 720 | 2141 | 2861
  DAS28-4 (ESR) </=3.2 Month 36 | 44.6 | 48.4 | 47.5
  DAS28-4 (ESR) </=3.2 Month 39: number analyzed (Participants) | 679 | 2056 | 2735
  DAS28-4 (ESR) </=3.2 Month 39 | 42.6 | 48.3 | 46.9
  DAS28-4 (ESR) </=3.2 Month 42: number analyzed (Participants) | 642 | 1890 | 2532
  DAS28-4 (ESR) </=3.2 Month 42 | 45.8 | 49.2 | 48.3
  DAS28-4 (ESR) </=3.2 Month 45: number analyzed (Participants) | 609 | 1641 | 2250
  DAS28-4 (ESR) </=3.2 Month 45 | 45.3 | 48.4 | 47.6
  DAS28-4 (ESR) </=3.2 Month 48: number analyzed (Participants) | 570 | 1471 | 2041
  DAS28-4 (ESR) </=3.2 Month 48 | 46.1 | 49.4 | 48.5
  DAS28-4 (ESR) </=3.2 Month 51: number analyzed (Participants) | 481 | 1344 | 1825
  DAS28-4 (ESR) </=3.2 Month 51 | 44.9 | 49.0 | 47.9
  DAS28-4 (ESR) </=3.2 Month 54: number analyzed (Participants) | 467 | 1194 | 1661
  DAS28-4 (ESR) </=3.2 Month 54 | 43.7 | 49.4 | 47.8
  DAS28-4 (ESR) </=3.2 Month 57: number analyzed (Participants) | 438 | 1006 | 1444
  DAS28-4 (ESR) </=3.2 Month 57 | 45.2 | 50.3 | 48.8
  DAS28-4 (ESR) </=3.2 Month 60: number analyzed (Participants) | 408 | 908 | 1316
  DAS28-4 (ESR) </=3.2 Month 60 | 46.3 | 49.9 | 48.8
  DAS28-4 (ESR) </=3.2 Month 63: number analyzed (Participants) | 388 | 825 | 1213
  DAS28-4 (ESR) </=3.2 Month 63 | 41.0 | 49.9 | 47.1
  DAS28-4 (ESR) </=3.2 Month 66: number analyzed (Participants) | 379 | 700 | 1079
  DAS28-4 (ESR) </=3.2 Month 66 | 38.8 | 49.7 | 45.9
  DAS28-4 (ESR) </=3.2 Month 69: number analyzed (Participants) | 355 | 483 | 838
  DAS28-4 (ESR) </=3.2 Month 69 | 45.6 | 50.3 | 48.3
  DAS28-4 (ESR) </=3.2 Month 72: number analyzed (Participants) | 338 | 284 | 622
  DAS28-4 (ESR) </=3.2 Month 72 | 44.7 | 48.2 | 46.3
  DAS28-4 (ESR) </=3.2 Month 75: number analyzed (Participants) | 299 | 169 | 468
  DAS28-4 (ESR) </=3.2 Month 75 | 43.1 | 48.5 | 45.1
  DAS28-4 (ESR) </=3.2 Month 78: number analyzed (Participants) | 291 | 91 | 382
  DAS28-4 (ESR) </=3.2 Month 78 | 44.7 | 45.1 | 44.8
  DAS28-4 (ESR) </=3.2 Month 81: number analyzed (Participants) | 284 | 54 | 338
  DAS28-4 (ESR) </=3.2 Month 81 | 49.3 | 48.1 | 49.1
  DAS28-4 (ESR) </=3.2 Month 84: number analyzed (Participants) | 271 | 44 | 315
  DAS28-4 (ESR) </=3.2 Month 84 | 47.2 | 45.5 | 47.0
  DAS28-4 (ESR) </=3.2 Month 87: number analyzed (Participants) | 263 | 41 | 304
  DAS28-4 (ESR) </=3.2 Month 87 | 47.9 | 46.3 | 47.7
  DAS28-4 (ESR) </=3.2 Month 90: number analyzed (Participants) | 237 | 39 | 276
  DAS28-4 (ESR) </=3.2 Month 90 | 46.0 | 46.2 | 46.0
  DAS28-4 (ESR) </=3.2 Month 93: number analyzed (Participants) | 191 | 28 | 219
  DAS28-4 (ESR) </=3.2 Month 93 | 48.2 | 50.0 | 48.4
  DAS28-4 (ESR) </=3.2 Month 96: number analyzed (Participants) | 142 | 16 | 158
  DAS28-4 (ESR) </=3.2 Month 96 | 47.2 | 43.8 | 46.8
  DAS28-4 (ESR) </=3.2 Month 99: number analyzed (Participants) | 65 | 11 | 76
  DAS28-4 (ESR) </=3.2 Month 99 | 43.1 | 54.5 | 44.7
  DAS28-4 (ESR) </=3.2 Month 102: number analyzed (Participants) | 22 | 4 | 26
  DAS28-4 (ESR) </=3.2 Month 102 | 45.5 | 50.0 | 46.2
  DAS28-4 (ESR) </=3.2 Month 105: number analyzed (Participants) | 14 | 3 | 17
  DAS28-4 (ESR) </=3.2 Month 105 | 42.9 | 66.7 | 47.1
  DAS28-4 (ESR) </=3.2 Month 108: number analyzed (Participants) | 8 | 1 | 9
  DAS28-4 (ESR) </=3.2 Month 108 | 50.0 | 0 | 44.4
  DAS28-3 (CRP) <2.6 Baseline: number analyzed (Participants) | 1112 | 3340 | 4452
  DAS28-3 (CRP) <2.6 Baseline | 0.5 | 0.9 | 0.8
  DAS28-3 (CRP) <2.6 Month 1: number analyzed (Participants) | 1096 | 3234 | 4330
  DAS28-3 (CRP) <2.6 Month 1 | 38.0 | 43.0 | 41.7
  DAS28-3 (CRP) <2.6 Month 2: number analyzed (Participants) | 1070 | 3180 | 4250
  DAS28-3 (CRP) <2.6 Month 2 | 39.7 | 47.1 | 45.2
  DAS28-3 (CRP) <2.6 Month 3: number analyzed (Participants) | 1057 | 3190 | 4247
  DAS28-3 (CRP) <2.6 Month 3 | 42.3 | 47.5 | 46.2
  DAS28-3 (CRP) <2.6 Month 6: number analyzed (Participants) | 1026 | 3106 | 4132
  DAS28-3 (CRP) <2.6 Month 6 | 45.2 | 49.0 | 48.1
  DAS28-3 (CRP) <2.6 Month 9: number analyzed (Participants) | 993 | 3008 | 4001
  DAS28-3 (CRP) <2.6 Month 9 | 47.1 | 50.7 | 49.8
  DAS28-3 (CRP) <2.6 Month 12: number analyzed (Participants) | 962 | 2874 | 3836
  DAS28-3 (CRP) <2.6 Month 12 | 47.8 | 51.8 | 50.8
  DAS28-3 (CRP) <2.6 Month 15: number analyzed (Participants) | 923 | 2761 | 3684
  DAS28-3 (CRP) <2.6 Month 15 | 50.6 | 52.3 | 51.9
  DAS28-3 (CRP) <2.6 Month 18: number analyzed (Participants) | 899 | 2654 | 3553
  DAS28-3 (CRP) <2.6 Month 18 | 51.3 | 54.1 | 53.4
  DAS28-3 (CRP) <2.6 Month 21: number analyzed (Participants) | 856 | 2556 | 3412
  DAS28-3 (CRP) <2.6 Month 21 | 51.1 | 55.5 | 54.4
  DAS28-3 (CRP) <2.6 Month 24: number analyzed (Participants) | 813 | 2456 | 3269
  DAS28-3 (CRP) <2.6 Month 24 | 51.9 | 55.3 | 54.4
  DAS28-3 (CRP) <2.6 Month 27: number analyzed (Participants) | 793 | 2345 | 3138
  DAS28-3 (CRP) <2.6 Month 27 | 53.2 | 55.8 | 55.2
  DAS28-3 (CRP) <2.6 Month 30: number analyzed (Participants) | 766 | 2271 | 3037
  DAS28-3 (CRP) <2.6 Month 30 | 53.3 | 56.8 | 55.9
  DAS28-3 (CRP) <2.6 Month 33: number analyzed (Participants) | 745 | 2209 | 2954
  DAS28-3 (CRP) <2.6 Month 33 | 54.1 | 56.0 | 55.6
  DAS28-3 (CRP) <2.6 Month 36: number analyzed (Participants) | 724 | 2142 | 2866
  DAS28-3 (CRP) <2.6 Month 36 | 52.9 | 55.6 | 54.9
  DAS28-3 (CRP) <2.6 Month 39: number analyzed (Participants) | 686 | 2057 | 2743
  DAS28-3 (CRP) <2.6 Month 39 | 54.2 | 56.9 | 56.2
  DAS28-3 (CRP) <2.6 Month 42: number analyzed (Participants) | 653 | 1893 | 2546
  DAS28-3 (CRP) <2.6 Month 42 | 54.2 | 56.8 | 56.2
  DAS28-3 (CRP) <2.6 Month 45: number analyzed (Participants) | 611 | 1644 | 2255
  DAS28-3 (CRP) <2.6 Month 45 | 56.3 | 58.6 | 58.0
  DAS28-3 (CRP) <2.6 Month 48: number analyzed (Participants) | 579 | 1469 | 2048
  DAS28-3 (CRP) <2.6 Month 48 | 55.4 | 59.3 | 58.2
  DAS28-3 (CRP) <2.6 Month 51: number analyzed (Participants) | 487 | 1348 | 1835
  DAS28-3 (CRP) <2.6 Month 51 | 56.1 | 57.3 | 56.9
  DAS28-3 (CRP) <2.6 Month 54: number analyzed (Participants) | 468 | 1198 | 1666
  DAS28-3 (CRP) <2.6 Month 54 | 52.6 | 57.8 | 56.3
  DAS28-3 (CRP) <2.6 Month 57: number analyzed (Participants) | 439 | 1011 | 1450
  DAS28-3 (CRP) <2.6 Month 57 | 55.6 | 57.7 | 57.0
  DAS28-3 (CRP) <2.6 Month 60: number analyzed (Participants) | 407 | 913 | 1320
  DAS28-3 (CRP) <2.6 Month 60 | 55.0 | 57.9 | 57.0
  DAS28-3 (CRP) <2.6 Month 63: number analyzed (Participants) | 390 | 824 | 1214
  DAS28-3 (CRP) <2.6 Month 63 | 51.0 | 58.1 | 55.8
  DAS28-3 (CRP) <2.6 Month 66: number analyzed (Participants) | 376 | 702 | 1078
  DAS28-3 (CRP) <2.6 Month 66 | 51.9 | 59.3 | 56.7
  DAS28-3 (CRP) <2.6 Month 69: number analyzed (Participants) | 355 | 483 | 838
  DAS28-3 (CRP) <2.6 Month 69 | 53.5 | 57.8 | 56.0
  DAS28-3 (CRP) <2.6 Month 72: number analyzed (Participants) | 337 | 285 | 622
  DAS28-3 (CRP) <2.6 Month 72 | 52.2 | 55.4 | 53.7
  DAS28-3 (CRP) <2.6 Month 75: number analyzed (Participants) | 304 | 170 | 474
  DAS28-3 (CRP) <2.6 Month 75 | 53.9 | 53.5 | 53.8
  DAS28-3 (CRP) <2.6 Month 78: number analyzed (Participants) | 292 | 91 | 383
  DAS28-3 (CRP) <2.6 Month 78 | 58.2 | 51.6 | 56.7
  DAS28-3 (CRP) <2.6 Month 81: number analyzed (Participants) | 285 | 54 | 339
  DAS28-3 (CRP) <2.6 Month 81 | 58.6 | 51.9 | 57.5
  DAS28-3 (CRP) <2.6 Month 84: number analyzed (Participants) | 269 | 44 | 313
  DAS28-3 (CRP) <2.6 Month 84 | 61.7 | 43.2 | 59.1
  DAS28-3 (CRP) <2.6 Month 87: number analyzed (Participants) | 264 | 41 | 305
  DAS28-3 (CRP) <2.6 Month 87 | 60.2 | 48.8 | 58.7
  DAS28-3 (CRP) <2.6 Month 90: number analyzed (Participants) | 240 | 39 | 279
  DAS28-3 (CRP) <2.6 Month 90 | 60.8 | 46.2 | 58.8
  DAS28-3 (CRP) <2.6 Month 93: number analyzed (Participants) | 196 | 28 | 224
  DAS28-3 (CRP) <2.6 Month 93 | 56.1 | 53.6 | 55.8
  DAS28-3 (CRP) <2.6 Month 96: number analyzed (Participants) | 144 | 16 | 160
  DAS28-3 (CRP) <2.6 Month 96 | 56.3 | 37.5 | 54.4
  DAS28-3 (CRP) <2.6 Month 99: number analyzed (Participants) | 64 | 11 | 75
  DAS28-3 (CRP) <2.6 Month 99 | 50.0 | 63.6 | 52.0
  DAS28-3 (CRP) <2.6 Month 102: number analyzed (Participants) | 13 | 3 | 16
  DAS28-3 (CRP) <2.6 Month 102 | 46.2 | 66.7 | 50.0
  DAS28-3 (CRP) <2.6 Month 105: number analyzed (Participants) | 12 | 2 | 14
  DAS28-3 (CRP) <2.6 Month 105 | 33.3 | 100 | 42.9
  DAS28-3 (CRP) <2.6 Month 108: number analyzed (Participants) | 7 | 1 | 8
  DAS28-3 (CRP) <2.6 Month 108 | 42.9 | 0 | 37.5
  DAS28-3 (CRP) <2.6 Month 111: number analyzed (Participants) | 3 | 1 | 4
  DAS28-3 (CRP) <2.6 Month 111 | 100 | 100 | 100
  DAS28-3 (CRP) </=3.2 Month 1: number analyzed (Participants) | 1096 | 3234 | 4330
  DAS28-3 (CRP) </=3.2 Month 1 | 55.3 | 61.9 | 60.2
  DAS28-3 (CRP) </=3.2 Month 2: number analyzed (Participants) | 1070 | 3180 | 4250
  DAS28-3 (CRP) </=3.2 Month 2 | 60.7 | 64.5 | 63.6
  DAS28-3 (CRP) </=3.2 Month 3: number analyzed (Participants) | 1057 | 3190 | 4247
  DAS28-3 (CRP) </=3.2 Month 3 | 60.6 | 66.3 | 64.9
  DAS28-3 (CRP) </=3.2 Month 6: number analyzed (Participants) | 1026 | 3106 | 4132
  DAS28-3 (CRP) </=3.2 Month 6 | 64.4 | 67.1 | 66.4
  DAS28-3 (CRP) </=3.2 Month 9: number analyzed (Participants) | 993 | 3008 | 4001
  DAS28-3 (CRP) </=3.2 Month 9 | 66.4 | 68.3 | 67.8
  DAS28-3 (CRP) </=3.2 Month 12: number analyzed (Participants) | 962 | 2874 | 3836
  DAS28-3 (CRP) </=3.2 Month 12 | 66.1 | 70.0 | 69.0
  DAS28-3 (CRP) </=3.2 Month 15: number analyzed (Participants) | 923 | 2761 | 3684
  DAS28-3 (CRP) </=3.2 Month 15 | 70.0 | 70.0 | 70.0
  DAS28-3 (CRP) </=3.2 Month 18: number analyzed (Participants) | 899 | 2654 | 3553
  DAS28-3 (CRP) </=3.2 Month 18 | 69.2 | 71.7 | 71.1
  DAS28-3 (CRP) </=3.2 Month 21: number analyzed (Participants) | 856 | 2556 | 3412
  DAS28-3 (CRP) </=3.2 Month 21 | 69.5 | 72.5 | 71.8
  DAS28-3 (CRP) </=3.2 Month 24: number analyzed (Participants) | 813 | 2456 | 3269
  DAS28-3 (CRP) </=3.2 Month 24 | 71.7 | 72.5 | 72.3
  DAS28-3 (CRP) </=3.2 Month 27: number analyzed (Participants) | 793 | 2345 | 3138
  DAS28-3 (CRP) </=3.2 Month 27 | 72.6 | 73.0 | 72.9
  DAS28-3 (CRP) </=3.2 Month 30: number analyzed (Participants) | 766 | 2271 | 3037
  DAS28-3 (CRP) </=3.2 Month 30 | 73.0 | 73.8 | 73.6
  DAS28-3 (CRP) </=3.2 Month 33: number analyzed (Participants) | 745 | 2209 | 2954
  DAS28-3 (CRP) </=3.2 Month 33 | 72.2 | 74.5 | 73.9
  DAS28-3 (CRP) </=3.2 Month 36: number analyzed (Participants) | 724 | 2142 | 2866
  DAS28-3 (CRP) </=3.2 Month 36 | 73.8 | 73.4 | 73.5
  DAS28-3 (CRP) </=3.2 Month 39: number analyzed (Participants) | 686 | 2057 | 2743
  DAS28-3 (CRP) </=3.2 Month 39 | 73.2 | 74.6 | 74.2
  DAS28-3 (CRP) </=3.2 Month 42: number analyzed (Participants) | 653 | 1893 | 2546
  DAS28-3 (CRP) </=3.2 Month 42 | 73.8 | 74.7 | 74.5
  DAS28-3 (CRP) </=3.2 Month 45: number analyzed (Participants) | 611 | 1644 | 2255
  DAS28-3 (CRP) </=3.2 Month 45 | 74.6 | 75.2 | 75.1
  DAS28-3 (CRP) </=3.2 Month 48: number analyzed (Participants) | 579 | 1469 | 2048
  DAS28-3 (CRP) </=3.2 Month 48 | 74.6 | 75.0 | 74.9
  DAS28-3 (CRP) </=3.2 Month 51: number analyzed (Participants) | 487 | 1348 | 1835
  DAS28-3 (CRP) </=3.2 Month 51 | 74.3 | 75.1 | 74.9
  DAS28-3 (CRP) </=3.2 Month 54: number analyzed (Participants) | 468 | 1198 | 1666
  DAS28-3 (CRP) </=3.2 Month 54 | 71.4 | 76.4 | 75.0
  DAS28-3 (CRP) </=3.2 Month 57: number analyzed (Participants) | 439 | 1011 | 1450
  DAS28-3 (CRP) </=3.2 Month 57 | 73.6 | 75.2 | 74.7
  DAS28-3 (CRP) </=3.2 Month 60: number analyzed (Participants) | 407 | 913 | 1320
  DAS28-3 (CRP) </=3.2 Month 60 | 72.5 | 77.0 | 75.6
  DAS28-3 (CRP) </=3.2 Month 63: number analyzed (Participants) | 390 | 824 | 1214
  DAS28-3 (CRP) </=3.2 Month 63 | 72.8 | 76.5 | 75.3
  DAS28-3 (CRP) </=3.2 Month 66: number analyzed (Participants) | 376 | 702 | 1078
  DAS28-3 (CRP) </=3.2 Month 66 | 71.5 | 78.1 | 75.8
  DAS28-3 (CRP) </=3.2 Month 69: number analyzed (Participants) | 355 | 483 | 838
  DAS28-3 (CRP) </=3.2 Month 69 | 69.9 | 77.0 | 74.0
  DAS28-3 (CRP) </=3.2 Month 72: number analyzed (Participants) | 337 | 285 | 622
  DAS28-3 (CRP) </=3.2 Month 72 | 74.8 | 73.3 | 74.1
  DAS28-3 (CRP) </=3.2 Month 75: number analyzed (Participants) | 304 | 170 | 474
  DAS28-3 (CRP) </=3.2 Month 75 | 77.0 | 72.9 | 75.5
  DAS28-3 (CRP) </=3.2 Month 78: number analyzed (Participants) | 292 | 91 | 383
  DAS28-3 (CRP) </=3.2 Month 78 | 74.3 | 70.3 | 73.4
  DAS28-3 (CRP) </=3.2 Month 81: number analyzed (Participants) | 285 | 54 | 339
  DAS28-3 (CRP) </=3.2 Month 81 | 75.8 | 68.5 | 74.6
  DAS28-3 (CRP) </=3.2 Month 84: number analyzed (Participants) | 269 | 44 | 313
  DAS28-3 (CRP) </=3.2 Month 84 | 79.2 | 68.2 | 77.6
  DAS28-4 (CRP) </=3.2 Month 87: number analyzed (Participants) | 264 | 41 | 305
  DAS28-4 (CRP) </=3.2 Month 87 | 81.1 | 70.7 | 79.7
  DAS28-3 (CRP) </=3.2 Month 90: number analyzed (Participants) | 240 | 39 | 279
  DAS28-3 (CRP) </=3.2 Month 90 | 77.1 | 74.4 | 76.7
  DAS28-3 (CRP) </=3.2 Month 93: number analyzed (Participants) | 196 | 28 | 224
  DAS28-3 (CRP) </=3.2 Month 93 | 75.0 | 67.9 | 74.1
  DAS28-3 (CRP) </=3.2 Month 96: number analyzed (Participants) | 144 | 16 | 160
  DAS28-3 (CRP) </=3.2 Month 96 | 77.1 | 87.5 | 78.1
  DAS28-3 (CRP) </=3.2 Month 99: number analyzed (Participants) | 64 | 11 | 75
  DAS28-3 (CRP) </=3.2 Month 99 | 76.6 | 81.8 | 77.3
  DAS28-3 (CRP) </=3.2 Month 102: number analyzed (Participants) | 13 | 3 | 16
  DAS28-3 (CRP) </=3.2 Month 102 | 84.6 | 66.7 | 81.3
  DAS28-3 (CRP) </=3.2 Month 105: number analyzed (Participants) | 12 | 2 | 14
  DAS28-3 (CRP) </=3.2 Month 105 | 50.0 | 100 | 57.1
  DAS28-3 (CRP) </=3.2 Month 108: number analyzed (Participants) | 7 | 1 | 8
  DAS28-3 (CRP) </=3.2 Month 108 | 42.9 | 0 | 37.5

12. Secondary Outcome: Extension Period: Percentage of Participants With DAS28-4 (ESR) and DAS28-3 (CRP) Less Than (<) 2.6 and Less Than or (<=) 3.2
Description: DAS28 is composite score, calculated using mathematical formula, derived from: 1) tender/painful joints count, out of 28 joints (TJC28), 2) swollen joints count, out of 28 joints (SJC28), 3) blood marker of inflammation (ESR [millimeter per hour] or CRP [milligram per liter]). DAS28-4 also include score of GH. GH is general health or participants' global assessment of disease activity on 100 mm visual analog scale (GH score: 0 mm [very well] to 100 mm [extremely bad], higher scores = worse health condition). DAS28-3(CRP) = (0.56*sqrt[TJC28] + 0.28*sqrt[SJC28] + 0.36*ln[CRP+1]) *1.10 + 1.15) and DAS28-4(ESR) = (0.56*sqrt[TJC28] + 0.28*sqrt[SJC28] + 0.70*ln[ESR] + 0.014*GH), where sqrt = square root, ln = natural logarithm. DAS28-4 ESR and DAS28-3 CRP: score range is from 0 (none) to 9.4 (extreme disease activity), with a higher score indicating more disease activity. Score of <=3.2 indicate low disease activity and score of <2.6 indicate disease remission.
Time Frame: Baseline (Day 1 at the entry of Extension period); Month 3, 6, 9 and 12 of Extension Period
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Extension Period: Tofacitinib 5 mg
Number analyzed (Participants) | 48
Percentage of participants
  DAS28-4 (ESR) <2.6: Baseline | 12.5
  DAS28-4 (ESR) <2.6: Month 3: number analyzed (Participants) | 44
  DAS28-4 (ESR) <2.6: Month 3 | 40.9
  DAS28-4 (ESR) <2.6: Month 6: number analyzed (Participants) | 35
  DAS28-4 (ESR) <2.6: Month 6 | 45.7
  DAS28-4 (ESR) <2.6: Month 9: number analyzed (Participants) | 15
  DAS28-4 (ESR) <2.6: Month 9 | 46.7
  DAS28-4 (ESR) <2.6: Month 12: number analyzed (Participants) | 2
  DAS28-4 (ESR) <2.6: Month 12 | 50.0
  DAS28-4 (ESR) <=3.2: Baseline | 29.2
  DAS28-4 (ESR) <=3.2: Month 3: number analyzed (Participants) | 44
  DAS28-4 (ESR) <=3.2: Month 3 | 68.2
  DAS28-4 (ESR) <=3.2: Month 6: number analyzed (Participants) | 35
  DAS28-4 (ESR) <=3.2: Month 6 | 68.6
  DAS28-4 (ESR) <=3.2: Month 9: number analyzed (Participants) | 15
  DAS28-4 (ESR) <=3.2: Month 9 | 66.7
  DAS28-4 (ESR) <=3.2: Month 12: number analyzed (Participants) | 2
  DAS28-4 (ESR) <=3.2: Month 12 | 50.0
  DAS28-3 (CRP) <2.6: Baseline: number analyzed (Participants) | 47
  DAS28-3 (CRP) <2.6: Baseline | 27.7
  DAS28-3 (CRP) <2.6: Month 3: number analyzed (Participants) | 42
  DAS28-3 (CRP) <2.6: Month 3 | 61.9
  DAS28-3 (CRP) <2.6: Month 6: number analyzed (Participants) | 34
  DAS28-3 (CRP) <2.6: Month 6 | 67.6
  DAS28-3 (CRP) <2.6: Month 9: number analyzed (Participants) | 15
  DAS28-3 (CRP) <2.6: Month 9 | 80.0
  DAS28-3 (CRP) <2.6: Month 12: number analyzed (Participants) | 1
  DAS28-3 (CRP) <2.6: Month 12 | 0
  DAS28-3 (CRP) <=3.2: Baseline: number analyzed (Participants) | 47
  DAS28-3 (CRP) <=3.2: Baseline | 53.2
  DAS28-3 (CRP) <=3.2: Month 3: number analyzed (Participants) | 42
  DAS28-3 (CRP) <=3.2: Month 3 | 85.7
  DAS28-3 (CRP) <=3.2: Month 6: number analyzed (Participants) | 34
  DAS28-3 (CRP) <=3.2: Month 6 | 85.3
  DAS28-3 (CRP) <=3.2: Month 9: number analyzed (Participants) | 15
  DAS28-3 (CRP) <=3.2: Month 9 | 80.0
  DAS28-3 (CRP) <=3.2: Month 12: number analyzed (Participants) | 1
  DAS28-3 (CRP) <=3.2: Month 12 | 0

13. Secondary Outcome: Initial Period: Health Assessment Questionnaire - Disability Index (HAQ-DI) Score
Description: Change from baseline by visit. HAQ-DI scores range from 0 to 3, where lower score implies less disease. A reduction from baseline in score indicates an improvement in condition. A clinically meaningful decrease from baseline is defined as a decrease of at least 0.22 units. The stated number of participants analyzed was the total number of participants in each group. The actual number of participants analyzed on each occasion varied, and is provided for each visit presented.
Time Frame: Every visit until study completion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib
Number analyzed (Participants) | 1123 | 3358 | 4481
Units on scale
  Month 1: number analyzed (Participants) | 1098 | 3264 | 4362
  Month 1 | -0.57 (0.62) | -0.61 (0.63) | -0.60 (0.63)
  Month 2: number analyzed (Participants) | 1067 | 3213 | 4280
  Month 2 | -0.58 (0.62) | -0.65 (0.65) | -0.63 (0.65)
  Month 3: number analyzed (Participants) | 1057 | 3196 | 4253
  Month 3 | -0.58 (0.63) | -0.66 (0.65) | -0.64 (0.65)
  Month 6: number analyzed (Participants) | 1029 | 3105 | 4134
  Month 6 | -0.58 (0.65) | -0.65 (0.66) | -0.64 (0.66)
  Month 9: number analyzed (Participants) | 990 | 2992 | 3982
  Month 9 | -0.58 (0.64) | -0.66 (0.66) | -0.64 (0.66)
  Month 12: number analyzed (Participants) | 960 | 2866 | 3826
  Month 12 | -0.58 (0.65) | -0.66 (0.67) | -0.64 (0.67)
  Month 15: number analyzed (Participants) | 926 | 2756 | 3682
  Month 15 | -0.61 (0.65) | -0.68 (0.68) | -0.66 (0.67)
  Month 18: number analyzed (Participants) | 898 | 2646 | 3544
  Month 18 | -0.60 (0.65) | -0.68 (0.67) | -0.66 (0.67)
  Month 21: number analyzed (Participants) | 849 | 2542 | 3391
  Month 21 | -0.60 (0.67) | -0.69 (0.68) | -0.67 (0.68)
  Month 24: number analyzed (Participants) | 815 | 2443 | 3258
  Month 24 | -0.60 (0.65) | -0.69 (0.68) | -0.67 (0.67)
  Month 27: number analyzed (Participants) | 789 | 2341 | 3130
  Month 27 | -0.62 (0.65) | -0.69 (0.68) | -0.67 (0.67)
  Month 30: number analyzed (Participants) | 757 | 2258 | 3015
  Month 30 | -0.58 (0.66) | -0.68 (0.69) | -0.66 (0.68)
  Month 33: number analyzed (Participants) | 741 | 2194 | 2935
  Month 33 | -0.60 (0.66) | -0.67 (0.69) | -0.66 (0.68)
  Month 36: number analyzed (Participants) | 720 | 2136 | 2856
  Month 36 | -0.63 (0.66) | -0.67 (0.68) | -0.66 (0.67)
  Month 39: number analyzed (Participants) | 683 | 2053 | 2736
  Month 39 | -0.59 (0.67) | -0.68 (0.69) | -0.66 (0.69)
  Month 42: number analyzed (Participants) | 649 | 1884 | 2533
  Month 42 | -0.59 (0.67) | -0.66 (0.68) | -0.65 (0.68)
  Month 45: number analyzed (Participants) | 609 | 1636 | 2245
  Month 45 | -0.59 (0.69) | -0.64 (0.69) | -0.63 (0.69)
  Month 48: number analyzed (Participants) | 575 | 1468 | 2043
  Month 48 | -0.58 (0.69) | -0.64 (0.69) | -0.62 (0.68)
  Month 51: number analyzed (Participants) | 482 | 1332 | 1814
  Month 51 | -0.59 (0.69) | -0.63 (0.66) | -0.62 (0.67)
  Month 54: number analyzed (Participants) | 463 | 1191 | 1654
  Month 54 | -0.57 (0.68) | -0.65 (0.67) | -0.63 (0.67)
  Month 57: number analyzed (Participants) | 434 | 1011 | 1445
  Month 57 | -0.57 (0.69) | -0.66 (0.68) | -0.63 (0.68)
  Month 60: number analyzed (Participants) | 405 | 916 | 1321
  Month 60 | -0.59 (0.68) | -0.66 (0.69) | -0.64 (0.69)
  Month 63: number analyzed (Participants) | 392 | 828 | 1220
  Month 63 | -0.57 (0.68) | -0.68 (0.70) | -0.64 (0.69)
  Month 66: number analyzed (Participants) | 375 | 702 | 1077
  Month 66 | -0.54 (0.70) | -0.67 (0.69) | -0.63 (0.70)
  Month 69: number analyzed (Participants) | 353 | 484 | 837
  Month 69 | -0.55 (0.70) | -0.66 (0.71) | -0.61 (0.71)
  Month 72: number analyzed (Participants) | 335 | 286 | 621
  Month 72 | -0.57 (0.71) | -0.62 (0.73) | -0.59 (0.72)
  Month 75: number analyzed (Participants) | 303 | 171 | 474
  Month 75 | -0.57 (0.72) | -0.58 (0.73) | -0.57 (0.72)
  Month 78: number analyzed (Participants) | 289 | 91 | 380
  Month 78 | -0.54 (0.73) | -0.61 (0.78) | -0.56 (0.74)
  Month 81: number analyzed (Participants) | 282 | 54 | 336
  Month 81 | -0.55 (0.73) | -0.64 (0.68) | -0.56 (0.72)
  Month 84: number analyzed (Participants) | 269 | 44 | 313
  Month 84 | -0.53 (0.73) | -0.56 (0.68) | -0.53 (0.72)
  Month 87: number analyzed (Participants) | 262 | 41 | 303
  Month 87 | -0.53 (0.70) | -0.53 (0.60) | -0.53 (0.69)
  Month 90: number analyzed (Participants) | 240 | 39 | 279
  Month 90 | -0.52 (0.72) | -0.54 (0.61) | -0.52 (0.70)
  Month 93: number analyzed (Participants) | 194 | 28 | 222
  Month 93 | -0.52 (0.75) | -0.50 (0.60) | -0.52 (0.73)
  Month 96: number analyzed (Participants) | 143 | 16 | 159
  Month 96 | -0.54 (0.77) | -0.48 (0.58) | -0.53 (0.75)
  Month 99: number analyzed (Participants) | 64 | 11 | 75
  Month 99 | -0.53 (0.80) | -0.44 (0.51) | -0.52 (0.76)
  Month 102: number analyzed (Participants) | 22 | 3 | 25
  Month 102 | -0.61 (0.82) | -0.29 (0.85) | -0.58 (0.81)
  Month 105: number analyzed (Participants) | 15 | 3 | 18
  Month 105 | -0.65 (0.91) | -0.50 (0.99) | -0.63 (0.90)
  Month 108: number analyzed (Participants) | 8 | 1 | 9
  Month 108 | -0.89 (0.97) | 0.13 (0) | -0.78 (0.97)
  Month 111: number analyzed (Participants) | 3 | 1 | 4
  Month 111 | -1.29 (1.34) | 0.25 (0) | -0.91 (1.34)
  Month 114: number analyzed (Participants) | 1 | 0 | 1
  Month 114 | -0.13 (0) |  | -0.13 (0)

14. Secondary Outcome: Extension Period: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Month 3, 6, 9 and 12
Description: HAQ-DI assesses the degree of difficulty a participant has experienced during the past week in 8 categories of daily living activities: dressing/grooming; arising; eating; walking; reach; grip; hygiene; and other activities. Each activity category consisted of 2-3 questionnaire. Each questionnaire was scored on a 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Any activity that required assistance from another individual or required the use of an assistive device was adjusted to a score of 2 to represent a more limited functional status. Overall score was computed as the sum of total scores divided by the number of questionnaire answered. Total possible HAQ-DI score range: 0 (least difficulty) and 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities.
Time Frame: Baseline (Month 0 at the entry of Initial Period); Month 3, 6, 9, and 12 of Extension Period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Extension Period: Tofacitinib 5 mg
Number analyzed (Participants) | 48
Units on a scale
  Baseline | 1.35 (0.63)
  Change at Month 3: number analyzed (Participants) | 46
  Change at Month 3 | -0.48 (0.58)
  Change at Month 6: number analyzed (Participants) | 35
  Change at Month 6 | -0.55 (0.65)
  Change at Month 9: number analyzed (Participants) | 15
  Change at Month 9 | -0.58 (0.70)
  Change at Month 12: number analyzed (Participants) | 2
  Change at Month 12 | -1.50 (1.94)

15. Secondary Outcome: Initial Period: Short-Form-36 Health Survey (SF-36) Score
Description: Change from Baseline for Physical Component and Mental Component Scores by visit. SF-36 is a health status measure of 8 general health domains, each scored on a 0 to 100 scale: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. These domains can be summarized as physical and mental component scores. The domain scores were "normed" and the resulting component scores treated as Z-scores with a scale of negative to positive infinity. A higher score implies less disease. The greater the change from baseline, the greater the improvement. The stated number of participants analyzed was the total number of participants in each group. The actual number of participants analyzed on each occasion varied, and is provided for each visit presented.
Time Frame: Every visit until study completion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib
Number analyzed (Participants) | 1123 | 3358 | 4481
Scores on scale
  Physical Component Month 3: number analyzed (Participants) | 983 | 2693 | 3676
  Physical Component Month 3 | 7.90 (8.70) | 8.85 (8.92) | 8.60 (8.87)
  Physical Component Month 6: number analyzed (Participants) | 961 | 2629 | 3590
  Physical Component Month 6 | 8.10 (8.94) | 9.02 (9.11) | 8.77 (9.07)
  Physical Component Month 9: number analyzed (Participants) | 534 | 2499 | 3033
  Physical Component Month 9 | 8.60 (9.07) | 8.80 (9.20) | 8.77 (9.18)
  Physical Component Month 12: number analyzed (Participants) | 903 | 2449 | 3352
  Physical Component Month 12 | 8.44 (8.53) | 8.78 (9.26) | 8.69 (9.07)
  Physical Component Month 15: number analyzed (Participants) | 733 | 2324 | 3057
  Physical Component Month 15 | 8.43 (8.88) | 8.98 (9.05) | 8.85 (9.01)
  Physical Component Month 18: number analyzed (Participants) | 855 | 2188 | 3043
  Physical Component Month 18 | 8.14 (8.89) | 8.99 (9.18) | 8.75 (9.11)
  Physical Component Month 21: number analyzed (Participants) | 767 | 2005 | 2772
  Physical Component Month 21 | 8.00 (8.70) | 8.85 (8.96) | 8.62 (8.90)
  Physical Component Month 24: number analyzed (Participants) | 797 | 2102 | 2899
  Physical Component Month 24 | 8.28 (8.73) | 9.00 (9.30) | 8.80 (9.15)
  Physical Component Month 27: number analyzed (Participants) | 739 | 1663 | 2402
  Physical Component Month 27 | 8.41 (8.84) | 8.64 (9.16) | 8.57 (9.06)
  Physical Component Month 30: number analyzed (Participants) | 708 | 1566 | 2274
  Physical Component Month 30 | 7.78 (8.81) | 8.56 (9.06) | 8.32 (8.99)
  Physical Component Month 33: number analyzed (Participants) | 682 | 1444 | 2126
  Physical Component Month 33 | 8.17 (8.87) | 8.39 (9.31) | 8.32 (9.17)
  Physical Component Month 36: number analyzed (Participants) | 676 | 1530 | 2206
  Physical Component Month 36 | 8.31 (8.97) | 8.43 (9.22) | 8.40 (9.14)
  Physical Component Month 39: number analyzed (Participants) | 609 | 1176 | 1785
  Physical Component Month 39 | 8.05 (9.26) | 8.13 (9.14) | 8.10 (9.18)
  Physical Component Month 42: number analyzed (Participants) | 573 | 923 | 1496
  Physical Component Month 42 | 7.81 (9.32) | 8.07 (9.13) | 7.97 (9.21)
  Physical Component Month 45: number analyzed (Participants) | 540 | 652 | 1192
  Physical Component Month 45 | 8.40 (9.87) | 8.33 (9.40) | 8.36 (9.61)
  Physical Component Month 48: number analyzed (Participants) | 537 | 1044 | 1581
  Physical Component Month 48 | 8.12 (9.56) | 8.27 (9.23) | 8.22 (9.34)
  Physical Component Month 51: number analyzed (Participants) | 417 | 304 | 721
  Physical Component Month 51 | 7.88 (9.69) | 8.55 (9.70) | 8.16 (9.69)
  Physical Component Month 54: number analyzed (Participants) | 396 | 175 | 571
  Physical Component Month 54 | 7.72 (9.41) | 8.82 (9.47) | 8.06 (9.43)
  Physical Component Month 57: number analyzed (Participants) | 372 | 105 | 477
  Physical Component Month 57 | 7.57 (9.72) | 8.12 (9.69) | 7.69 (9.71)
  Physical Component Month 60: number analyzed (Participants) | 371 | 259 | 630
  Physical Component Month 60 | 7.94 (9.74) | 9.29 (9.43) | 8.49 (9.63)
  Physical Component Month 63: number analyzed (Participants) | 345 | 68 | 413
  Physical Component Month 63 | 7.73 (9.76) | 7.90 (8.98) | 7.76 (9.63)
  Physical Component Month 66: number analyzed (Participants) | 327 | 56 | 383
  Physical Component Month 66 | 7.92 (9.41) | 7.58 (7.88) | 7.87 (9.20)
  Physical Component Month 69: number analyzed (Participants) | 267 | 40 | 307
  Physical Component Month 69 | 7.68 (9.32) | 9.12 (7.06) | 7.87 (9.06)
  Physical Component Month 72: number analyzed (Participants) | 316 | 54 | 370
  Physical Component Month 72 | 7.90 (9.93) | 8.70 (10.24) | 8.02 (9.97)
  Physical Component Month 75: number analyzed (Participants) | 84 | 12 | 96
  Physical Component Month 75 | 9.03 (10.96) | 5.75 (9.05) | 8.62 (10.75)
  Physical Component Month 78: number analyzed (Participants) | 55 | 7 | 62
  Physical Component Month 78 | 10.22 (11.10) | 7.39 (7.09) | 9.90 (10.72)
  Physical Component Month 81: number analyzed (Participants) | 49 | 4 | 53
  Physical Component Month 81 | 10.51 (10.17) | 7.90 (13.05) | 10.31 (10.28)
  Physical Component Month 84: number analyzed (Participants) | 93 | 11 | 104
  Physical Component Month 84 | 8.93 (11.56) | 7.14 (8.01) | 8.74 (11.22)
  Physical Component Month 87: number analyzed (Participants) | 26 | 2 | 28
  Physical Component Month 87 | 11.92 (10.49) | 15.23 (3.64) | 12.16 (10.15)
  Physical Component Month 90: number analyzed (Participants) | 12 | 1 | 13
  Physical Component Month 90 | 13.50 (10.98) | 16.50 (0) | 13.73 (10.55)
  Physical Component Month 93: number analyzed (Participants) | 1 | 0 | 1
  Physical Component Month 93 | 26.71 (0) |  | 26.71 (0)
  Physical Component Month 96: number analyzed (Participants) | 5 | 0 | 5
  Physical Component Month 96 | 4.61 (9.75) |  | 4.61 (9.75)
  Physical Component Month 99: number analyzed (Participants) | 1 | 0 | 1
  Physical Component Month 99 | -8.26 (0) |  | -8.26 (0)
  Mental Component Month 3: number analyzed (Participants) | 983 | 2693 | 3676
  Mental Component Month 3 | 4.37 (10.88) | 4.91 (11.18) | 4.77 (11.10)
  Mental Component Month 6: number analyzed (Participants) | 961 | 2629 | 3590
  Mental Component Month 6 | 3.94 (10.85) | 4.81 (11.12) | 4.58 (11.06)
  Mental Component Month 9: number analyzed (Participants) | 534 | 2499 | 3033
  Mental Component Month 9 | 4.65 (10.78) | 5.04 (11.17) | 4.97 (11.10)
  Mental Component Month 12: number analyzed (Participants) | 903 | 2449 | 3352
  Mental Component Month 12 | 3.77 (11.03) | 4.81 (11.43) | 4.53 (11.33)
  Mental Component Month 15: number analyzed (Participants) | 733 | 2324 | 3057
  Mental Component Month 15 | 4.14 (11.21) | 4.79 (11.52) | 4.63 (11.45)
  Mental Component Month 18: number analyzed (Participants) | 855 | 2188 | 3043
  Mental Component Month 18 | 4.12 (11.11) | 4.87 (11.41) | 4.66 (11.33)
  Mental Component Month 21: number analyzed (Participants) | 767 | 2005 | 2772
  Mental Component Month 21 | 4.21 (11.08) | 4.87 (11.22) | 4.68 (11.18)
  Mental Component Month 24: number analyzed (Participants) | 797 | 2102 | 2899
  Mental Component Month 24 | 4.12 (11.06) | 5.08 (11.32) | 4.82 (11.26)
  Mental Component Month 27: number analyzed (Participants) | 739 | 1663 | 2402
  Mental Component Month 27 | 3.67 (10.53) | 4.91 (11.28) | 4.53 (11.07)
  Mental Component Month 30: number analyzed (Participants) | 708 | 1566 | 2274
  Mental Component Month 30 | 3.58 (11.14) | 4.68 (11.71) | 4.34 (11.54)
  Mental Component Month 33: number analyzed (Participants) | 682 | 1444 | 2126
  Mental Component Month 33 | 3.91 (10.65) | 4.82 (11.74) | 4.53 (11.40)
  Mental Component Month 36: number analyzed (Participants) | 676 | 1530 | 2206
  Mental Component Month 36 | 3.83 (10.94) | 4.81 (11.60) | 4.51 (11.40)
  Mental Component Month 39: number analyzed (Participants) | 609 | 1176 | 1785
  Mental Component Month 39 | 3.60 (11.02) | 4.59 (11.75) | 4.25 (11.51)
  Mental Component Month 42: number analyzed (Participants) | 573 | 923 | 1496
  Mental Component Month 42 | 3.23 (11.40) | 4.55 (11.63) | 4.04 (11.56)
  Mental Component Month 45: number analyzed (Participants) | 540 | 652 | 1192
  Mental Component Month 45 | 3.16 (11.63) | 4.40 (11.64) | 3.83 (11.56)
  Mental Component Month 48: number analyzed (Participants) | 537 | 1044 | 1581
  Mental Component Month 48 | 3.48 (11.71) | 4.73 (11.83) | 4.31 (11.80)
  Mental Component Month 51: number analyzed (Participants) | 417 | 304 | 721
  Mental Component Month 51 | 3.61 (12.12) | 4.83 (11.82) | 4.13 (12.00)
  Mental Component Month 54: number analyzed (Participants) | 396 | 175 | 571
  Mental Component Month 54 | 3.44 (11.77) | 6.49 (12.67) | 4.38 (12.12)
  Mental Component Month 57: number analyzed (Participants) | 372 | 105 | 477
  Mental Component Month 57 | 3.24 (12.24) | 5.10 (11.74) | 3.65 (12.15)
  Mental Component Month 60: number analyzed (Participants) | 371 | 259 | 630
  Mental Component Month 60 | 3.05 (12.06) | 5.18 (12.22) | 3.93 (12.16)
  Mental Component Month 63: number analyzed (Participants) | 345 | 68 | 413
  Mental Component Month 63 | 3.04 (11.61) | 4.22 (10.32) | 3.23 (11.40)
  Mental Component Month 66: number analyzed (Participants) | 327 | 56 | 383
  Mental Component Month 66 | 2.96 (11.32) | 3.47 (8.33) | 3.04 (10.93)
  Mental Component Month 69: number analyzed (Participants) | 267 | 40 | 307
  Mental Component Month 69 | 3.90 (12.35) | 4.90 (9.84) | 4.03 (12.04)
  Mental Component Month 72: number analyzed (Participants) | 316 | 54 | 370
  Mental Component Month 72 | 3.78 (11.48) | 5.32 (12.80) | 4.00 (11.68)
  Mental Component Month 75: number analyzed (Participants) | 84 | 12 | 96
  Mental Component Month 75 | 5.04 (12.22) | 1.52 (11.38) | 4.60 (12.12)
  Mental Component Month 78: number analyzed (Participants) | 55 | 7 | 62
  Mental Component Month 78 | 4.12 (13.37) | 1.05 (13.28) | 3.77 (13.29)
  Mental Component Month 81: number analyzed (Participants) | 49 | 4 | 53
  Mental Component Month 81 | 6.09 (10.40) | 2.60 (14.75) | 5.83 (10.64)
  Mental Component Month 84: number analyzed (Participants) | 93 | 11 | 104
  Mental Component Month 84 | 5.73 (13.07) | -2.36 (11.63) | 4.87 (13.11)
  Mental Component Month 87: number analyzed (Participants) | 26 | 2 | 28
  Mental Component Month 87 | 7.52 (13.03) | 16.93 (2.66) | 8.19 (12.79)
  Mental Component Month 90: number analyzed (Participants) | 12 | 1 | 13
  Mental Component Month 90 | 4.61 (11.75) | 18.75 (0) | 5.65 (11.86)
  Mental Component Month 93: number analyzed (Participants) | 1 | 0 | 1
  Mental Component Month 93 | 14.03 (0) |  | 14.03 (0)
  Mental Component Month 96: number analyzed (Participants) | 5 | 0 | 5
  Mental Component Month 96 | 7.58 (9.73) |  | 7.58 (9.73)
  Mental Component Month 99: number analyzed (Participants) | 1 | 0 | 1
  Mental Component Month 99 | 22.28 (0) |  | 22.28 (0)

16. Secondary Outcome: Initial Period: FACIT Fatigue Scale, EuroQol EQ 5D, Work Limitations Questionnaire, and RA Healthcare Resource Utilization Questionnaire (RA-HCRU)
Description: Change from Baseline Scores for each: FACIT Fatigue Scale (score range 0 to 52, higher score indicates higher quality of life and an increase from baseline score indicates improvement), EuroQol EQ 5D (index values derived from a measure of central tendency and a measure of dispersion, an increase from baseline indicates improvement, score range 0 to 1), Work Limitations (WL) Physical Demands (covers ability to perform job tasks that involve bodily strength, a decrease from baseline indicates improvement, score range 0 to 100, higher scores indicating greater limitation), and RA Healthcare Resource Utilization Work Performance in Past 3 Months on Days Bothered by RA (assesses healthcare use over previous 3 months, a decrease from baseline indicates improvement, score range 0 to 10).
  The stated number of participants analyzed was the total number of participants in each group. The actual number of participants analyzed on each occasion varied, and is provided for each visit presented.
Time Frame: Every visit until study completion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib
Number analyzed (Participants) | 1123 | 3358 | 4481
Scores on a scale
  FACIT Month 6: number analyzed (Participants) | 370 | 2544 | 2914
  FACIT Month 6 | 6.29 (8.98) | 7.33 (10.57) | 7.19 (10.39)
  FACIT Month 12: number analyzed (Participants) | 582 | 2396 | 2978
  FACIT Month 12 | 5.98 (9.74) | 7.33 (10.56) | 7.06 (10.41)
  FACIT Month 18: number analyzed (Participants) | 729 | 2168 | 2897
  FACIT Month 18 | 6.14 (10.06) | 7.40 (10.65) | 7.09 (10.51)
  FACIT Month 24: number analyzed (Participants) | 704 | 2053 | 2757
  FACIT Month 24 | 5.90 (9.76) | 7.42 (10.56) | 7.03 (10.38)
  FACIT Month 30: number analyzed (Participants) | 618 | 1525 | 2143
  FACIT Month 30 | 5.36 (10.08) | 7.00 (10.91) | 6.52 (10.70)
  FACIT Month 36: number analyzed (Participants) | 589 | 1497 | 2086
  FACIT Month 36 | 5.95 (9.87) | 6.87 (10.94) | 6.61 (10.66)
  FACIT Month 42: number analyzed (Participants) | 491 | 898 | 1389
  FACIT Month 42 | 5.35 (10.36) | 6.83 (10.86) | 6.31 (10.71)
  FACIT Month 48: number analyzed (Participants) | 464 | 1025 | 1489
  FACIT Month 48 | 6.01 (10.33) | 6.88 (10.95) | 6.61 (10.77)
  FACIT Month 54: number analyzed (Participants) | 330 | 169 | 499
  FACIT Month 54 | 6.16 (10.49) | 8.51 (11.58) | 6.96 (10.92)
  FACIT Month 60: number analyzed (Participants) | 318 | 256 | 574
  FACIT Month 60 | 5.96 (10.69) | 8.88 (11.65) | 7.27 (11.21)
  FACIT Month 66: number analyzed (Participants) | 277 | 55 | 332
  FACIT Month 66 | 5.64 (10.93) | 6.67 (10.58) | 5.81 (10.86)
  FACIT Month 72: number analyzed (Participants) | 272 | 51 | 323
  FACIT Month 72 | 5.73 (11.10) | 8.63 (10.71) | 6.18 (11.07)
  FACIT Month 78: number analyzed (Participants) | 32 | 7 | 39
  FACIT Month 78 | 12.06 (11.15) | 0.71 (14.84) | 10.03 (12.48)
  FACIT Month 84: number analyzed (Participants) | 74 | 11 | 85
  FACIT Month 84 | 9.13 (12.88) | 2.91 (12.36) | 8.32 (12.91)
  FACIT Month 90: number analyzed (Participants) | 6 | 1 | 7
  FACIT Month 90 | 18.67 (9.14) | 10.00 (0) | 17.43 (8.96)
  FACIT Month 96: number analyzed (Participants) | 3 | 0 | 3
  FACIT Month 96 | 6.00 (2.65) |  | 6.00 (2.65)
  EuroQol Month 6: number analyzed (Participants) | 323 | 2021 | 2344
  EuroQol Month 6 | 0.20 (0.31) | 0.22 (0.32) | 0.22 (0.32)
  EuroQol Month 12: number analyzed (Participants) | 538 | 1897 | 2435
  EuroQol Month 12 | 0.22 (0.30) | 0.22 (0.33) | 0.22 (0.32)
  EuroQol Month 18: number analyzed (Participants) | 684 | 1748 | 2432
  EuroQol Month 18 | 0.20 (0.32) | 0.23 (0.33) | 0.22 (0.33)
  EuroQol Month 24: number analyzed (Participants) | 664 | 1619 | 2283
  EuroQol Month 24 | 0.20 (0.31) | 0.23 (0.33) | 0.22 (0.32)
  EuroQol Month 30: number analyzed (Participants) | 616 | 1456 | 2072
  EuroQol Month 30 | 0.19 (0.31) | 0.22 (0.33) | 0.21 (0.32)
  EuroQol Month 36: number analyzed (Participants) | 582 | 1397 | 1979
  EuroQol Month 36 | 0.21 (0.30) | 0.23 (0.33) | 0.22 (0.32)
  EuroQol Month 42: number analyzed (Participants) | 483 | 874 | 1357
  EuroQol Month 42 | 0.18 (0.31) | 0.24 (0.33) | 0.22 (0.32)
  EuroQol Month 48: number analyzed (Participants) | 464 | 1010 | 1474
  EuroQol Month 48 | 0.19 (0.31) | 0.23 (0.33) | 0.22 (0.32)
  EuroQol Month 54: number analyzed (Participants) | 330 | 167 | 497
  EuroQol Month 54 | 0.22 (0.32) | 0.32 (0.36) | 0.22 (0.32)
  EuroQol Month 60: number analyzed (Participants) | 317 | 255 | 572
  EuroQol Month 60 | 0.20 (0.33) | 0.27 (0.35) | 0.23 (0.34)
  EuroQol Month 66: number analyzed (Participants) | 276 | 53 | 329
  EuroQol Month 66 | 0.21 (0.33) | 0.24 (0.34) | 0.21 (0.33)
  EuroQol Month 72: number analyzed (Participants) | 273 | 50 | 323
  EuroQol Month 72 | 0.22 (0.32) | 0.28 (0.35) | 0.23 (0.32)
  EuroQol Month 78: number analyzed (Participants) | 32 | 7 | 39
  EuroQol Month 78 | 0.36 (0.37) | 0.10 (0.51) | 0.31 (0.40)
  EuroQol Month 84: number analyzed (Participants) | 75 | 11 | 86
  EuroQol Month 84 | 0.27 (0.35) | 0.21 (0.43) | 0.27 (0.36)
  EuroQol Month 90: number analyzed (Participants) | 6 | 1 | 7
  EuroQol Month 90 | 0.47 (0.32) | 0.84 (0) | 0.52 (0.32)
  EuroQol Month 96: number analyzed (Participants) | 3 | 0 | 3
  EuroQol Month 96 | 0.09 (0.04) |  | 0.09 (0.04)
  WL: Physical Demands Month 6: number analyzed (Participants) | 109 | 900 | 1009
  WL: Physical Demands Month 6 | -5.34 (39.81) | -3.67 (38.17) | -3.85 (38.33)
  WL: Physical Demands Month 12: number analyzed (Participants) | 96 | 808 | 904
  WL: Physical Demands Month 12 | -5.31 (37.81) | -4.02 (39.25) | -4.16 (39.08)
  WL: Physical Demands Month 18: number analyzed (Participants) | 83 | 706 | 789
  WL: Physical Demands Month 18 | -7.97 (35.46) | -2.29 (37.48) | -2.89 (37.29)
  WL: Physical Demands Month 24: number analyzed (Participants) | 63 | 544 | 607
  WL: Physical Demands Month 24 | -2.62 (36.05) | -4.46 (37.54) | -4.27 (37.36)
  WL: Physical Demands Month 30: number analyzed (Participants) | 51 | 444 | 495
  WL: Physical Demands Month 30 | -10.12 (37.17) | -3.75 (37.67) | -4.41 (37.63)
  WL: Physical Demands Month 36: number analyzed (Participants) | 35 | 350 | 385
  WL: Physical Demands Month 36 | -7.31 (34.69) | -3.95 (39.58) | -4.25 (39.14)
  WL: Physical Demands Month 42: number analyzed (Participants) | 24 | 246 | 270
  WL: Physical Demands Month 42 | -13.51 (33.91) | -4.81 (38.98) | -5.58 (38.58)
  WL: Physical Demands Month 48: number analyzed (Participants) | 19 | 126 | 145
  WL: Physical Demands Month 48 | -25.86 (34.47) | 0.73 (38.68) | -2.76 (39.09)
  WL: Physical Demands Month 54: number analyzed (Participants) | 2 | 20 | 22
  WL: Physical Demands Month 54 | -39.17 (62.46) | -13.27 (45.69) | -15.63 (46.18)
  WL: Physical Demands Month 60: number analyzed (Participants) | 0 | 3 | 3
  WL: Physical Demands Month 60 |  | -27.78 (34.94) | -27.78 (34.94)
  WL: Physical Demands Month 66: number analyzed (Participants) | 0 | 1 | 1
  WL: Physical Demands Month 66 |  | 8.33 (0) | 8.33 (0)
  RA-HCRU Month 6: number analyzed (Participants) | 189 | 1419 | 1608
  RA-HCRU Month 6 | -2.01 (6.20) | -2.08 (4.15) | -2.07 (4.44)
  RA-HCRU Month 12: number analyzed (Participants) | 180 | 1329 | 1509
  RA-HCRU Month 12 | -2.41 (6.43) | -2.26 (3.76) | -2.28 (4.17)
  RA-HCRU Month 18: number analyzed (Participants) | 161 | 1162 | 1323
  RA-HCRU Month 18 | -1.88 (2.93) | -2.24 (3.90) | -2.19 (3.80)
  RA-HCRU Month 24: number analyzed (Participants) | 162 | 1101 | 1263
  RA-HCRU Month 24 | -2.03 (3.18) | -2.22 (3.26) | -2.19 (3.25)
  RA-HCRU Month 30: number analyzed (Participants) | 126 | 785 | 911
  RA-HCRU Month 30 | -1.67 (3.02) | -2.16 (4.17) | -2.10 (4.04)
  RA-HCRU Month 36: number analyzed (Participants) | 106 | 759 | 865
  RA-HCRU Month 36 | -2.38 (2.91) | -2.32 (4.14) | -2.33 (4.01)
  RA-HCRU Month 42: number analyzed (Participants) | 68 | 455 | 523
  RA-HCRU Month 42 | -1.68 (2.84) | -2.18 (4.70) | -2.11 (4.51)
  RA-HCRU Month 48: number analyzed (Participants) | 66 | 527 | 593
  RA-HCRU Month 48 | -1.88 (3.24) | -2.15 (4.67) | -2.12 (4.53)
  RA-HCRU Month 54: number analyzed (Participants) | 3 | 39 | 42
  RA-HCRU Month 54 | -2.00 (1.00) | -2.59 (3.42) | -2.55 (3.30)
  RA-HCRU Month 60: number analyzed (Participants) | 4 | 94 | 98
  RA-HCRU Month 60 | -2.00 (3.56) | -2.88 (2.85) | -2.85 (2.87)
  RA-HCRU Month 66: number analyzed (Participants) | 0 | 0 | 0
  RA-HCRU Month 72: number analyzed (Participants) | 0 | 4 | 4
  RA-HCRU Month 72 |  | -1.25 (6.70) | -1.25 (6.70)
  RA-HCRU Month 78: number analyzed (Participants) | 0 | 0 | 0
  RA-HCRU Month 84: number analyzed (Participants) | 0 | 0 | 0
  RA-HCRU Month 90: number analyzed (Participants) | 0 | 0 | 0
  RA-HCRU Month 96: number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Initial Period: Preservation of Joint Structure in Participants Who Had Baseline Radiographs Obtained in Their Qualifying Index Study
Description: Modified Total Sharp Score per visit. Baseline score was the last available assessment from the index study. The Modified Total Sharp Score measures disease progression; increased scores indicate disease progression. Score range 0 (normal) to 448 (worst possible total score). The stated number of participants analyzed was the total number of participants in each group. The actual number of participants analyzed on each occasion varied, and is provided for each visit presented.
  TSS=Total Sharp Score
Time Frame: Every 6 months until study completion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib
Number analyzed (Participants) | 1123 | 3358 | 4481
Scores on a scale
  Modified TSS Baseline: number analyzed (Participants) | 95 | 1061 | 1156
  Modified TSS Baseline | 20.55 (33.37) | 24.13 (43.57) | 23.84 (42.83)
  Modified TSS Month 6: number analyzed (Participants) | 82 | 937 | 1019
  Modified TSS Month 6 | 22.58 (35.10) | 25.12 (44.42) | 24.91 (43.74)
  Modified TSS Month 12: number analyzed (Participants) | 85 | 918 | 1003
  Modified TSS Month 12 | 21.26 (33.75) | 24.73 (44.08) | 24.44 (43.30)
  Modified TSS Month 24: number analyzed (Participants) | 77 | 801 | 878
  Modified TSS Month 24 | 22.07 (35.85) | 24.85 (43.21) | 24.61 (42.61)
  Modified TSS Month 36: number analyzed (Participants) | 35 | 379 | 414
  Modified TSS Month 36 | 25.88 (37.74) | 28.22 (44.95) | 28.02 (44.35)

18. Secondary Outcome: Vaccine Sub-study. Percent Achieving a Satisfactory Humoral Response to the Pneumococcal Vaccine as Defined by ≥ 2-fold Increase in Antibody Concentrations
Description: Number (%) of participants achieving a satisfactory humoral response to the pneumococcal vaccine as defined by ≥2-fold increase in antibody concentration from vaccine sub-study visit 2 (vaccination baseline) in ≥6 of 12 anti-pneumococcal antigens (serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) The number of participants was the number with a determinate antibody titer to the given vaccine antigen within the population.
  95% CI is based on Clopper-Pearson exact method for response rate.
Time Frame: From vaccine sub-study visit 2 (baseline) to sub-study visit 4
Population: Evaluable Immunogenicity Population
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Tofacitinib 10 mg BID Continuous Visit 3; Tofacitinib 10 mg BID Continuous Visit 4: Participants receiving continuous tofacitinib treatment
- Tofacitinib 10 mg BID Interrupted Visit 3; Tofacitinib 10 mg BID Interrupted Visit 4: Participants whose treatment with tofacitinib was interrupted for 2 weeks post-randomization
Arm/Group | Tofacitinib 10 mg BID Continuous Visit 3 | Tofacitinib 10 mg BID Interrupted Visit 3 | Tofacitinib 10 mg BID Continuous Visit 4 | Tofacitinib 10 mg BID Interrupted Visit 4
Number analyzed (Participants) | 91 | 91 | 92 | 91
Percent of participants | 18.7 [11.3 to 28.2] | 38.5 [28.4 to 49.2] | 75.0 [64.9 to 83.4] | 84.6 [75.5 to 91.3]

19. Secondary Outcome: Vaccine Sub-study. Percent Achieving a Satisfactory Humoral Response to the Seasonal Influenza Vaccine as Defined by ≥ 4-fold Increase in Antibody Titers
Description: Number of participants achieving a satisfactory humoral response to the seasonal influenza vaccine as defined by ≥4-fold increase in antibody titers from visit 2 (vaccination baseline) in ≥2 of 3 influenza antigens (HAI B, HAI H1N1, and HAI H3N2) The number of participants was the number with a determinate antibody titer to the given vaccine antigen within the population.
  95% CI is based on Clopper-Pearson exact method for response rate.
Time Frame: From vaccine sub-study visit 2 (baseline) to sub-study visit 4
Population: Evaluable Immunogenicity Population
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Tofacitinib 10 mg BID Continuous Visit 3 | Tofacitinib 10 mg BID Interrupted Visit 3 | Tofacitinib 10 mg BID Continuous Visit 4 | Tofacitinib 10 mg BID Interrupted Visit 4
Number analyzed (Participants) | 91 | 91 | 92 | 91
Percent of participants | 31.9 [22.5 to 42.5] | 53.8 [43.1 to 64.4] | 66.3 [55.7 to 75.8] | 63.7 [53.0 to 73.6]

20. Secondary Outcome: Vaccine Sub-study. Percentage of Participants Achieving Protective Antibody Titers to the Seasonal Influenza Vaccine as Measured by a Hemagglutination Inhibition (HI) Assay Titer of ≥ 1:40 in ≥ 2 of 3 Influenza Antigens at Vaccine Sub-study Visit 3 and 4
Description: Number (%) of participants achieving protective antibody titers to the seasonal influenza vaccine as measured by an HAI assay titer of ≥1:40 in ≥2 of 3 influenza antigens measured at vaccine sub-study visits 3 and 4.
  The number of participants was the number with a determinate antibody titer to the given vaccine antigen within the population.
  95% CI is based on Clopper-Pearson exact method for response rate.
Time Frame: From vaccine sub-study visit 2 (baseline) to sub-study visit 4
Population: Evaluable Immunogenicity Population
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Tofacitinib 10 mg BID Continuous Visit 3 | Tofacitinib 10 mg BID Interrupted Visit 3 | Tofacitinib 10 mg BID Continuous Visit 4 | Tofacitinib 10 mg BID Interrupted Visit 4
Number analyzed (Participants) | 91 | 91 | 92 | 91
Percent of participants | 56.0 [45.2 to 66.4] | 69.2 [58.7 to 78.5] | 75.0 [64.9 to 83.4] | 82.4 [73.0 to 89.6]

21. Secondary Outcome: Vaccine Sub-study. Percentage of Participants Who Respond to Each of the 12 Pneumococcal Antigens as Defined by ≥ 2-fold Increase in Antibody Concentrations From Vaccine Sub-study Visit 2 (Vaccination Baseline) Measured at Vaccine Sub-study Visit 4
Description: as for outcome 18
Time Frame: From vaccine sub-study visit 2 (baseline) to sub-study visit 4
Population: Evaluable Immunogenicity Population
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Tofacitinib 10 mg BID Continuous: Participants receiving continuous tofacitinib treatment
- Tofacitinib 10 mg BID Interrupted: Participants whose treatment with tofacitinib was interrupted for 2 weeks post-randomization
Arm/Group | Tofacitinib 10 mg BID Continuous | Tofacitinib 10 mg BID Interrupted
Number analyzed (Participants) | 92 | 91
Percent of participants
  Serotype 1 | 75 [64.9 to 83.4] | 82.4 [73.0 to 89.6]
  Serotype 3 | 53.3 [42.6 to 63.7] | 71.4 [61.0 to 80.4]
  Serotype 4 | 76.1 [66.1 to 84.4] | 76.9 [66.9 to 85.1]
  Serotype 5 | 42.4 [32.1 to 53.1] | 49.5 [38.8 to 60.1]
  Serotype 6B | 48.9 [38.3 to 59.6] | 56 [45.2 to 66.4]
  Serotype 7F | 71.7 [61.4 to 80.6] | 78 [68.1 to 86.0]
  Serotype 9V | 64.1 [53.5 to 73.9] | 78 [68.1 to 86.0]
  Serotype 14 | 71.7 [61.4 to 80.6] | 75.8 [65.7 to 84.2]
  Serotype 18C | 73.9 [63.7 to 82.5] | 83.5 [74.3 to 90.5]
  Serotype 19A | 54.3 [43.6 to 64.8] | 56.0 [45.2 to 66.4]
  Serotype 19F | 60.9 [50.1 to 70.9] | 71.4 [61.0 to 80.4]
  Serotype 23F | 53.3 [42.6 to 63.7] | 70.3 [59.8 to 79.5]

22. Secondary Outcome: Vaccine Sub-study. Percentage of Participants Who Respond to Each of the 3 Influenza Antigens as Defined by ≥ 4-fold Increase in Antibody Titers From Vaccine Sub-study Visit 2 (Vaccination Baseline) Measured at Vaccine Sub-study Visit 4
Description: Number (%) of participants achieving a satisfactory humoral response to the seasonal influenza vaccine defined as ≥4-fold increase in antibody titers from visit 2 (vaccination baseline) in ≥2 of 3 influenza antigens (HAI B, HAI H1N1, and HAI H3N2).
  The number of participants was the number with a determinate antibody titer to the given vaccine antigen within the population.
  95% CI is based on Clopper-Pearson exact method for response rate.
Time Frame: From vaccine sub-study visit 2 (baseline) to sub-study visit 4
Population: Evaluable Immunogenicity Population
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Tofacitinib 10 mg BID Continuous Visit 4 | Tofacitinib 10 mg BID Interrupted Visit 4
Number analyzed (Participants) | 92 | 91
Percent of participants
  Antigen B | 45.7 [35.2 to 56.4] | 51.6 [40.9 to 62.3]
  Antigen H1N1 | 71.7 [61.4 to 80.6] | 63.7 [53.0 to 73.6]
  Antigen H3N2 | 66.3 [55.7 to 75.8] | 74.7 [64.5 to 83.3]

23. Secondary Outcome: Vaccine Sub-study. Fold Increase of Anti-pneumococcal Antibody Levels to Each of the 12 Pneumococcal Antigens Above Vaccination Baseline Values (Vaccine Sub-study Visit 2) at Vaccine Sub-study Visit 4
Description: Geometric Mean Fold Increase From Baseline of Pneumococcal Antigens Measured at Visit 4.
  n was the number of participants with valid and determinate assay results for the specified serotype at the given visit.
  The stated number of participants analyzed was the total number of participants. The actual number of participants analyzed for some serotypes varied, and is provided where it differed from the total number of participants.
  Confidence Intervals (CIs) were back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: From vaccine sub-study visit 2 (baseline) to sub-study visit 4
Population: Evaluable Immunogenicity Population
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change in Antibody Level
Groups:
- Tofacitinib 10 mg Continuous: Participants receiving continuous tofacitinib treatment
Arm/Group | Tofacitinib 10 mg Continuous | Tofacitinib 10 mg BID Interrupted
Number analyzed (Participants) | 92 | 91
Fold Change in Antibody Level
  Serotype 1: number analyzed (Participants) | 89 | 86
  Serotype 1 | 5.87 [4.57 to 7.55] | 9.26 [6.89 to 12.44]
  Serotype 3: number analyzed (Participants) | 91 | 89
  Serotype 3 | 2.34 [1.97 to 2.79] | 4.20 [3.31 to 5.32]
  Serotype 4: number analyzed (Participants) | 91 | 89
  Serotype 4 | 5.32 [4.22 to 6.71] | 6.29 [4.65 to 8.51]
  Serotype 5 | 2.02 [1.75 to 2.34] | 2.53 [2.12 to 3.02]
  Serotype 6B | 2.32 [1.98 to 2.73] | 3.06 [2.53 to 3.69]
  Serotype 7F: number analyzed (Participants) | 92 | 89
  Serotype 7F | 4.69 [3.73 to 5.90] | 6.41 [4.97 to 8.28]
  Serotype 9V: number analyzed (Participants) | 92 | 90
  Serotype 9V | 3.17 [2.70 to 3.72] | 4.39 [3.62 to 5.34]
  Serotype 14 | 5.23 [4.00 to 6.86] | 7.34 [5.50 to 9.79]
  Serotype 18C | 3.97 [3.28 to 4.79] | 7.41 [5.77 to 9.53]
  Serotype 19A | 2.33 [1.99 to 2.72] | 2.93 [2.46 to 3.50]
  Serotype 19F: number analyzed (Participants) | 90 | 90
  Serotype 19F | 2.97 [2.44 to 3.62] | 4.60 [3.64 to 5.80]
  Serotype 23F: number analyzed (Participants) | 92 | 90
  Serotype 23F | 2.74 [2.27 to 3.32] | 4.54 [3.58 to 5.75]

24. Secondary Outcome: Vaccine Sub-study. Fold Increase of Anti-influenza Antibody Levels to Each of the 3 Influenza Antigens Above Vaccination Baseline Values (Vaccine Sub-study Visit 2) at Vaccine Sub-study Visit 4
Description: Geometric Mean Fold Increase From Baseline of Influenza Antigens Measured at Visit 4.
  n was the number of participants with valid and determinate assay results for the specified HAI strain at the given visit.
  Confidence Intervals (CIs) were back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: From vaccine sub-study visit 2 (baseline) to sub-study visit 4
Population: Evaluable Immunogenicity Population
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change in Antibody Level
Arm/Group | Tofacitinib 10 mg BID Continuous | Tofacitinib 10 mg BID Interrupted
Number analyzed (Participants) | 92 | 91
Fold Change in Antibody Level
  Antigen B | 3.33 [2.57 to 4.32] | 4.17 [3.25 to 5.34]
  Antigen H1N1 | 7.94 [5.96 to 10.58] | 6.71 [4.94 to 9.12]
  Antigen H3N2 | 7.80 [5.58 to 10.91] | 8.51 [6.45 to 11.21]

25. Secondary Outcome: Vaccine Sub-study. Concentrations of Anti-pneumococcal Antibodies at Vaccine Sub-study Visit 3 and 4
Description: Mean pneumococcal concentrations (ug/mL) at vaccine baseline (visit 2) and post-vaccination visits (visits 3 and 4) by serotype. The stated number of participants analyzed was the total number of participants in each group. The actual number of participants analyzed for each serotype varied, and is provided for each individually.
  ug/mL=micrograms per milliliter
Time Frame: From vaccine sub-study visit 2 (baseline) to sub-study visit 4
Population: Evaluable Immunogenicity Population
Measure: Geometric Mean (95% Confidence Interval); unit: Concentration (ug/mL)
Groups:
- Tofacitinib 10 mg BID Continuous Visit 2; Tofacitinib 10 mg BID Continuous Visit 3; Tofacitinib 10 mg BID Continuous Visit 4: Participants receiving continuous tofacitinib treatment
- Tofacitinib 10 mg BID Interrupted Visit 2; Tofacitinib 10 mg BID Interrupted Visit 3: Participants whose treatment with tofacitinib was interrupted for 2 weeks post-randomization
- Tofacitinib 10 mg BID Interrupted Visit 4: Patients whose treatment with tofacitinib was interrupted for 2 weeks post-randomization
Arm/Group | Tofacitinib 10 mg BID Continuous Visit 2 | Tofacitinib 10 mg BID Interrupted Visit 2 | Tofacitinib 10 mg BID Continuous Visit 3 | Tofacitinib 10 mg BID Interrupted Visit 3 | Tofacitinib 10 mg BID Continuous Visit 4 | Tofacitinib 10 mg BID Interrupted Visit 4
Number analyzed (Participants) | 92 | 91 | 92 | 91 | 92 | 91
Concentration (ug/mL)
  Serotype 9V: number analyzed (Participants) | 92 | 90 | 91 | 91 | 92 | 91
  Serotype 9V | 1.31 [1.08 to 1.60] | 1.12 [0.89 to 1.42] | 2.00 [1.64 to 2.44] | 2.26 [1.78 to 2.87] | 4.16 [3.29 to 5.27] | 4.80 [3.75 to 6.16]
  Serotype 14: number analyzed (Participants) | 92 | 91 | 91 | 91 | 92 | 91
  Serotype 14 | 2.31 [1.79 to 2.98] | 2.05 [1.59 to 2.63] | 4.02 [3.04 to 5.32] | 5.03 [3.77 to 6.71] | 12.09 [8.76 to 16.69] | 15.01 [10.80 to 20.88]
  Serotype 18C: number analyzed (Participants) | 92 | 91 | 91 | 91 | 92 | 91
  Serotype 18C | 1.08 [0.86 to 1.36] | 0.89 [0.70 to 1.14] | 1.81 [1.43 to 2.29] | 2.41 [1.82 to 3.18] | 4.27 [3.34 to 5.47] | 6.61 [5.01 to 8.74]
  Serotype 19F: number analyzed (Participants) | 90 | 90 | 90 | 91 | 92 | 91
  Serotype 19F | 1.17 [0.92 to 1.50] | 1.18 [0.89 to 1.58] | 1.61 [1.25 to 2.08] | 2.17 [1.61 to 2.91] | 3.52 [2.60 to 4.76] | 5.47 [3.98 to 7.52]
  Serotype 23F: number analyzed (Participants) | 92 | 90 | 90 | 91 | 92 | 91
  Serotype 23F | 1.25 [1.01 to 1.56] | 1.16 [0.93 to 1.44] | 1.80 [1.44 to 2.25] | 2.24 [1.75 to 2.88] | 3.44 [2.66 to 4.44] | 5.27 [3.96 to 7.02]

26. Secondary Outcome: Vaccine Sub-study. Titers of Anti-influenza Antibodies at Vaccine Sub-study Visit 3 and 4
Description: Mean influenza antibody titers at visits 3 and 4.
Time Frame: From vaccine sub-study visit 2 (baseline) to sub-study visit 4
Population: Evaluable Immunogenicity Population
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody Titer
Arm/Group | Tofacitinib 10 mg BID Continuous Visit 2 | Tofacitinib 10 mg BID Interrupted Visit 2 | Tofacitinib 10 mg BID Continuous Visit 3 | Tofacitinib 10 mg BID Interrupted Visit 3 | Tofacitinib 10 mg BID Continuous Visit 4 | Tofacitinib 10 mg BID Interrupted Visit 4
Number analyzed (Participants) | 92 | 91 | 91 | 91 | 92 | 91
Antibody Titer
  HAI B | 11.43 [9.38 to 13.91] | 10.85 [8.90 to 13.22] | 23.29 [17.92 to 30.27] | 37.45 [28.17 to 49.78] | 38.06 [28.71 to 50.47] | 45.19 [35.01 to 58.34]
  HAI H1N1 | 15.14 [11.67 to 19.64] | 20.26 [14.86 to 27.62] | 52.75 [37.97 to 73.28] | 105.2 [70.76 to 156.5] | 120.2 [89.83 to 160.8] | 136.0 [97.67 to 189.4]
  HAI H3N2 | 18.18 [13.53 to 24.44] | 17.30 [12.98 to 23.07] | 55.07 [38.19 to 79.43] | 83.10 [57.38 to 120.4] | 141.8 [102.9 to 195.4] | 147.2 [107.8 to 201.0]

ADVERSE EVENTS:
Time Frame: 114 months for Initial Period; 13 months for Extension Period
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) | Initial Period: Tofacitinib 10 mg BID | Initial Period: All Tofacitinib | Extension Period: Tofacitinib 5 mg
All-Cause Mortality (participants affected / at risk) | 25/1123 | 30/3358 | 55/4481 | 0/48
Serious Adverse Events (participants affected / at risk) | 346/1123 | 997/3358 | 1343/4481 | 5/48
Other Adverse Events (participants affected / at risk) | 807/1123 | 2422/3358 | 3229/4481 | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) (N=1123) | Initial Period: Tofacitinib 10 mg BID (N=3358) | Initial Period: All Tofacitinib (N=4481) | Extension Period: Tofacitinib 5 mg (N=48)
Anaemia (Blood and lymphatic system disorders) | 4 | 10 | 14 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 3 | 4 | 0
Mastocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 4 | 8 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 3 | 5 | 8 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 1 | 3 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 14 | 20 | 0
Atrial flutter (Cardiac disorders) | 2 | 1 | 3 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 2 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 2 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 2 | 0
Cardiac failure (Cardiac disorders) | 3 | 5 | 8 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 3 | 7 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 3 | 1 | 4 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 1 | 0
Coronary artery disease (Cardiac disorders) | 4 | 11 | 15 | 0
Coronary artery stenosis (Cardiac disorders) | 2 | 0 | 2 | 0
Coronary artery thrombosis (Cardiac disorders) | 1 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 1 | 0
Long QT syndrome (Cardiac disorders) | 0 | 1 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 1 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 8 | 13 | 21 | 0
Myocardial ischaemia (Cardiac disorders) | 4 | 3 | 7 | 0
Palpitations (Cardiac disorders) | 2 | 1 | 3 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 2 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 2 | 3 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 2 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1 | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 1 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 1 | 0
Tourette's disorder (Congenital, familial and genetic disorders) | 0 | 1 | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 2 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 3 | 4 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 1 | 0
Goitre (Endocrine disorders) | 3 | 7 | 10 | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 4 | 4 | 0
Cataract (Eye disorders) | 2 | 8 | 10 | 0
Glaucoma (Eye disorders) | 0 | 2 | 2 | 0
Keratitis interstitial (Eye disorders) | 0 | 1 | 1 | 0
Necrotising retinitis (Eye disorders) | 1 | 0 | 1 | 0
Optic disc drusen (Eye disorders) | 0 | 1 | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 2 | 2 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 1 | 2 | 0
Uveitis (Eye disorders) | 0 | 2 | 2 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 3 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 5 | 6 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 8 | 10 | 0
Diverticular perforation (Gastrointestinal disorders) | 3 | 5 | 8 | 0
Diverticulum (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Duodenal polyp (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Enterocele (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Fistula of small intestine (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 4 | 7 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 2 | 3 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 4 | 5 | 0
Pancreatitis acute (Gastrointestinal disorders) | 4 | 4 | 8 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 3 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 3 | 4 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Abscess sterile (General disorders) | 0 | 1 | 1 | 0
Asthenia (General disorders) | 2 | 1 | 3 | 0
Chest discomfort (General disorders) | 2 | 1 | 3 | 0
Chest pain (General disorders) | 5 | 12 | 17 | 0
Death (General disorders) | 3 | 1 | 4 | 0
Drug ineffective (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0
Fibrosis (General disorders) | 0 | 1 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 1 | 0
Hernia (General disorders) | 0 | 1 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 2 | 4 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 3 | 0
Oedema (General disorders) | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 5 | 5 | 10 | 0
Sudden death (General disorders) | 0 | 1 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 2 | 2 | 4 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholangitis chronic (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 1 | 3 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 4 | 5 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 3 | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 10 | 13 | 23 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Gallbladder non-functioning (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatic congestion (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 2 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 1 | 2 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 1 | 0
Abscess (Infections and infestations) | 0 | 1 | 1 | 0
Abscess limb (Infections and infestations) | 1 | 3 | 4 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 6 | 11 | 17 | 0
Appendicitis perforated (Infections and infestations) | 0 | 3 | 3 | 0
Arthritis bacterial (Infections and infestations) | 1 | 4 | 5 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 3 | 3 | 0
Bacteraemia (Infections and infestations) | 1 | 2 | 3 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 1 | 0
Bartholin's abscess (Infections and infestations) | 0 | 1 | 1 | 0
Bone tuberculosis (Infections and infestations) | 1 | 1 | 2 | 0
Bronchiolitis (Infections and infestations) | 1 | 1 | 2 | 0
Bronchitis (Infections and infestations) | 3 | 5 | 8 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 1 | 0
Bursitis infective (Infections and infestations) | 0 | 2 | 2 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 14 | 16 | 0
Cellulitis gangrenous (Infections and infestations) | 0 | 1 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 2 | 2 | 0
Chronic tonsillitis (Infections and infestations) | 1 | 1 | 2 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 2 | 2 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1 | 0
Colonic abscess (Infections and infestations) | 0 | 2 | 2 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 1 | 1 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 3 | 3 | 0
Device related infection (Infections and infestations) | 1 | 3 | 4 | 0
Diabetic gangrene (Infections and infestations) | 0 | 1 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 3 | 4 | 7 | 0
Diverticulitis (Infections and infestations) | 5 | 12 | 17 | 0
Encephalitis (Infections and infestations) | 1 | 1 | 2 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 2 | 2 | 4 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 2 | 2 | 0
Eye infection fungal (Infections and infestations) | 0 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 13 | 15 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 4 | 4 | 0
Gastrointestinal viral infection (Infections and infestations) | 2 | 0 | 2 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 2 | 2 | 0
HIV infection (Infections and infestations) | 0 | 1 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 2 | 2 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 1 | 0
Hepatitis E (Infections and infestations) | 0 | 1 | 1 | 0
Herpes dermatitis (Infections and infestations) | 1 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 16 | 18 | 0
Herpes zoster cutaneous disseminated (Infections and infestations) | 0 | 1 | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 5 | 5 | 0
Herpes zoster oticus (Infections and infestations) | 0 | 1 | 1 | 0
Incision site infection (Infections and infestations) | 0 | 1 | 1 | 0
Infected seroma (Infections and infestations) | 0 | 1 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 1 | 0
Infectious colitis (Infections and infestations) | 0 | 1 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 1 | 0
Infective spondylitis (Infections and infestations) | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 3 | 0 | 3 | 0
Joint abscess (Infections and infestations) | 0 | 1 | 1 | 0
Joint tuberculosis (Infections and infestations) | 1 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1 | 0
Lyme disease (Infections and infestations) | 0 | 1 | 1 | 0
Lymph node tuberculosis (Infections and infestations) | 0 | 3 | 3 | 0
Meningitis (Infections and infestations) | 0 | 1 | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 1 | 1 | 0
Meningococcal bacteraemia (Infections and infestations) | 1 | 0 | 1 | 0
Meningoencephalitis bacterial (Infections and infestations) | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 1 | 2 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 1 | 2 | 0
Ophthalmic herpes simplex (Infections and infestations) | 0 | 2 | 2 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 4 | 4 | 0
Otitis media (Infections and infestations) | 0 | 1 | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 1 | 0
Peritoneal tuberculosis (Infections and infestations) | 0 | 1 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 3 | 4 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 1 | 0
Pertussis (Infections and infestations) | 0 | 1 | 1 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 21 | 70 | 91 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 2 | 2 | 0
Pneumonia cryptococcal (Infections and infestations) | 0 | 2 | 2 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 2 | 2 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 2 | 2 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 1 | 2 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 2 | 2 | 0
Postoperative wound infection (Infections and infestations) | 0 | 5 | 5 | 0
Primary syphilis (Infections and infestations) | 0 | 1 | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 1 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 7 | 8 | 0
Pulpitis dental (Infections and infestations) | 0 | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 3 | 2 | 5 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 5 | 6 | 0
Pyoderma streptococcal (Infections and infestations) | 0 | 1 | 1 | 0
Pyometra (Infections and infestations) | 0 | 1 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 1 | 0
Renal abscess (Infections and infestations) | 0 | 1 | 1 | 0
Renal cyst infection (Infections and infestations) | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 5 | 5 | 0
Retinitis (Infections and infestations) | 1 | 0 | 1 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 1 | 1 | 0
Secondary syphilis (Infections and infestations) | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 5 | 8 | 13 | 0
Sepsis syndrome (Infections and infestations) | 0 | 1 | 1 | 0
Septic shock (Infections and infestations) | 3 | 4 | 7 | 0
Sinusitis (Infections and infestations) | 0 | 4 | 4 | 0
Sinusitis aspergillus (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis fungal (Infections and infestations) | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 2 | 2 | 0
Splenic abscess (Infections and infestations) | 0 | 1 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 3 | 3 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1 | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Streptococcal infection (Infections and infestations) | 1 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1 | 0
Superinfection (Infections and infestations) | 0 | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 2 | 3 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 1 | 0
Toxic shock syndrome (Infections and infestations) | 0 | 1 | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 1 | 2 | 0
Tuberculosis of central nervous system (Infections and infestations) | 1 | 0 | 1 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 8 | 14 | 22 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 2 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1 | 1 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 1 | 0
Wound infection bacterial (Infections and infestations) | 0 | 1 | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 7 | 9 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Exposure via father (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 9 | 16 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 3 | 7 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 12 | 14 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 4 | 5 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 6 | 2 | 8 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 11 | 13 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 4 | 5 | 0
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 3 | 4 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 3 | 4 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 0
Maternal exposure timing unspecified (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 3 | 4 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 4 | 3 | 7 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 5 | 5 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 5 | 5 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 4 | 4 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 10 | 12 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 7 | 7 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Twiddler's syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 3 | 4 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 4 | 5 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Airway peak pressure increased (Investigations) | 0 | 1 | 1 | 0
B-lymphocyte count increased (Investigations) | 1 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 2 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 1 | 0
Cardiac murmur (Investigations) | 0 | 1 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 4 | 4 | 0
Human papilloma virus test positive (Investigations) | 0 | 1 | 1 | 0
Liver function test increased (Investigations) | 0 | 1 | 1 | 0
Metamyelocyte count increased (Investigations) | 0 | 1 | 1 | 0
Myelocyte count increased (Investigations) | 0 | 1 | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 1 | 1 | 0
Transaminases increased (Investigations) | 0 | 2 | 2 | 0
Troponin I increased (Investigations) | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 2 | 2 | 0
Weight increased (Investigations) | 0 | 2 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 6 | 9 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3 | 4 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 4 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 3 | 3 | 0
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 8 | 9 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 0
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 13 | 17 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Finger deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 5 | 12 | 17 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Hand deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 11 | 14 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 | 4 | 9 | 0
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 21 | 63 | 84 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 5 | 7 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 11 | 23 | 34 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 7 | 7 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 8 | 9 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 8 | 10 | 0
Synovial disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
5q minus syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 12 | 15 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Benign tracheal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 12 | 16 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 4 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Choroid plexus papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 4 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 5 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8 | 11 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Marginal zone lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3 | 0
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 7 | 7 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3 | 0
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 10 | 12 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 7 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 14 | 21 | 0
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1 | 1 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 2 | 2 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 1 | 0
Cerebellar ataxia (Nervous system disorders) | 0 | 2 | 2 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 2 | 2 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 4 | 5 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 6 | 8 | 0
Cervical cord compression (Nervous system disorders) | 0 | 2 | 2 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 3 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 2 | 2 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 2 | 3 | 0
Headache (Nervous system disorders) | 0 | 2 | 2 | 0
Hemianopia (Nervous system disorders) | 0 | 1 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 1 | 0
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 1 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 3 | 3 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 1 | 2 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 2 | 2 | 0
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0 | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1 | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1 | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 1 | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 2 | 3 | 0
Neuritis (Nervous system disorders) | 1 | 0 | 1 | 0
Pachymeningitis (Nervous system disorders) | 0 | 1 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 2 | 2 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 2 | 2 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 2 | 0
Quadriparesis (Nervous system disorders) | 0 | 1 | 1 | 0
Radicular syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 9 | 10 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 1 | 1 | 0
Serotonin syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Small fibre neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0
Spinal claudication (Nervous system disorders) | 0 | 2 | 2 | 0
Spinal subdural haematoma (Nervous system disorders) | 0 | 1 | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 5 | 6 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 11 | 13 | 0
Vasculitis cerebral (Nervous system disorders) | 0 | 1 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 3 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 2 | 2 | 0
Device electrical impedance issue (Product Issues) | 0 | 1 | 1 | 0
Device loosening (Product Issues) | 0 | 2 | 2 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 1 | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 2 | 0
Depression (Psychiatric disorders) | 0 | 3 | 3 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 1 | 0
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 1 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 6 | 6 | 12 | 0
Anuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Mixed incontinence (Renal and urinary disorders) | 0 | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 5 | 7 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 2 | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 3 | 4 | 0
Renal failure (Renal and urinary disorders) | 3 | 1 | 4 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1 | 0
Ureteral necrosis (Renal and urinary disorders) | 0 | 1 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 4 | 4 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2 | 2 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 2 | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 4 | 4 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Breast hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 1 | 2 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 3 | 3 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 1 | 2 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Endometrial dysplasia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 2 | 3 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 8 | 9 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 2 | 3 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 1 | 2 | 0
Uterine prolapse (Reproductive system and breast disorders) | 3 | 1 | 4 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 2 | 2 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 11 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 16 | 19 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 8 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Activities of daily living impaired (Social circumstances) | 0 | 1 | 1 | 0
Physical abuse (Social circumstances) | 0 | 1 | 1 | 0
Arthrodesis (Surgical and medical procedures) | 0 | 1 | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1 | 1 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 3 | 5 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 1 | 2 | 0
Arteriosclerosis (Vascular disorders) | 1 | 1 | 2 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 6 | 9 | 15 | 0
Extremity necrosis (Vascular disorders) | 1 | 1 | 2 | 0
Haematoma (Vascular disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 7 | 10 | 0
Hypertensive crisis (Vascular disorders) | 3 | 8 | 11 | 0
Hypotension (Vascular disorders) | 0 | 2 | 2 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 1 | 0
Peripheral venous disease (Vascular disorders) | 0 | 2 | 2 | 0
Shock (Vascular disorders) | 1 | 0 | 1 | 0
Thromboangiitis obliterans (Vascular disorders) | 0 | 1 | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 1 | 3 | 0
Varicose vein (Vascular disorders) | 0 | 5 | 5 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 1 | 0
Herpes zoster 1 (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia 1 (Infections and infestations) | 0 | 0 | 0 | 1
Humerus fracture 1 (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Basal cell carcinoma 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Depression 1 (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Period: Tofacitinib 5 Milligram(mg) Twice Daily (BID) (N=1123) | Initial Period: Tofacitinib 10 mg BID (N=3358) | Initial Period: All Tofacitinib (N=4481) | Extension Period: Tofacitinib 5 mg (N=48)
Anemia (Blood and lymphatic system disorders) | 64 | 176 | 240 | 0
Diarrhoea (Gastrointestinal disorders) | 72 | 213 | 285 | 0
Nausea (Gastrointestinal disorders) | 56 | 175 | 231 | 0
Bronchitis (Infections and infestations) | 141 | 430 | 571 | 0
Herpes zoster (Infections and infestations) | 117 | 373 | 490 | 0
Influenza (Infections and infestations) | 78 | 199 | 277 | 0
Nasopharyngitis (Infections and infestations) | 138 | 517 | 655 | 0
Pharyngitis (Infections and infestations) | 58 | 148 | 206 | 0
Sinusitis (Infections and infestations) | 70 | 239 | 309 | 0
Upper respiratory tract infection (Infections and infestations) | 228 | 613 | 841 | 0
Urinary tract infection (Infections and infestations) | 161 | 447 | 608 | 0
Fall (Injury, poisoning and procedural complications) | 64 | 209 | 273 | 0
Alanine aminotransferase increased (Investigations) | 63 | 122 | 185 | 0
Blood creatine phosphokinase increased (Investigations) | 91 | 247 | 338 | 0
Blood creatinine increased (Investigations) | 60 | 116 | 176 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 62 | 153 | 215 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 87 | 265 | 352 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 106 | 291 | 397 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 103 | 293 | 396 | 0
Headache (Nervous system disorders) | 67 | 201 | 268 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 65 | 202 | 267 | 0
Hypertension (Vascular disorders) | 139 | 311 | 450 | 0
Bronchitis 1 (Infections and infestations) | 0 | 0 | 0 | 3

LIMITATIONS AND CAVEATS:
1 serious adverse event in the reporting group "Tofacitinib 5 milligram (mg) twice daily (BID)" of Initial Period could not be coded ("septic shock and pneumonia") and has not been included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the investigator is that the sponsor can review results communications at least 30 days prior to public release and can embargo communications regarding trial results for a period that is no more than an additional 60 days. Investigators will, on request, remove any previously undisclosed confidential information (other than the study results themselves) before disclosure.